CLINICAL TRIAL: NCT02528188
Title: A PHASE 3 RANDOMIZED, DOUBLE-BLIND, ACTIVE-CONTROLLED, MULTICENTER STUDY OF THE LONG-TERM SAFETY AND EFFICACY OF SUBCUTANEOUS ADMINISTRATION OF TANEZUMAB IN SUBJECTS WITH OSTEOARTHRITIS OF THE HIP OR KNEE
Brief Title: Long Term Safety and Efficacy Study of Tanezumab in Subjects With Osteoarthritis of the Hip or Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4091058; 2012-003721-22 (EudraCT Number); OA SAFETY STUDY (Other: Alias Study Number)
Record Dates: First submitted 2015-07-19; First posted 2015-08-19 (Estimated); Results first posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2019-12

CONDITIONS: Chronic Pain; Osteoarthritis, Hip; Osteoarthritis, Knee
MeSH Terms: conditions — Chronic Pain; Osteoarthritis, Hip; Osteoarthritis, Knee | interventions — Anti-Inflammatory Agents, Non-Steroidal; tanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NSAID (Active Comparator): Subcutaneous injection of placebo for tanezumab every 8 weeks plus oral NSAID (naproxen 500 mg, celecoxib 100 mg or diclofenac 75 mg) twice daily for 56 weeks
  Interventions: Drug: NSAID
- Tanezumab 2.5 mg (Experimental): Subcutaneous injection of tanezumab 2.5 mg every 8 weeks plus oral placebo for NSAID (naproxen, celecoxib or diclofenac ER) twice daily for 56 weeks
  Interventions: Biological: Tanezumab 2.5 mg
- Tanezumab 5 mg (Experimental): Subcutaneous injection of tanezumab 5 mg every 8 weeks plus oral placebo for NSAID (naproxen, celecoxib or diclofenac) twice daily for 56 weeks
  Interventions: Biological: Tanezumab 5 mg

INTERVENTIONS:
Drug: NSAID — Orally administered NSAID (naproxen 500 mg, celecoxib 100 mg or diclofenac 75 mg) twice daily for 56 weeks
  Arms: NSAID
Biological: Tanezumab 2.5 mg — Subcutaneous injection of tanezumab 2.5 mg every 8 weeks for 56 weeks
  Arms: Tanezumab 2.5 mg
Biological: Tanezumab 5 mg — Subcutaneous injection of tanezumab 5 mg every 8 weeks for 56 weeks
  Arms: Tanezumab 5 mg

SUMMARY:
The purpose of this study is to compare the long-term joint safety and efficacy (pain relief) of the investigational study drug, tanezumab compared to non-steroidal anti inflammatory drugs (NSAIDs) in subjects with osteoarthritis of the hips or knees.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of osteoarthritis of the index hip or knee based on American College of Rheumatology criteria with Kellgren Lawrence X ray Grade of 2 as diagnosed by the Central Reader
* Currently receiving a stable dose regimen of oral NSAID (naproxen, celecoxib, diclofenac, aceclofenac, loxoprofen, ibuprofen, meloxicam, nabumetone, sulindac or ketoprofen) as described in the protocol along with a history of insufficient pain relief from, inability to tolerate or contraindication to taking acetaminophen and, tramadol or opioid treatments. Subjects must also maintain a stabilized, protocol specified NSAID dose regimen for at least the final 2 or 3 weeks of the Screening period
* WOMAC Pain subscale score of at least 5 in the index knee or hip at Screening
* Be willing to discontinue all non study pain medications for osteoarthritis and not use prohibited pain medications throughout the duration of the study
* Female subjects of childbearing potential must agree to comply with protocol specified contraceptive requirements

Exclusion Criteria:

* Subjects exceeding protocol defined BMI or body weight limits
* History of other diseases specified in the protocol (eg, inflammatory joint diseases, crystalline diseases such as gout or pseudogout) that may involve the index joint and that could interfere with efficacy assessments
* Radiographic evidence of protocol specified bone or joint conditions in any screening radiograph as determined by the central radiology reviewer
* A history of osteonecrosis or osteoporotic fracture
* History of significant trauma or surgery to a knee, hip or shoulder within the previous year
* Planned surgical procedure during the duration of the study
* Presence of conditions (eg, fibromyaliga, radiculopathy) associated with moderate to severe pain that may confound assessments or self evaluation of osteoarthritis pain
* Signs or symptoms of carpal tunnel syndrome in the year prior to Screening
* Considered unfit for surgery based upon American Society of Anesthesiologists physical classification system for surgery grading, or subjects who would not be willing to undergo joint replacement surgery if required
* Contraindications to magnetic resonance imaging
* History of intolerance or hypersensitivity to the oral NSAID (naproxen, celecoxib or diclofenac) the subject could be randomized to receive or any of its excipients or existence of a medical condition or use of concomitant medication for which the use of this NSAID is contraindicated
* History of intolerance or hypersensitivity to acetaminophen or any of its excipients or existence of a medical condition or use of concomitant medication for which the use of acetaminophen is contraindicated
* Use of prohibited medications without the appropriate washout period prior to Screening or Initial Pain Assessment Period
* History of cancer within 5 years of Screening, except for cutaneous basal cell or squamous cell cancer resolved by excision
* Subjects with signs and symptoms of clinically significant cardiac disease as described in the protocol
* Diagnosis of a transient ischemic attack in the 6 months prior to Screening, diagnosis of stroke with residual deficits that would preclude completion of required study activities
* History, diagnosis, or signs and symptoms of clinically significant neurological disease such as but not limited to peripheral or autonomic neuropathy
* History, diagnosis, signs or symptoms of any clinically significant psychiatric disorder
* History of known alcohol, analgesic or drug abuse within 2 years of Screening
* Previous exposure to exogenous NGF or to an anti-NGF antibody
* History of allergic or anaphylactic reaction to a therapeutic or diagnostic monoclonal antibody or IgG fusion protein
* Poorly controlled hypertension as defined in the protocol or taking an antihypertensive that has not been stable for at least 1 month prior to Screening
* Evidence of protocol defined orthostatic hypotension at Screening
* Disqualifying score on the Survey of Autonomic Symptoms questionnaire at Screening
* Screening AST, ALT, serum creatinine or HbA1c values that exceed protocol defined limits
* Presence of drugs of abuse in screening urine toxicology panel
* Positive hepatitis B, hepatitis C or HIV test results indicative of current infection
* Participation in other investigational drug studies within protocol defined time limits
* Pregnant, breastfeeding or female subjects of childbearing potential who are unwilling or unable to follow protocol required contraceptive requirements
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that in the judgment of the investigator, would make the subject inappropriate for entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3021 (Actual)
Dates: Start 2015-07-21 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2019-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (500):
- United States (299):
  - Central Alabama Research, Birmingham, Alabama
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Alabama Orthopaedic Surgeons, Birmingham, Alabama
  - Rheumatology Associates of North Alabama, PC, Huntsville, Alabama
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Ferguson Family Medicine, Mesa, Arizona
  - Arizona Arthritis & Rheumatology Associates, P.C., Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Valley Pain Consultants, Scottsdale, Arizona
  - Clinical Research Consortium, Tempe, Arizona
  - Noble Clinical Research, LLC, Tucson, Arizona
  - Quality of Life Medical & Research Centers, LLC, Tucson, Arizona
  - Tucson Orthopaedic Institute - Research Center, Tucson, Arizona
  - CHI St. Vincent Medical Group Hot Springs, Hot Springs, Arkansas
  - Chrystal Johnson, Little Rock, Arkansas
  - KLR Business Group, Inc., dba Arkansas Clinical Research, Little Rock, Arkansas
  - Larry Watkins, MD, Little Rock, Arkansas
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Orange County Research Institute, Anaheim, California
  - Advanced Research Center, Anaheim, California
  - CITrials, Bellflower, California
  - Osteoporosis Medical Center, Beverly Hills, California
  - Hope Clinical Research, Canoga Park, California
  - Med Center, Carmichael, California
  - Core Healthcare Group, Cerritos, California
  - Pleitez Medical Clinic, Covina, California
  - Triwest Research Associates, LLC, El Cajon, California
  - T. Joseph Raoof MD, INC/Encino Research Center, Encino, California
  - San Diego Imaging Escondido, Escondido, California
  - Med Investigations, Inc., Fair Oaks, California
  - Research Center of Fresno, Inc., Fresno, California
  - Neuro-Pain Medical Center, Fresno, California
  - Collaborative Neuroscience Network, LLC., Garden Grove, California
  - Allied Clinical Research, Gold River, California
  - HealthCare Partners Clinical Research, LLC., Huntington Beach, California
  - Marvel Clinical Research LLC, Huntington Beach, California
  - BioSolutions Clinical Research Center, La Mesa, California
  - eStudySite, La Mesa, California
  - Arthritis & Osteoporosis Medical Center, La Palma, California
  - Center For United Research, Inc., Lakewood, California
  - Collaborative Neuroscience Network, LLC., Long Beach, California
  - Aeon Research, Inc., Los Angeles, California
  - American Institute of Research, Los Angeles, California
  - InterMed Medical Group, Los Angeles, California
  - IMD Medical Group, Los Angeles, California
  - Catalina Research Institute, LLC, Montclair, California
  - Providence Clinical Research, North Hollywood, California
  - Renaissance Imaging Medical Associates, Inc, Northridge, California
  - NRC Research Institute, Orange, California
  - Advances in Medicine, Palm Desert, California
  - Probe Clinical Research Corporation, Riverside, California
  - University of California, Davis Health System, Sacramento, California
  - University of California, Davis Medical Center, Sacramento, California
  - Clinical Trials Research, Sacramento, California
  - Northern California Research, Sacramento, California
  - Center for Clinical Trials of Sacramento, Inc., Sacramento, California
  - Artemis Institute for Clinical Research, San Diego, California
  - San Diego Imaging, Kearny Mesa, San Diego, California
  - Sharp and Children's MRI Center, LLC, San Diego, California
  - Artemis Institute for Clinical Research, San Marcos, California
  - CITrials, Santa Ana, California
  - Syrentis Clinical Research, Santa Ana, California
  - Shariar Cohen, MD Corp., Thousand Oaks, California
  - Westlake Medical Research, Thousand Oaks, California
  - Bayview Research Group, Valley Village, California
  - Renaissance Imaging Medical Associates, Inc, Van Nuys, California
  - Buhay & Maglunog MDS, West Covina, California
  - Prohealth Advanced Imaging, West Hills, California
  - Advanced Rx Clinical Research Group, Inc, Westminster, California
  - Medvin Clinical Research, Whittier, California
  - Elite Clinical Trials, Wildomar, California
  - Mountain View Clinical Research, Inc., Denver, Colorado
  - Mountain View Clinical Research, Inc, Denver, Colorado
  - New England Research Associates, LLC, Bridgeport, Connecticut
  - Clinical Research Center of CT, Danbury, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Delaware Arthritis, Lewes, Delaware
  - Javed Rheumatology Associates, Inc., Newark, Delaware
  - JEM Research Institute, Atlantis, Florida
  - AARDS Research, Inc., Aventura, Florida
  - RASF-Clinical Research, Inc, Boca Raton, Florida
  - Orthopedic Research Institute, Boynton Beach, Florida
  - Meridien Research, Brooksville, Florida
  - Orthopaedic Associates of West Florida, Clearwater, Florida
  - Tampa Bay Medical Research, Inc, Clearwater, Florida
  - Midland Florida Clinical Research Center, LLC, DeLand, Florida
  - S&W Clinical Research, Fort Lauderdale, Florida
  - Centre for Rheumatology, Immunology and Arthritis, Fort Lauderdale, Florida
  - Clinical Physiology Associates, Fort Myers, Florida
  - IMA, Fort Myers, Florida
  - SIMEDHealth, LLC, Gainesville, Florida
  - South Florida Clinical Trials, Hialeah, Florida
  - Pines Clinical Research Inc., Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Care Partners Clinical Research, Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Columbus Clinical Services LLC, Miami, Florida
  - Pharmax Research Clinic, Inc., Miami, Florida
  - Clintex Research Group, Miami, Florida
  - Center for Arthritis and Rheumatic Diseases, Miami, Florida
  - Larkin Imaging Center, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - International Research Associates, LLC, Miami, Florida
  - M&M Medical Center, Inc., Miami, Florida
  - Quality Research & Medical Center LLC, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - American Family Medical, Ocala, Florida
  - Sensible Healthcare, LLC., Ocoee, Florida
  - Journey Research, Inc., Oldsmar, Florida
  - Sunshine Research Center, Opa-locka, Florida
  - Compass Research, LLC, Orlando, Florida
  - Rheumatology Associates of Central Florida, P.A., Orlando, Florida
  - Omega Research Consultants, LLC, Orlando, Florida
  - Oviedo Medical Research, LLC, Oviedo, Florida
  - Pensacola Research Consultants, Inc., d.b.a. Avanza Medical Research Center, Pensacola, Florida
  - Sacred Heart Orthopedics, Pensacola, Florida
  - Orthopaedic Center of South Florida, Plantation, Florida
  - St. Johns Center for Clinical Research, Ponte Vedra, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Accord Clinical Research, LLC, Port Orange, Florida
  - Gulfcoast Research Institute, LLC, Sarasota, Florida
  - Kennedy White Orthopaedic Center, Sarasota, Florida
  - Meridien Research, St. Petersburg, Florida
  - Precision Clinical Research, LLC., Sunrise, Florida
  - Phoenix Clinical Research, LLC., Tamarac, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - BayCare Medical Group, Inc, Tampa, Florida
  - Compass Research North LLC, The Villages, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Perimeter Institute for Clinical Research, Inc. DBA:/PICR Clinic, Atlanta, Georgia
  - Masters of Clinical Research, Inc., Augusta, Georgia
  - River Birch Research Alliance, LLC, Blue Ridge, Georgia
  - Arthritis Center of North Georgia, Gainesville, Georgia
  - Center for Advanced Research & Education, Gainesville, Georgia
  - Drug Studies America, Marietta, Georgia
  - Better Health Clinical Research, Inc., Newnan, Georgia
  - Atlanta Orthopaedic Institute, LLC, Stockbridge, Georgia
  - Herman Clinical Research, LLC, Suwanee, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - North Georgia Internal Medicine, Woodstock, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Idaho Sports Medicine Institute, Boise, Idaho
  - Injury Care Research, LLC, Boise, Idaho
  - Institute Of Arthritis Research, Idaho Falls, Idaho
  - Advanced Clinical Research, Meridian, Idaho
  - Medex Healthcare Research, Inc., Chicago, Illinois
  - Chicago Clinical Research Institute Inc., Chicago, Illinois
  - Northwestern Memorial Hospital-Arkes Pavilion, Diagnostic Testing Center, Chicago, Illinois
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Affinity Clinical Research Institute, Oak Lawn, Illinois
  - Southwest Center for Healthy Joints, S.C., Oak Lawn, Illinois
  - Methodist Research Administration Office, Peoria, Illinois
  - UnityPoint Clinic Rheumatology, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OrthoIllinois, Rockford, Illinois
  - Quest Diagnostics, Rockford, Illinois
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Buynak Clinical Research, P.C., Valparaiso, Indiana
  - Mid-America Physiatrists, P.A., Overland Park, Kansas
  - Phoenix Medical Research, Inc., Prairie Village, Kansas
  - Professional Research Network of Kansas, LLC, Wichita, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Otrimed Corporation, Edgewood, Kentucky
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - Baton Rouge General Medical Center-Internal Medicine Clinic, Baton Rouge, Louisiana
  - Baton Rouge General Medical Center-Midcity, Baton Rouge, Louisiana
  - Baton Rouge General Medical Center-Bluebonnet, Baton Rouge, Louisiana
  - Baton Rouge General Medical Center-Clinical Trials Office, Baton Rouge, Louisiana
  - Centex Studies, Inc., Lake Charles, Louisiana
  - Klein & Associates, M.D., P.A., Cumberland, Maryland
  - Arthritis Treatment Center, Frederick, Maryland
  - Klein & Associates, M.D., P.A., Hagerstown, Maryland
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Beacon Clinical Research, LLC, Quincy, Massachusetts
  - MedVadis Research Corporation, Watertown, Massachusetts
  - Great Lakes Research Group, Incorporated, Bay City, Michigan
  - Onyx Clinical Research, Caro, Michigan
  - Orthopaedic Associates of Michigan, PC, Grand Rapids, Michigan
  - June D.O. PC, Lansing, Michigan
  - Great Lakes Research Group, Pinconning, Michigan
  - Michigan Orthopaedic Spine Surgeons, Rochester Hills, Michigan
  - Medical Research Associates Inc., Traverse City, Michigan
  - Oakland Medical Research Center, Troy, Michigan
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Landmark Internal Medicine, Southaven, Mississippi
  - University of Missouri Health Care-Investigational Pharmacy, Columbia, Missouri
  - University of Missouri Health Care, Columbia, Missouri
  - University of Missouri School of Medicine- Clinical Research Center, Columbia, Missouri
  - Advance Clinical Research, Inc., St Louis, Missouri
  - Medex Healthcare Research, Inc., St Louis, Missouri
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - Affiliated Clinical Research, Inc., Las Vegas, Nevada
  - Impact Clinical Trials, Las Vegas, Nevada
  - Office of Stephen H. Miller, MD, Las Vegas, Nevada
  - Clinical Research Consortium, Las Vegas, Nevada
  - Office of Robert P. Kaplan, DO, Las Vegas, Nevada
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - G. Timothy Kelly, MD, Las Vegas, Nevada
  - ActivMed Practices & Research, Inc., Portsmouth, New Hampshire
  - Ocean Rheumatology, PA, Toms River, New Jersey
  - Premier Research, Trenton, New Jersey
  - Arthritis, Rheumatic and Back Disease Associates, PA, Voorhees Township, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - New Mexico Clinical Research & Osteoporosis Center, Inc., Albuquerque, New Mexico
  - Lovelace Scientific Resources Inc., Albuquerque, New Mexico
  - NYU Langone Ambulatory Care Brooklyn Heights, Brooklyn, New York
  - Drug Trials Brooklyn, Brooklyn, New York
  - SPRI Clinical Trials, LLC, Brooklyn, New York
  - Drug Trials America, Hartsdale, New York
  - NYU Langone Arena Oncology, Laura and Issac Perlmutter Cancer Center, Infusion Center, Lake Success, New York
  - NYU Langone Arena Oncology, Laura and Issac Perlmutter Cancer Center, Lake Success, New York
  - NYU Langone Rheumatology Associates Long Island, Lake Success, New York
  - Lenox Hill Radiology, New York, New York
  - Manhattan Medical Research Practice PLLC, New York, New York
  - The Medical Research Network, LLC, New York, New York
  - AAIR Research Center, Rochester, New York
  - Upstate Clinical Research Associates, LLC, Williamsville, New York
  - Northstate Clinical Research, PLLC, Lenoir, North Carolina
  - Wake Internal Medicine Consultants, Inc, Raleigh, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Lillestol Research, LLC, Fargo, North Dakota
  - Plains Clinical Research Center, LLC, Fargo, North Dakota
  - Valley Medical Research/Valley Medical Primary Care, Centerville, Ohio
  - Hightop Medical Research Center, Cincinnati, Ohio
  - New Horizons Clinical Research, Cincinnati, Ohio
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Aventiv Research Inc., Columbus, Ohio
  - Remington-Davis, Incorporated, Columbus, Ohio
  - Optimed Research LTD, Columbus, Ohio
  - Dayton Clinical Research, Dayton, Ohio
  - PriMed Clinical Research, Dayton, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Springboro Health Center, Springboro, Ohio
  - AC Clinical Research, Tiffin, Ohio
  - Glendale Medical Center, Toledo, Ohio
  - Bone Joint & Spine Surgeons, Inc., Toledo, Ohio
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - University Orthopedics Center, Altoona, Pennsylvania
  - Heritage Valley Medical Group, Inc., Beaver, Pennsylvania
  - Brandywine Clinical Research, Downingtown, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - The Clinical Trial Center LLC, Jenkintown, Pennsylvania
  - Founders Research Corporation, Philadelphia, Pennsylvania
  - The Arthritis Group, Philadelphia, Pennsylvania
  - Clinical Research Center of Reading, LLC, Wyomissing, Pennsylvania
  - Main Street Physician's Care - Waterway, Little River, South Carolina
  - Main Street Physician's Care - Loris, Loris, South Carolina
  - North Myrtle Beach Family Practice, North Myrtle Beach, South Carolina
  - Clinical Research Solutions, Jackson, Tennessee
  - Physicians Quality Care, Jackson, Tennessee
  - PMG Research, Inc. d/b/a PMG Research of Knoxville, Jefferson City, Tennessee
  - PCET Research Center, LLC, Knoxville, Tennessee
  - Diagnostic Imaging PC, Memphis, Tennessee
  - ARC Clinical Research at Wilson Parke, Austin, Texas
  - Tekton Research, Inc., Austin, Texas
  - Urgent Care MD's, Baytown, Texas
  - Texas Orthopedic Specialists, PLLC, Bedford, Texas
  - Galenos Research, Dallas, Texas
  - Abigail R. Neiman, MD, PA, Houston, Texas
  - Advances in Health, Houston, Texas
  - Mercury Clinical Research, Inc., Houston, Texas
  - Centex Studies, Inc., Houston, Texas
  - Memorial Pulmonology, Houston, Texas
  - BI Research Center, Houston, Texas
  - Clinical Investigations of Texas, Plano, Texas
  - ClinRX Research, Richardson, Texas
  - Quality Research, Inc., San Antonio, Texas
  - Lee Medical Associates PA, San Antonio, Texas
  - Progressive Clinical Research, PA, San Antonio, Texas
  - Sun Research Institute, San Antonio, Texas
  - Panacea Clinical Research, San Antonio, Texas
  - Accurate Clinical Research Inc., San Antonio, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Victorium Clinical Research, San Antonio, Texas
  - DCT-Stone Oak, LLC dba Discovery Clinical Trials, San Antonio, Texas
  - South Texas Radiology Imaging Centers, San Antonio, Texas
  - Envision Imaging, Southlake, Texas
  - Oakbend Medical Center, Sugar Land, Texas
  - ClinPoint Trials, Waxahachie, Texas
  - Mercury Clinical Research, Webester, Texas
  - Clinics of North Texas, Wichita Falls, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - Granger Medical Clinic-Riverton, Riverton, Utah
  - Millennium Clinical Trials, LLC, Arlington, Virginia
  - Charlottesville Medical Research Center, LLC, Charlottesville, Virginia
  - Millennium Clinical Trials, Fairfax, Virginia
  - National Clinical Research-Norfolk, Inc., Norfolk, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Optimed Research, LTD, Bellingham, Washington
  - Swedish Medical Center Investigational Drug Services Pharmacy, Seattle, Washington
  - Seattle Rheumatology Associates, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
- Australia (18):
  - Genesis Research Services, Broadmeadow, New South Wales
  - Hunter Imaging Group, Cardiff, New South Wales
  - Optimus Clinical Research Pty Ltd, Kogarah, New South Wales
  - Southern Radiology, Miranda, New South Wales
  - Royal Hospital for Women, Randwick, New South Wales
  - Castlereagh Imaging, St Leonards, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Australian Clinical Research Network, Sydney, New South Wales
  - Spectrum Medical Imaging, Sydney, New South Wales
  - AusTrials Pty Ltd, Sherwood, Queensland
  - CMAX Clinical Research Pty Ltd, Adelaide, South Australia
  - Royal Adelaide Hospital Pharmacy, Adelaide, South Australia
  - Bensons Radiology, North Adelaide, South Australia
  - Emeritus Research, Camberwell, Victoria
  - Capital Radiology-Malvern, Melbourne, Victoria
  - Capital Radiology-Clayton, Melbourne, Victoria
  - SKG Radiology Hollywood, Nedlands, Western Australia
  - RK Will Pty Ltd, Victoria Park, Western Australia
- Brazil (3):
  - CMIP-Centro Mineiro de Pesquisa LTDA, Juiz de Fora, Minas Gerais
  - CCBR - Centro de Pesquisas e Analises Clinicas LTDA, Rio de Janeiro, Rio de Janeiro
  - CEPIC - Centro Paulista de Investigacao Clinica e Servicos Medicos Ltda, São Paulo, São Paulo
- Bulgaria (9):
  - Diagnostic Consultative Center "Sveti Georgi" EOOD, Plovdiv
  - Medical Center "Health for all" - EOOD, Plovdiv
  - UMHAT Kaspela - EOOD Rheumatology Clinic, Plovdiv
  - UMHAT Kaspela - EOOD, Plovdiv
  - "Medical Center Teodora" EOOD, Rousse
  - Diagnostic Consultative Center 17 Sofia EOOD, Sofia
  - UMHAT Sveti Ivan Rilski- EAD, Sofia
  - UMHAT "Sofiamed" OOD, Block 2, Sofia
  - "Medical Center- Dr. Hayvazov" EOOD, Sofia
- Colombia (2):
  - Centro Integral de Reumatologia Reumalab S.A.S., Medellín, Antioquia
  - Centro de Investigacion en Reumatologia y Especialidades Medicas SAS CIREEM SAS, Bogotá, Bogota DC
- Medicinski centar Kuna&Peric, Zagreb, Croatia
- Japan (53):
  - National Hospital Organization Toyohashi Medical Center, Toyohashi, Aichi-ken
  - Funabashi Municipal Medical Center, Funabashi, Chiba
  - Matsudo City General Hospital, Matsudo, Chiba
  - Kanbara Clinic, Kitakyushu, Fukuoka
  - Hidaka Orthopedic Hospital, Kurume, Fukuoka
  - Obase Hospital, Miyako-gun, Fukuoka
  - Himeno Hospital, Yamegun, Fukuoka
  - Ikeda Kinen Hospital, Sukagawa, Fukushima
  - Zenshukai Hospital, Maebashi, Gunma
  - Mazda Hospital, Aki-gun, Hiroshima
  - Medical Corporation Okimoto Clinic, Kure, Hiroshima
  - Medical Corporation Emu Emukai, Matterhorn Rehabilitation Hospital, Kure, Hiroshima
  - Takahashi Orthopedics Clinic, Chitose, Hokkaido
  - Obihiro Orthopaedic Hospital, Obihiro, Hokkaido
  - Okubo Hospital, Akashi, Hyōgo
  - Omuro Orthopedic Clinic, Himeji, Hyōgo
  - Medical corporate corporation hoshikai Onishi medical clinic, Kako-gun, Hyōgo
  - Kobe Red Cross Hospital, Kobe, Hyōgo
  - Mito Saiseikai General Hospital, Mito, Ibaraki
  - National Hospital Organization Kanazawa Medical Center, Kanazawa, Ishikawa-ken
  - Kokan Clinic, Kawasaki, Kanagawa
  - Misugikai Medical Corporation Otokoyama Hospital, Yawata, Kyoto
  - Nakajo Orthopedic Clinic, Sendai, Miyagi
  - Marunouchi Hospital, Matsumoto, Nagano
  - Oita University Hospital, Yufu, Oita Prefecture
  - Sobajima Clinic/Orthopedics, Higashiosaka, Osaka
  - Rinku General Medical Center, Izumisano, Osaka
  - Kishiwada Tokushukai Hospital, Kishiwada, Osaka
  - Social Welfare Organization Saiseikai Imperial Gift Foundation,Inc. Osaka Saiseikai Nakatsu Hospital, Osaka, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Shimane University Hospital, Izumo, Shimane
  - Fujieda Municipal General Hospital, Fujieda, Shizuoka
  - JA Shizuoka Kohseiren Enshu Hospital, Hamamatsu, Shizuoka
  - Japanese Red Cross Hamamatsu Hospital, Hamamatsu, Shizuoka
  - Sonodakai Joint Replacement Center Hospital, Adachi-ku, Tokyo
  - Medical Plaza Edogawa, Edogawa-ku, Tokyo
  - Sato Orthopaedic Clinic, Edogawa-ku, Tokyo
  - Fussa Hospital, Fussa, Tokyo
  - Jukoukai hospital, Koto-ku, Tokyo
  - Kitasato University Kitasato Institute Hospital, Minato-ku, Tokyo
  - Tamagawa Hospital, Setagaya-ku, Tokyo
  - Kohno Clinical Medicine Research Institute Daisan Kitashinagawa Hospital, Shinagawa-ku, Tokyo
  - Ohimachi Orthopaedic Clinic, Shinagawa-ku, Tokyo
  - Japan Organization of Occupational Health and Safety Sanin Rosai Hospital, Yonago, Tottori
  - National Hospital Organization Chiba Medical Center, Chiba
  - Chihaya Hospital, Fukuoka
  - Kuroda Orthopedic Hospital, Fukuoka
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital, Hiroshima
  - Hiroshima Prefectural Hospital, Hiroshima
  - Kumamoto Orthopaedic Hospital, Kumamoto
  - Nagayoshi General Hospital, Osaka
  - Iwasaki Orthopedic Surgery, Saitama
  - Saitama Municipal Hospital, Saitama
- Lithuania (3):
  - Saules seimos medicinos centras, Kaunas
  - Klaipeda University Hospital, Klaipėda
  - Republican Siauliai Hospital, Šiauliai
- Mexico (2):
  - Centro Hospitalario Mac, S.A. de C.V., Guadajara, Jalisco
  - Consultorio Medico del Dr. Federico Galvan Villegas, Guadalajara, Jalisco
- New Zealand (22):
  - Lakeland Clinical Trials, Rotorua, BOP
  - Otago Radiology, Dunedin, Otago
  - RMC Medical Research Ltd, Dunedin, Otago
  - South Pacific Clinical Trials, Auckland
  - TRG Imaging Lincoln Road, Auckland
  - Auckland Bone Density Ltd, Auckland
  - North Shore Hospital, Waitemata District Health Board, Auckland
  - Star Unit, North Shore Hospital, Waitemata District Health Board, Auckland
  - The Radiology Group, Auckland
  - Southern Clinical Trials- Waitemata Ltd, Auckland
  - Auckland Bone Density, Auckland
  - Optimal Clinical Trials, Auckland
  - Auckland Radiology Parnell Branch, Auckland
  - Southern Clinical Trials Ltd, Christchurch
  - Collingwood Street Pharmacy, Nelson
  - Nelson Radiology, Nelson
  - Porter Rheumatology Ltd, Nelson
  - Bay Radiology, Tauranga
  - P3 Research Ltd, Tauranga
  - Clinical Horizons NZ Ltd, Tauranga
  - P3 Research Ltd, Wellington
  - Pacific Radiology, Wellington
- Peru (8):
  - Unidad de Investigacion en Medicina Interna y Enfermedades criticas-Hogar Clinica San Juan de Dios, Cayma, Arequipa
  - Centro De Investigacion Clinica Trujillo EIRL/Clinica Peruano Americana S.A., Trujillo, La Libertad
  - ABK REUMA S.R.L. de Medicentro Biociencias/BIO CIENCIAS PERU S.R.L., Lima
  - Centro de Investigación Reumatología CAA-Clinica Anglo Americana, Lima
  - Investigaciones en Reumatologia / Centro Medico Corpac S.A., Lima
  - Centro de Investigaciones Medicas-Hospital Maria Auxiliadora, Lima
  - Investigaciones Clinicas S.A.C. / Instituto de Ginecologia y Reproduccion S.A., Lima
  - Investigaciones Clinicas S.A.C./Instituto de Ginecologia y Reproduccion S.A., Lima
- Philippines (2):
  - Philippine General Hospital, Manila, NCR
  - Manila Doctors Hospital, Manila
- Russia (10):
  - Moscow Municipal Rheumatology Center, Moscow
  - SBHI "City Clinical Hospital No. 1 n.a N.I. Pirogov", Moscow
  - SBHI "City Clinical Hospital No. 1 n.a. N.I. Pirogov", Moscow
  - Federal State Budgetary Scientific Research institution of fundamental and clinical immunology, Novosibirsk
  - Federal State Budgetary Scientific Institution, Novosibirsk
  - State Budgetary Institution of Ryazan Region, Ryazan
  - Medical Technologies Ltd, Saint Petersburg
  - Limited Liability Company "Medical Center "Reavita Med SPb", Saint Petersburg
  - Medinet LLC, Saint Petersburg
  - FSBI 'SRITO n.a. R.R. Vreden' MoH RF, Saint Petersburg
- Serbia (5):
  - Institute for Rehabilitation, Belgrade
  - Institute of Rheumatology, Belgrade
  - Institute for treatment and rehabilitation "Niska Banja", Niška Banja
  - Special Hospital for Rheumatic Diseases Novi Sad, Novi Sad
  - General hospital "Dr Laza K. Lazarevic" Sabac, Šabac
- Slovakia (6):
  - Reumatologia s.r.o., Bratislava
  - Nestatna Reumatologicka Ambulancia, Poliklinika Karlova Ves, Bratislava
  - MUDr. STRANAI s.r.o., Košice
  - Reum.hapi s.r.o., Nové Mesto nad Váhom
  - MEDIPA s.r.o., Piešťany
  - Thermium s.r.o., Piešťany
- South Korea (27):
  - Daegu Catholic University Medical Center, Daegu
  - Department of Radiology, Daegu
  - Division of Rheumatology, Department of Internal Medicine, Daegu Catholic University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Clinical Trial Center Pharmacy, Daejeon
  - Department of Radiology, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Department of Radiology, Gwangju
  - Pharmacy of Clinical Trial Center, Gwangju
  - Clinical Trial Pharmacy, Seoul
  - Department of Radiology, Seoul
  - Korea University Anam Hospital, Seoul
  - Clinical Trials Center Pharmacy, Seoul
  - Seoul National University Hospital, Seoul
  - Clinical Trial Center Pharmacy, Seoul
  - Yonsei University Health System, Severance Hospital, Seoul
  - Clinical Research Pharmacy, Seoul
  - Department of Clinical Research Pharmacy, Konkuk University Medical Center, Seoul
  - Division of Rheumatology, Department of Internal Medicine, Konkuk University Medical Center, Seoul
  - Konkuk University Medical Center, Seoul
  - Department of Orthopedic Surgery, Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - Clinical Research Pharmacy, SMG SNU Boramae Medical Center, Seoul
  - Department of Clinical Research Pharmacy, SMG-SNU Boramae Medical Center, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Clinical Trial Pharmacy, Yangcheon-gu, Seoul
- Taiwan (8):
  - Changhua Christian Hospital Clinical Trial Pharmacy, Changhua
  - Changhua Christian Hospital, Changhua
  - Chang Gung Memorial Hospital-Kaohsiung Branch Clinical Trial Pharmacy, Kaohsiung City
  - Chang Gung Memorial Hospital-Kaohsiung Branch, Kaohsiung City
  - Chung Shan Medical University Hospital Clinical Trial Pharmacy, Taichung
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - Department of Pharmacy, China Medical University Hospital, Taichung
- Ukraine (22):
  - Regional Communal Institution Chernivtsi Regional Clinical Hospital, Chernivtsi
  - Communal Non-profit Institution "City Clinical Hospital No.27" of Kharkiv City Council, Kharkiv
  - Government Institution "L.T. Malaya Therapy National Institute of the NAMS of Ukraine", Kharkiv
  - Chair of Internal Medicine #2, Kyiv
  - Oleksandrivska Clinical Hospital Of Kyiv, Kyiv
  - Kyiv City Clinical Hospital 3,Rheumatology Department, Kyiv
  - Clinic of NI "NSC"M.D.Strazhesko Institute of Cardiology" of NAMS of Ukraine,, Kyiv
  - Polyclinic of Administration of Medical Services and Rehabilitation of State Stock Holding Company, Kyiv
  - Clinic of SI "Institute of Gerontology named after D.F Chebotarov of NAMS of Ukraine", Kyiv
  - Clinic of SI Institute of Gerontology named after D.F Chebotarov of NAMS of Ukraine, Kyiv
  - National Medical University named after O O Bogomolets,, Kyiv
  - Polyclinic Of Administration of Medical Services and Rehabilitation of SSHC Artem, Kyiv
  - Communal Non-profit Institution "City Clinical Hospital #5 of Lviv", Therapeutics Department, Lviv
  - Communal Institution "Odesa Regional Clinical Hospital", Odesa
  - Multi-field Medical Center (University Clinic No.1) of Odesa National Medical University,, Odesa
  - Communal Institution Ternopil University Hospital, Ternopil
  - Vinnytsia Regional Clinical Hospital named after M.I. Pyrogov, Rheumatology Department,, Vinnytsia
  - Communal Non-commercial Enterprise "Vinnytsia City Clinical Hospital No 1", Vinnytsia
  - Medical Clinical Investigational Centre of Medical Centre Health Clinic LTD, Vinnytsia
  - Scientific and Research Institute of Invalid Rehabilitation (Educational and Scientific Medical, Vinnytsia
  - Vinnytsya Medical National University named after M.I. Pyrogov, Chair of Internal Medicine #3, Vinnytsia
  - Communal Institution Zaporizhzhya Regional Clinical Hospital, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Schnitzer TJ, Conaghan PG, Berenbaum F, Abraham L, Cappelleri JC, Bushmakin AG, Viktrup L, Yang R, Brown MT. Effect size varies based on calculation method and may affect interpretation of treatment effect: an illustration using randomised clinical trials in osteoarthritis. Adv Rheumatol. 2024 Apr 22;64(1):31. doi: 10.1186/s42358-024-00358-y. PMID 38650049
- [Derived] Guermazi A, Roemer FW, Kompel AJ, Diaz LE, Crema MD, Brown MT, Hickman A, Pixton GC, Viktrup L, Fountaine RJ, Burr A, Sherlock SP, West CR. Inter-Reader Consistency and Exclusionary Findings During Radiographic Screening for Phase 3 Trials of Tanezumab in Patients With Osteoarthritis. Osteoarthr Imaging. 2022 Sep-Dec;2(3-4):100082. doi: 10.1016/j.ostima.2022.100082. Epub 2022 Nov 15. PMID 38343426
- [Derived] Carrino JA, McAlindon TE, Schnitzer TJ, Guermazi A, Hochberg MC, Conaghan PG, Brown MT, Burr A, Fountaine RJ, Pixton GC, Viktrup L, Verburg KM, West CR. Characterization of adverse joint outcomes in patients with osteoarthritis treated with subcutaneous tanezumab. Osteoarthritis Cartilage. 2023 Dec;31(12):1612-1626. doi: 10.1016/j.joca.2023.08.010. Epub 2023 Aug 29. PMID 37652258
- [Derived] Shoji S, Suzuki A, Nouri P, Cai CH, Gaitonde P, Marshall S. Prediction of relative change in free nerve growth factor following subcutaneous administration of tanezumab, a novel monoclonal antibody to nerve growth factor. CPT Pharmacometrics Syst Pharmacol. 2023 Sep;12(9):1358-1370. doi: 10.1002/psp4.13015. Epub 2023 Jul 31. PMID 37470295
- [Derived] Hunter DJ, Schnitzer TJ, Hall J, Semel D, Davignon I, Cappelleri JC, Bushmakin AG, Abraham L. Time to first and sustained improvement in WOMAC domains among patients with osteoarthritis receiving tanezumab. Osteoarthr Cartil Open. 2022 Jul 2;4(3):100294. doi: 10.1016/j.ocarto.2022.100294. eCollection 2022 Sep. PMID 36474952
- [Derived] Atkinson J, Edwards RA, Bonfanti G, Barroso J, Schnitzer TJ. A Two-Step, Trajectory-Focused, Analytics Approach to Attempt Prediction of Analgesic Response in Patients with Moderate-to-Severe Osteoarthritis. Adv Ther. 2023 Jan;40(1):252-264. doi: 10.1007/s12325-022-02336-6. Epub 2022 Oct 27. PMID 36301512
- [Derived] Mease P, Kuritzky L, Wright WL, Mallick-Searle T, Fountaine R, Yang R, Sadrarhami M, Faison W, Johnston E, Viktrup L. Efficacy and safety of tanezumab, NSAIDs, and placebo in patients with moderate to severe hip or knee osteoarthritis and a history of depression, anxiety, or insomnia: post-hoc analysis of phase 3 trials. Curr Med Res Opin. 2022 Nov;38(11):1909-1922. doi: 10.1080/03007995.2022.2113689. Epub 2022 Aug 28. PMID 35980115
- [Derived] Schnitzer TJ, Bonfanti G, Atkinson J, Donevan S, Viktrup L, Barroso J, Whalen E, Edwards RA. Characterizing 16-Week Responder Profiles Using Group-Based Trajectory Modeling in Over 4300 Clinical Trial Participants Receiving Pharmaceutical Treatment for Moderate to Severe Osteoarthritis. Adv Ther. 2022 Oct;39(10):4742-4756. doi: 10.1007/s12325-022-02290-3. Epub 2022 Aug 12. PMID 35960482
- [Derived] Neogi T, Hunter DJ, Churchill M, Shirinsky I, White A, Guermazi A, Omata M, Fountaine RJ, Pixton G, Viktrup L, Brown MT, West CR, Verburg KM. Observed efficacy and clinically important improvements in participants with osteoarthritis treated with subcutaneous tanezumab: results from a 56-week randomized NSAID-controlled study. Arthritis Res Ther. 2022 Mar 29;24(1):78. doi: 10.1186/s13075-022-02759-0. PMID 35351194
- [Derived] Conaghan PG, Dworkin RH, Schnitzer TJ, Berenbaum F, Bushmakin AG, Cappelleri JC, Viktrup L, Abraham L. WOMAC Meaningful Within-patient Change: Results From 3 Studies of Tanezumab in Patients With Moderate-to-severe Osteoarthritis of the Hip or Knee. J Rheumatol. 2022 Jun;49(6):615-621. doi: 10.3899/jrheum.210543. Epub 2022 Mar 1. PMID 35232805
- [Derived] Brown MT, Sandroni P, Low PA, Gorson KC, Hunter DJ, Pixton GC, Fountaine RJ, Viktrup L, West CR, Verburg KM. Neurological safety of subcutaneous tanezumab versus NSAID in patients with osteoarthritis. J Neurol Sci. 2022 Mar 15;434:120184. doi: 10.1016/j.jns.2022.120184. Epub 2022 Feb 14. PMID 35217440
- [Derived] Hochberg MC, Carrino JA, Schnitzer TJ, Guermazi A, Walsh DA, White A, Nakajo S, Fountaine RJ, Hickman A, Pixton G, Viktrup L, Brown MT, West CR, Verburg KM. Long-Term Safety and Efficacy of Subcutaneous Tanezumab Versus Nonsteroidal Antiinflammatory Drugs for Hip or Knee Osteoarthritis: A Randomized Trial. Arthritis Rheumatol. 2021 Jul;73(7):1167-1177. doi: 10.1002/art.41674. Epub 2021 Jun 7. PMID 33538113
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091058&StudyName=A%20Phase%203%20Randomized%2C%20Double-blind%2C%20Active-controlled%2C%20Multicenter%20Study%20Of%20The%20Long-term%20Safety%20And%20Efficacy%20Of%20Subcutaneous%20Administration%20Of%20Tanezumab%20In%20Subjects%20With%20Osteoarthritis%20Of%20The%20Hip%20Or%20Knee

RESULTS

PARTICIPANT FLOW:
Groups:
- Tanezumab 2.5 mg: Tanezumab (RN624 or PF-04383119) 2.5 milligram (mg) injection administered subcutaneously (SC) once every 8 weeks, from Baseline (Day 1) up to Week 48 and oral placebo tablets matched to naproxen, celecoxib or diclofenac extended release (ER), twice daily, from Baseline up to Week 56.
- Tanezumab 5 mg: Tanezumab (RN624 or PF-04383119) 5 mg injection administered SC once every 8 weeks, from Baseline up to Week 48 and oral placebo tablets matched to naproxen, celecoxib or diclofenac ER, twice daily, from Baseline up to week 56.
- NSAID: Non-steroidal anti-inflammatory drug (NSAID) tablets (naproxen 500 mg, celecoxib 100 mg, or diclofenac ER 75 mg), administered orally, twice daily, from Baseline up to week 56 and placebo matched to tanezumab (RN624 or PF-04383119) injection administered SC once every 8 weeks, from Baseline up to Week 48.
Period: Overall Study
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Started | 1008 | 1005 | 1008
Treated | 1002 | 998 | 996
Completed | 741 | 729 | 757
Not Completed | 267 | 276 | 251
Not completed — Adverse Event | 23 | 22 | 8
Not completed — Protocol Violation | 4 | 6 | 4
Not completed — Lack of Efficacy | 19 | 21 | 22
Not completed — Withdrawal by Subject | 97 | 104 | 100
Not completed — Lost to Follow-up | 25 | 21 | 31
Not completed — Death | 4 | 4 | 0
Not completed — Other | 89 | 91 | 74
Not completed — Randomized but not treated | 6 | 7 | 12

BASELINE CHARACTERISTICS:
Population: Safety population included all participants treated with tanezumab or placebo SC.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID | Total
Number analyzed (Participants) | 1002 | 998 | 996 | 2996
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.30 (9.17) | 61.15 (9.57) | 60.25 (9.46) | 60.57 (9.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 637 | 654 | 662 | 1953
  Male | 365 | 344 | 334 | 1043
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 705 | 712 | 680 | 2097
  Black or African American | 166 | 162 | 186 | 514
  Asian | 110 | 95 | 99 | 304
  Other | 21 | 29 | 31 | 81

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adjudicated Primary Composite Joint Safety Outcome
Description: Any participant with incidence of an adjudicated outcome of primary osteonecrosis, rapidly progressive osteoarthritis (OA) type 1 or type 2, subchondral insufficiency fracture, or pathological fracture. Rapidly progressive OA type 1 events were those that the Adjudication Committee considered to have significant loss of joint space width (JSW) (greater than or equal to [>=] 2 millimeters [mm]) within approximately 1 year without gross structural failure. Rapidly progressive OA type 2 events were those considered to have abnormal loss/destruction of bone including limited or total collapse of at least one subchondral surface (e.g., medial femoral condyle) that is not normally present in conventional end-stage OA.
Time Frame: Baseline up to Week 80
Population: Safety population included all participants treated with tanezumab or placebo SC.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
percentage of participants | 3.9 [2.8 to 5.3] | 7.1 [5.6 to 8.9] | 1.5 [0.8 to 2.5]
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Test type: Superiority; p = 0.0123, Exact methods for risk difference; Risk Difference (RD) = 2.39, 95% CI 2-sided [0.58 to 4.68]
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; Test type: Superiority; p < 0.0001, Exact methods for risk difference; Risk Difference (RD) = 5.61, 95% CI 2-sided [3.55 to 8.14]

2. Primary Outcome: Observation Time-Adjusted Event Rate of Participants With Adjudicated Primary Composite Joint Safety Outcome
Description: Observation time was defined as the start day of first SC study medication until either the (i) date of completion of or withdrawal from study, if a participant did not have the event, or (ii) date of the event (earliest event within each participant in the case of multiple events). Primary joint safety outcome included participants with adjudicated outcome of primary osteonecrosis, rapidly progressive OA type 1 or type 2, subchondral insufficiency fracture, or pathological fracture. Event rate was calculated as the number of events per 1000 participant-years at risk.
Time Frame: Baseline up to Week 80
Population: Safety population included all participants treated with tanezumab or placebo SC.
Measure: Number (95% Confidence Interval); unit: events per 1000 participant-years
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
events per 1000 participant-years | 38.3 [28.0 to 52.5] | 71.5 [56.7 to 90.2] | 14.8 [8.9 to 24.6]
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Test type: Superiority; p = 0.0012, Poisson model for rate difference; Rate Difference = 23.5, 95% CI 2-sided [9.3 to 37.7]
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; Test type: Superiority; p < 0.0001, Poisson model for rate difference; Rate Difference = 56.7, 95% CI 2-sided [38.4 to 74.9]

3. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale at Week 16
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA. The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to OA of index joint (knee or hip) during past 48 hours. It was calculated as the mean of scores from 5 individual questions, which may not be a whole (integer) number, scored on a numerical rating scale (NRS). Scores for each question and WOMAC Pain subscale score on NRS ranged from 0 (no pain) to 10 (extreme pain), where higher scores indicated higher pain.
Time Frame: Baseline, Week 16
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or matching placebo).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
units on a scale | -3.22 (0.11) | -3.33 (0.11) | -3.07 (0.11)
Statistical Analysis 1: Comparison: Tanezumab 5 mg vs NSAID; Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC pain subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority — A graphical testing procedure was applied to maintain Type I error. Tanezumab 5 mg versus NSAID was tested first and if all primary endpoints were found significant, then the testing was continued for Tanezumab 2.5 mg versus NSAID and the key secondary endpoint (>=50% reduction from baseline in WOMAC Pain at Week 16). Primary endpoints were tested sequentially within a dose in order of WOMAC pain, WOMAC physical function, and PGA; p = 0.0148, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -0.26, 95% CI 2-sided [-0.46 to -0.05], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Tanezumab 2.5 mg vs NSAID; Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. Analysis of covariance (ANCOVA) model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC pain subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.1597, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -0.15, 95% CI 2-sided [-0.36 to 0.06], Standard Error of Mean 0.11

4. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale at Week 16
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA. Physical function refers to participant's ability to move around and perform usual activities of daily living. The WOMAC physical function subscale is a 17-item questionnaire used to assess the degree of difficulty experienced due to OA in index joint (knee or hip) during past 48 hours. It was calculated as mean of the scores from 17 individual questions, which may not be a whole (integer) number, scored on a NRS. Scores for each question and WOMAC physical function subscale score on NRS ranged from 0 (no difficulty) to 10 (extreme difficulty), where higher scores indicated extreme difficulty/worse physical function.
Time Frame: Baseline, Week 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
units on a scale | -3.27 (0.11) | -3.39 (0.11) | -3.08 (0.11)
Statistical Analysis 1: Comparison: Tanezumab 5 mg vs NSAID; Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC physical function subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0030, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -0.31, 95% CI 2-sided [-0.52 to -0.11], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: Tanezumab 2.5 mg vs NSAID; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0691, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -0.19, 95% CI 2-sided [-0.40 to 0.02], Standard Error of Mean 0.11

5. Primary Outcome: Change From Baseline in Patient's Global Assessment (PGA) of Osteoarthritis at Week 16
Description: PGA of OA was assessed by asking a question from participants: "Considering all the ways your OA in your knee or hip (index joint) affects you, how are you doing today?" Participants responded on a scale ranging from 1-5, using Interactive Response Technology (IRT), where 1=very good (no symptom and no limitation of normal activities), 2= good (mild symptoms and no limitation of normal activities), 3= fair (moderate symptoms and limitation of some normal activities), 4= poor (severe symptoms and inability to carry out most normal activities), and 5= very poor (very severe symptoms and inability to carry out all normal activities). Higher scores indicated worsening of condition.
Time Frame: Baseline, Week 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
units on a scale | -0.96 (0.04) | -0.97 (0.04) | -0.94 (0.04)
Statistical Analysis 1: Comparison: Tanezumab 5 mg vs NSAID; Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline PGA and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.3431, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -0.04, 95% CI 2-sided [-0.11 to 0.04], Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Tanezumab 2.5 mg vs NSAID; [analysis description as in outcome 5, analysis 1]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.6332, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -0.02, 95% CI 2-sided [-0.09 to 0.06], Standard Error of Mean 0.04

6. Secondary Outcome: Percentage of Participants With Adjudicated Secondary Composite Joint Safety Outcome
Description: Any participant with incidence of an adjudicated outcome of primary osteonecrosis, rapidly progressive OA type 2, subchondral insufficiency fracture, or pathological fracture. Rapidly progressive OA type 2 events were those considered to have abnormal loss/destruction of bone including limited or total collapse of at least one subchondral surface (e.g., medial femoral condyle) that is not normally present in conventional end-stage OA.
Time Frame: Baseline up to Week 80
Population: Safety population included all participants treated with tanezumab or placebo SC.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
percentage of participants | 1.0 [0.5 to 1.8] | 2.2 [1.4 to 3.3] | 0.5 [0.2 to 1.2]
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Test type: Superiority; p = 0.4082, Exact methods for risk difference; Risk Difference (RD) = 0.50, 95% CI 2-sided [-0.75 to 2.28]
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; Test type: Superiority; p = 0.0238, Exact methods for risk difference; Risk Difference (RD) = 1.70, 95% CI 2-sided [0.31 to 3.63]

7. Secondary Outcome: Observation Time-Adjusted Event Rate of Participants With Adjudicated Secondary Composite Joint Safety Outcome
Description: Observation time was defined as the start day of first SC study medication until either the (i) date of completion of or withdrawal from study, if a participant did not have the event, or (ii) date of the event (earliest event within each participant in the case of multiple events). Secondary joint safety outcome included primary osteonecrosis, rapidly progressive OA (type-2), subchondral insufficiency fracture, or pathological fracture. Event rate was calculated as the number of events per 1000 participant-years at risk.
Time Frame: Baseline up to Week 80
Population: Safety population included all participants treated with tanezumab or placebo SC.
Measure: Number (95% Confidence Interval); unit: events per 1000 participant-years
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
events per 1000 participant-years | 9.7 [5.2 to 18.1] | 21.8 [14.4 to 33.1] | 4.9 [2.1 to 11.8]
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Test type: Superiority; p = 0.2035, Poisson model for rate difference; Rate Difference = 4.8, 95% CI 2-sided [-2.6 to 12.2]
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; Test type: Superiority; p = 0.0010, Poisson model for rate difference; Rate Difference = 16.9, 95% CI 2-sided [6.8 to 27.0]

8. Secondary Outcome: Percentage of Participants With Individual Adjudicated Joint Safety Outcome
Description: Any participant with incidence of an adjudicated outcome of rapidly progressive OA (type-1 only), rapidly progressive OA (type-2 only), rapidly progressive OA (type-1 or type-2 combined), subchondral insufficiency fracture, primary osteonecrosis, and pathological fracture. Rapidly progressive OA type 1 events were those that the Adjudication Committee considered to have significant loss of JSW >=2 mm within approximately 1 year without gross structural failure. Rapidly progressive OA type 2 events were those considered to have abnormal loss/destruction of bone including limited or total collapse of at least one subchondral surface (e.g., medial femoral condyle) that is not normally present in conventional end-stage OA.
Time Frame: Baseline up to Week 80
Population: Safety population included all participants treated with tanezumab or placebo SC.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
percentage of participants
  Rapidly Progressive OA Type 1 or 2 | 3.2 [2.2 to 4.5] | 6.3 [4.9 to 8.0] | 1.2 [0.6 to 2.1]
  Rapidly Progressive OA type 1 | 2.9 [1.9 to 4.1] | 4.9 [3.7 to 6.4] | 1.1 [0.6 to 2.0]
  Rapidly Progressive OA type 2 | 0.3 [0.1 to 0.9] | 1.4 [0.8 to 2.3] | 0.1 [0.0 to 0.6]
  Primary Osteonecrosis | 0.1 [0.0 to 0.6] | 0.1 [0.0 to 0.6] | 0 [0.0 to 0.4]
  Pathological Fracture | 0 [0.0 to 0.4] | 0 [0.0 to 0.4] | 0 [0.0 to 0.4]
  Subchondral Insufficiency Fracture | 0.6 [0.2 to 1.3] | 0.7 [0.3 to 1.4] | 0.4 [0.1 to 1.0]
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Rapidly progressive OA Type 1 or 2; Test type: Superiority; p = 0.0248, Exact methods for risk difference; Risk Difference = 1.99, 95% CI 2-sided [0.31 to 4.17]
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; Rapidly Progressive OA Type 1 or 2; Test type: Superiority; p < 0.0001, Exact methods for risk difference; Risk difference = 5.11, 95% CI 2-sided [3.16 to 7.54]
Statistical Analysis 3: Comparison: Tanezumab 2.5 mg vs NSAID; Rapidly Progressive OA Type 1; Test type: Superiority; p = 0.0366, Exact methods for risk difference; Risk difference = 1.79, 95% CI 2-sided [0.16 to 3.92]
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs NSAID; Rapidly Progressive OA Type 1; Test type: Superiority; p = 0.0001, Exact methods for risk difference; Risk difference = 3.81, 95% CI 2-sided [1.99 to 6.12]
Statistical Analysis 5: Comparison: Tanezumab 2.5 mg vs NSAID; Rapidly Progressive OA Type 2; Test type: Superiority; p = 0.6168, Exact methods for risk difference; Risk difference = 0.20, 95% CI 2-sided [-0.76 to 1.71]
Statistical Analysis 6: Comparison: Tanezumab 5 mg vs NSAID; Rapidly Progressive OA Type 2; Test type: Superiority; p = 0.0388, Exact methods for risk difference; Risk difference = 1.30, 95% CI 2-sided [0.17 to 2.97]
Statistical Analysis 7: Comparison: Tanezumab 2.5 mg vs NSAID; Primary osteonecrosis; Test type: Superiority; p = 0.7245, Exact methods for risk difference; Risk difference = 0.10, 95% CI 2-sided [-0.74 to 1.51]
Statistical Analysis 8: Comparison: Tanezumab 5 mg vs NSAID; Primary osteonecrosis; Test type: Superiority; p = 0.7182, Exact methods for risk difference; Risk difference = 0.10, 95% CI 2-sided [-0.74 to 1.52]
Statistical Analysis 9: Comparison: Tanezumab 2.5 mg vs NSAID; Subchondral insufficiency fracture; Test type: Superiority; p = 0.6824, Exact methods for risk difference; Risk difference = 0.20, 95% CI 2-sided [-0.96 to 1.90]
Statistical Analysis 10: Comparison: Tanezumab 5 mg vs NSAID; Subchondral insufficiency fracture; Test type: Superiority; p = 0.5632, Exact methods for risk difference; Risk difference = 0.30, 95% CI 2-sided [-0.86 to 2.03]

9. Secondary Outcome: Observation Time-Adjusted Event Rate of Participants With Individual Adjudicated Joint Safety Outcome
Description: Observation time was defined as the start day of first SC study medication until either the (i) date of completion of or withdrawal from study, if a participant did not have the event, or (ii) date of the event (earliest event within each participant in the case of multiple events). Individual joint safety outcome included rapidly progressive OA (type-1 only), rapidly progressive OA (type-2 only), rapidly progressive OA (type-1 or type-2 combined), subchondral insufficiency fracture, primary osteonecrosis, and pathological fracture. Event rate was calculated as the number of events per 1000 participant-years at risk.
Time Frame: Baseline up to Week 80
Population: Safety population included all participants treated with tanezumab or placebo SC.
Measure: Number (95% Confidence Interval); unit: events per 1000 participant-years
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
events per 1000 participant-years
  Rapidly Progressive OA Type 1 or 2 | 31.4 [22.2 to 44.4] | 63.3 [49.5 to 81.1] | 11.9 [6.7 to 20.9]
  Rapidly Progressive OA Type 1 | 28.4 [19.8 to 40.9] | 49.1 [37.1 to 65.0] | 10.9 [6.0 to 19.6]
  Rapidly Progressive OA Type 2 | 2.9 [0.9 to 9.1] | 13.9 [8.2 to 23.4] | 1.0 [0.1 to 7.0]
  Primary Osteonecrosis | 1.0 [0.1 to 6.9] | 1.0 [0.1 to 7.0] | 0 [NA to NA] — 95% CI was not estimable since no participants had events.
  Pathological Fracture | 0 [NA to NA] — 95% CI was not estimable since no participants had events. | 0 [NA to NA] — 95% CI was not estimable since no participants had events. | 0 [NA to NA] — 95% CI was not estimable since no participants had events.
  Subchondral Insufficiency Fracture | 5.8 [2.6 to 13.0] | 6.9 [3.3 to 14.5] | 3.9 [1.5 to 10.5]
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Rapidly Progressive OA Type 1 or 2; Test type: Superiority; p = 0.0027, Poisson model for rate difference; Rate Difference = 19.56, 95% CI 2-sided [6.78 to 32.35]
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; Rapidly Progressive OA Type 1 or 2; Test type: Superiority; p < 0.0001, Poisson model for rate difference; Rate Difference = 51.48, 95% CI 2-sided [34.47 to 68.50]
Statistical Analysis 3: Comparison: Tanezumab 2.5 mg vs NSAID; Rapidly Progressive OA Type 1; Test type: Superiority; p = 0.0047, Poisson model for rate difference; Rate Difference = 17.58, 95% CI 2-sided [5.39 to 29.76]
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs NSAID; Rapidly Progressive OA Type 1; Test type: Superiority; p < 0.0001, Poisson model for rate difference; Rate Difference = 38.22, 95% CI 2-sided [23.05 to 53.40]
Statistical Analysis 5: Comparison: Tanezumab 2.5 mg vs NSAID; Rapidly Progressive OA Type 2; Test type: Superiority; p = 0.3214, Poisson model for rate difference; Rate Difference = 1.94, 95% CI 2-sided [-1.89 to 5.76]
Statistical Analysis 6: Comparison: Tanezumab 5 mg vs NSAID; Rapidly Progressive OA Type 2; Test type: Superiority; p = 0.0008, Poisson model for rate difference; Rate Difference = 12.88, 95% CI 2-sided [5.36 to 20.39]
Statistical Analysis 7: Comparison: Tanezumab 2.5 mg vs NSAID; Subchondral Insufficiency Fracture; Test type: Superiority; p = 0.5394, Poisson model for rate difference; Rate Difference = 1.90, 95% CI 2-sided [-4.17 to 7.96]
Statistical Analysis 8: Comparison: Tanezumab 5 mg vs NSAID; Subchondral Insufficiency Fracture; Test type: Superiority; p = 0.3636, Poisson model for rate difference; Rate Difference = 2.98, 95% CI 2-sided [-3.44 to 9.39]
Statistical Analysis 9: Comparison: Tanezumab 2.5 mg vs NSAID; Primary osteonecrosis; Test type: Superiority; Poisson model for rate difference = 1.0 — 95% CI was not estimable since there were less number of participants with events
Statistical Analysis 10: Comparison: Tanezumab 5 mg vs NSAID; Primary osteonecrosis; Test type: Superiority; Rate Difference = 1.0 — 95% CI was not estimable since there were less number of participants with events

10. Secondary Outcome: Percentage of Participants With Total Joint Replacement or Adjudicated Primary Composite Joint Safety Outcome
Description: Percentage of participants with total joint replacement (hip, knee or shoulder) or adjudicated primary composite joint safety outcomes were reported. Adjudicated primary composite joint safety outcomes included primary osteonecrosis, rapidly progressive OA type 1 or type 2, subchondral insufficiency fracture, or pathological fracture.
Time Frame: Baseline up to Week 80
Population: Safety population included all participants treated with tanezumab or placebo SC.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
percentage of participants | 8.6 [6.9 to 10.5] | 13.1 [11.1 to 15.4] | 3.7 [2.6 to 5.1]
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Test type: Superiority; p = 0.0002, Exact methods for risk difference — The event of adjudicated primary osteonecrosis in the tanezumab 2.5 mg treatment group is not included in this analysis. Conclusions for this analysis do not change as the comparison to NSAID is already statistically significant in favor of NSAID; Risk Difference (RD) = 4.87, 95% CI 2-sided [2.43 to 7.74]
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; Test type: Superiority; p < 0.0001, Exact methods for risk difference; Risk Difference (RD) = 9.41, 95% CI 2-sided [6.73 to 12.52]

11. Secondary Outcome: Observation Time-Adjusted Event Rate of Participants With Total Joint Replacement or Adjudicated Primary Composite Joint Safety Outcome
Description: Observation time was defined as the start day of first SC study medication until either the (i) date of completion of or withdrawal from study, if a participant did not have the event, or (ii) date of the event (earliest event within each participant in the case of multiple events). Adjudicated primary composite joint safety outcomes included primary osteonecrosis, rapidly progressive OA type 1 or type 2, subchondral insufficiency fracture, or pathological fracture. Event rate was calculated as the number of events per 1000 participant-years at risk.
Time Frame: Baseline up to Week 80
Population: Safety population included all participants treated with tanezumab or placebo SC.
Measure: Number (95% Confidence Interval); unit: events per 1000 participant-years
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
events per 1000 participant-years | 84.9 [68.7 to 104.9] | 132.5 [111.7 to 157.3] | 36.7 [26.6 to 50.6]
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Test type: Superiority; p < 0.0001, Poisson model for rate difference — [p-value comment as in outcome 10, analysis 1]; Rate Difference = 48.25, 95% CI 2-sided [26.76 to 69.74]
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; Test type: Superiority; p < 0.0001, Poisson model for rate difference; Rate Difference = 95.83, 95% CI 2-sided [70.25 to 121.42]

12. Secondary Outcome: Change From Baseline in Medial or Lateral Joint Space Width of the Index Knee (Kellgren-Lawrence Grade 2 or 3) at Weeks 56 and 80
Description: Change from baseline in JSW was defined as change in JSW compared to baseline in participants with Kellgren-Lawrence grade 2 or 3 over the course of the study. It was measured radiographically in the medial and lateral tibiofemoral of knee in participants with OA. Kellgren-Lawrence grade system was a method of classifying the severity of knee OA using five grades i.e. 0 [no radiographic features of OA], 1 [doubtful joint space narrowing (JSN) and possible osteophytic lipping], 2 [definite osteophytes and possible JSN on anteroposterior weight-bearing radiograph], 3 [multiple osteophytes, definite JSN, sclerosis, possible bony deformity], 4 [large osteophytes, marked JSN, severe sclerosis and definite bony deformity]. Higher grade indicating worse knee function. The number of participants with progression of OA in the index knee are summarized separately by the compartment of OA at baseline (medial or lateral).
Time Frame: Baseline, Weeks 56 and 80
Population: Safety population included all participants treated with tanezumab or placebo SC. Here "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure, and "Number analyzed" signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Least Squares Mean (Standard Error); unit: millimeter
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 651 | 668 | 695
millimeter
  Change in Medial JSW at Week 56: number analyzed (Participants) | 486 | 506 | 523
  Change in Medial JSW at Week 56 | -0.25 (0.03) | -0.34 (0.03) | -0.19 (0.03)
  Change in Medial JSW at Week 80: number analyzed (Participants) | 402 | 413 | 432
  Change in Medial JSW at Week 80 | -0.33 (0.04) | -0.37 (0.04) | -0.25 (0.03)
  Change in Lateral JSW at Week 56: number analyzed (Participants) | 110 | 94 | 114
  Change in Lateral JSW at Week 56 | -0.26 (0.07) | -0.32 (0.07) | -0.27 (0.07)
  Change in Lateral JSW at Week 80: number analyzed (Participants) | 88 | 75 | 98
  Change in Lateral JSW at Week 80 | -0.46 (0.08) | -0.32 (0.09) | -0.37 (0.08)
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Change in medial JSW width at Week 56: ANCOVA model included treatment, baseline JSW as covariate, and study site as a random effect; Test type: Superiority; p = 0.0979, ANCOVA; LS Mean Difference = -0.07, 95% CI 2-sided [-0.15 to 0.01], Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; Change in medial JSW at Week 56: ANCOVA model included treatment, baseline JSW as covariate, and study site as a random effect; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -0.16, 95% CI 2-sided [-0.24 to -0.08], Standard Error of Mean 0.04
Statistical Analysis 3: Comparison: Tanezumab 2.5 mg vs NSAID; Change in medial JSW at Week 80: ANCOVA model included treatment, baseline JSW as covariate, and study site as a random effect; Test type: Superiority; p = 0.1162, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-0.17 to 0.02], Standard Error of Mean 0.05
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 12, analysis 3]; Test type: Superiority; p = 0.0128, ANCOVA; LS Mean Difference = -0.12, 95% CI 2-sided [-0.22 to -0.03], Standard Error of Mean 0.05
Statistical Analysis 5: Comparison: Tanezumab 2.5 mg vs NSAID; Change in lateral JSW at Week 56: ANCOVA model included treatment, baseline JSW as covariate, and study site as a random effect; Test type: Superiority; p = 0.8885, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-0.17 to 0.20], Standard Error of Mean 0.09
Statistical Analysis 6: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 12, analysis 5]; Test type: Superiority; p = 0.6345, ANCOVA; LS Mean Difference = -0.05, 95% CI 2-sided [-0.24 to 0.15], Standard Error of Mean 0.10
Statistical Analysis 7: Comparison: Tanezumab 2.5 mg vs NSAID; Change in lateral JSW at Week 80: ANCOVA model included treatment, baseline JSW as covariate, and study site as a random effect; Test type: Superiority; p = 0.4406, ANCOVA; LS Mean Difference = -0.09, 95% CI 2-sided [-0.32 to 0.14], Standard Error of Mean 0.12
Statistical Analysis 8: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 12, analysis 7]; Test type: Superiority; p = 0.7109, ANCOVA; LS Mean Difference = 0.05, 95% CI 2-sided [-0.19 to 0.28], Standard Error of Mean 0.12

13. Secondary Outcome: Change From Baseline in Joint Space Width of the Index Hip (Kellgren-Lawrence Grade 2 or 3) at Weeks 56 and 80
Description: Change from baseline in JSW was defined as narrowing in JSW compared to baseline in participants with Kellgren-Lawrence grade 2 or 3 over the course of the study. It was measured radiographically in the index hip in participants with OA. Kellgren-Lawrence grade system was a method of classifying the severity of hip OA using five grades i.e. 0 (no radiographic features of OA), 1 (doubtful JSN and possible osteophytic lipping), 2 (definite osteophytes and possible JSN on anteroposterior weight-bearing radiograph), 3 (multiple osteophytes, definite JSN, sclerosis, possible bony deformity), 4 (large osteophytes, marked JSN, severe sclerosis and definite bony deformity). Higher grade indicating worse hip function.
Time Frame: Baseline, Weeks 56 and 80
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: millimeter
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 123 | 132 | 120
millimeter
  Change at Week 56: number analyzed (Participants) | 110 | 112 | 107
  Change at Week 56 | -0.35 (0.06) | -0.40 (0.06) | -0.21 (0.06)
  Change at Week 80: number analyzed (Participants) | 89 | 89 | 86
  Change at Week 80 | -0.46 (0.07) | -0.35 (0.07) | -0.28 (0.07)
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Change at Week 56: ANCOVA model included treatment, baseline JSW as covariate, and study site as a random effect; Test type: Superiority; p = 0.1020, ANCOVA; LS Mean Difference = -0.14, 95% CI 2-sided [-0.30 to 0.03], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; Change at Week 56: ANCOVA model included treatment, baseline JSW as covariate, and study site as a random effect; Test type: Superiority; p = 0.0230, ANCOVA; LS Mean Difference = -0.19, 95% CI 2-sided [-0.35 to -0.03], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: Tanezumab 2.5 mg vs NSAID; Change at Week 80: ANCOVA model included treatment, baseline JSW as covariate, and study site as a random effect; Test type: Superiority; p = 0.0645, ANCOVA; LS Mean Difference = -0.18, 95% CI 2-sided [-0.37 to 0.01], Standard Error of Mean 0.10
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs NSAID; Change at Week 80: ANCOVA model included treatment, baseline JSW as covariate, and study site as a random effect; Test type: Superiority; p = 0.5005, ANCOVA; LS Mean Difference = -0.07, 95% CI 2-sided [-0.26 to 0.13], Standard Error of Mean 0.10

14. Secondary Outcome: Number of Participants With Progression of Osteoarthritis in the Index Knee (Kellgren-Lawrence Grade 2 or 3) According to Bland and Altman Method at Weeks 56 and 80
Description: Progression of OA according to Bland-Altman as defined by a decrease JSW >=1.96 times within-participant standard deviation of change in JSW. The number of participants with progression of OA in the index knee are summarized separately by the compartment of OA at baseline (medial or lateral). Kellgren-Lawrence grade system was a method of classifying the severity of knee OA using five grades i.e. 0 [no radiographic features of OA], 1 [doubtful joint space narrowing (JSN) and possible osteophytic lipping], 2 [definite osteophytes and possible JSN on anteroposterior weight-bearing radiograph], 3 [multiple osteophytes, definite JSN, sclerosis, possible bony deformity], 4 [large osteophytes, marked JSN, severe sclerosis and definite bony deformity]. Higher grade indicating worse knee function.
Time Frame: Weeks 56 and 80
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 651 | 668 | 695
Participants
  Decreased medial JSW at Week 56: number analyzed (Participants) | 486 | 506 | 523
  Decreased medial JSW at Week 56 | 33 | 43 | 20
  Decreased medial JSW at Week 80: number analyzed (Participants) | 402 | 413 | 432
  Decreased medial JSW at Week 80 | 29 | 38 | 16
  Decreased lateral JSW at Week 56: number analyzed (Participants) | 110 | 94 | 114
  Decreased lateral JSW at Week 56 | 5 | 8 | 9
  Decreased lateral JSW at Week 80: number analyzed (Participants) | 88 | 75 | 98
  Decreased lateral JSW at Week 80 | 9 | 4 | 7
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Decrease in medial JSW at Week 56: Logistic regression model included treatment, and baseline JSW as covariate; Test type: Superiority; p = 0.0358, Regression, Logistic; Odds Ratio (OR) = 1.85, 95% CI 2-sided [1.04 to 3.29]
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; Decrease in medial JSW at Week 56: Logistic regression model included treatment, and baseline JSW as covariate; Test type: Superiority; p = 0.0021, Regression, Logistic; Odds Ratio (OR) = 2.37, 95% CI 2-sided [1.37 to 4.12]
Statistical Analysis 3: Comparison: Tanezumab 2.5 mg vs NSAID; Decrease in medial JSW at Week 80: Logistic regression model included treatment, and baseline JSW as covariate; Test type: Superiority; p = 0.0301, Regression, Logistic; Odds Ratio (OR) = 2.01, 95% CI 2-sided [1.07 to 3.77]
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs NSAID; Decrease in medial JSW at Week 80: Logistic regression model included treatment, and baseline JSW as covariate; Test type: Superiority; p = 0.0016, Regression, Logistic; Odds Ratio (OR) = 2.65, 95% CI 2-sided [1.45 to 4.85]
Statistical Analysis 5: Comparison: Tanezumab 2.5 mg vs NSAID; Decrease in lateral JSW at Week 56: Logistic regression model included treatment, and baseline JSW as covariate; Test type: Superiority; p = 0.3002, Regression, Logistic; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.18 to 1.70]
Statistical Analysis 6: Comparison: Tanezumab 5 mg vs NSAID; Decrease in lateral JSW at Week 56: Logistic regression model included treatment, and baseline JSW as covariate; Test type: Superiority; p = 0.8997, Regression, Logistic; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.39 to 2.89]
Statistical Analysis 7: Comparison: Tanezumab 2.5 mg vs NSAID; Decrease in lateral JSW at Week 80: Logistic regression model included treatment, and baseline JSW as covariate; Test type: Superiority; p = 0.4559, Regression, Logistic; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.53 to 4.18]
Statistical Analysis 8: Comparison: Tanezumab 5 mg vs NSAID; Decrease in lateral JSW at Week 80: Logistic regression model included treatment, and baseline JSW as covariate; Test type: Superiority; p = 0.5996, Regression, Logistic; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.20 to 2.54]

15. Secondary Outcome: Number of Participants With Progression of Osteoarthritis in the Index Hip (Kellgren-Lawrence Grade 2 or 3) According to Bland and Altman Method at Weeks 56 and 80
Description: Progression of OA according to Bland-Altman methodology as defined by a decrease in JSW >=1.96 times within-participant standard deviation of the change in JSW in the index hip. The number of participants with progression of OA in the index hip per Bland-Altman methodology are reported. Kellgren-Lawrence grade system was a method of classifying the severity of hip OA using five grades i.e. 0 (no radiographic features of OA), 1 (doubtful JSN and possible osteophytic lipping), 2 (definite osteophytes and possible JSN on anteroposterior weight-bearing radiograph), 3 (multiple osteophytes, definite JSN, sclerosis, possible bony deformity), 4 (large osteophytes, marked JSN, severe sclerosis and definite bony deformity). Higher grade indicating worse hip function.
Time Frame: Weeks 56 and 80
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 123 | 132 | 120
Participants
  Week 56: number analyzed (Participants) | 110 | 112 | 107
  Week 56 | 10 | 10 | 3
  Week 80: number analyzed (Participants) | 89 | 89 | 86
  Week 80 | 9 | 9 | 3
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Decrease at Week 56: Logistic regression model included treatment, and baseline JSW as covariate; Test type: Superiority; p = 0.0714, Regression, Logistic; Odds Ratio (OR) = 3.37, 95% CI 2-sided [0.90 to 12.65]
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; Decrease at Week 56: Logistic regression model included treatment, and baseline JSW as covariate; Test type: Superiority; p = 0.0681, Regression, Logistic; Odds Ratio (OR) = 3.42, 95% CI 2-sided [0.91 to 12.84]
Statistical Analysis 3: Comparison: Tanezumab 2.5 mg vs NSAID; Decrease at Week 80: Logistic regression model included treatment, and baseline JSW as covariate; Test type: Superiority; p = 0.0967, Regression, Logistic; Odds Ratio (OR) = 3.12, 95% CI 2-sided [0.81 to 11.95]
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs NSAID; Decrease at Week 80: Logistic regression model included treatment, and baseline JSW as covariate; Test type: Superiority; p = 0.0976, Regression, Logistic; Odds Ratio (OR) = 3.11, 95% CI 2-sided [0.81 to 11.90]

16. Secondary Outcome: Change From Baseline in WOMAC Pain Subscale at Weeks 2, 4, 8, 24, 32, 40, 48 and 56
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA. The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to OA of index joint (knee or hip) during past 48 hours. It was calculated as the mean of scores from 5 individual questions scored on a NRS, which may not be a whole (integer) number. Scores for each question and WOMAC Pain subscale score on NRS ranged from 0 (no pain) to 10 (extreme pain), where higher scores indicated higher pain.
Time Frame: Baseline, Weeks 2, 4, 8, 24, 32, 40, 48 and 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
units on scale
  Change at Week 2 | -1.65 (0.08) | -1.49 (0.08) | -1.55 (0.08)
  Change at Week 4 | -2.25 (0.09) | -2.29 (0.09) | -1.98 (0.09)
  Change at Week 8 | -2.41 (0.10) | -2.65 (0.10) | -2.27 (0.10)
  Change at Week 24 | -2.73 (0.13) | -2.86 (0.13) | -2.67 (0.13)
  Change at Week 32 | -2.64 (0.13) | -2.68 (0.13) | -2.57 (0.13)
  Change at Week 40 | -2.56 (0.13) | -2.57 (0.13) | -2.52 (0.13)
  Change at Week 48 | -2.54 (0.13) | -2.48 (0.13) | -2.47 (0.13)
  Change at Week 56 | -2.44 (0.13) | -2.37 (0.13) | -2.42 (0.14)
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Change at Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC pain subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.2212, ANCOVA; LS Mean Difference = -0.10, 95% CI 2-sided [-0.27 to 0.06], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; p = 0.4557, ANCOVA; LS Mean Difference = 0.06, 95% CI 2-sided [-0.10 to 0.23], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: Tanezumab 2.5 mg vs NSAID; Change at Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC pain subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0029, ANCOVA; LS Mean Difference = -0.27, 95% CI 2-sided [-0.45 to -0.09], Standard Error of Mean 0.09
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 16, analysis 3]; Test type: Superiority; p = 0.0005, ANCOVA; LS Mean Difference = -0.32, 95% CI 2-sided [-0.50 to -0.14], Standard Error of Mean 0.09
Statistical Analysis 5: Comparison: Tanezumab 2.5 mg vs NSAID; Change at Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC pain subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.1273, ANCOVA; LS Mean Difference = -0.14, 95% CI 2-sided [-0.33 to 0.04], Standard Error of Mean 0.09
Statistical Analysis 6: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 16, analysis 5]; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -0.38, 95% CI 2-sided [-0.57 to -0.20], Standard Error of Mean 0.09
Statistical Analysis 7: Comparison: Tanezumab 2.5 mg vs NSAID; Change at Week 24: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC pain subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.6349, ANCOVA; LS Mean Difference = -0.06, 95% CI 2-sided [-0.31 to 0.19], Standard Error of Mean 0.13
Statistical Analysis 8: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 16, analysis 7]; Test type: Superiority; p = 0.1339, ANCOVA; LS Mean Difference = -0.19, 95% CI 2-sided [-0.44 to 0.06], Standard Error of Mean 0.13
Statistical Analysis 9: Comparison: Tanezumab 2.5 mg vs NSAID; Change at Week 32: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC pain subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.6237, ANCOVA; LS Mean Difference = -0.07, 95% CI 2-sided [-0.33 to 0.20], Standard Error of Mean 0.13
Statistical Analysis 10: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 16, analysis 9]; Test type: Superiority; p = 0.4224, ANCOVA; LS Mean Difference = -0.11, 95% CI 2-sided [-0.37 to 0.16], Standard Error of Mean 0.13
Statistical Analysis 11: Comparison: Tanezumab 2.5 mg vs NSAID; Change at Week 40: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC pain subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.7526, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.31 to 0.22], Standard Error of Mean 0.14
Statistical Analysis 12: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 16, analysis 11]; Test type: Superiority; p = 0.7328, ANCOVA; LS Mean Difference = -0.05, 95% CI 2-sided [-0.31 to 0.22], Standard Error of Mean 0.13
Statistical Analysis 13: Comparison: Tanezumab 2.5 mg vs NSAID; Change at Week 48: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC pain subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.5888, ANCOVA; LS Mean Difference = -0.07, 95% CI 2-sided [-0.33 to 0.19], Standard Error of Mean 0.13
Statistical Analysis 14: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 16, analysis 13]; Test type: Superiority; p = 0.9345, ANCOVA; LS Mean Difference = -0.01, 95% CI 2-sided [-0.28 to 0.26], Standard Error of Mean 0.14
Statistical Analysis 15: Comparison: Tanezumab 2.5 mg vs NSAID; Change at Week 56: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC pain subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.8782, ANCOVA; LS Mean Difference = -0.02, 95% CI 2-sided [-0.29 to 0.25], Standard Error of Mean 0.14
Statistical Analysis 16: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 16, analysis 15]; Test type: Superiority; p = 0.7076, ANCOVA; LS Mean Difference = 0.05, 95% CI 2-sided [-0.22 to 0.32], Standard Error of Mean 0.14

17. Secondary Outcome: Change From Baseline in WOMAC Pain Subscale at Week 64
Description: as for outcome 16
Time Frame: Baseline, Week 64
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either Tanezumab or matching placebo). Here, "Number analyzed" =participants who were evaluable at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
units on a scale
  Baseline: number analyzed (Participants) | 1000 | 995 | 994
  Baseline | 7.01 (1.12) | 7.02 (1.12) | 6.96 (1.08)
  Change at Week 64: number analyzed (Participants) | 437 | 419 | 445
  Change at Week 64 | -3.47 (2.45) | -3.12 (2.40) | -3.85 (2.07)

18. Secondary Outcome: Change From Baseline in WOMAC Physical Function Subscale at Weeks 2, 4, 8, 24, 32, 40, 48 and 56
Description: as for outcome 4
Time Frame: Baseline, Weeks 2, 4, 8, 24, 32, 40, 48 and 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
units on a scale
  Change at Week 2 | -1.76 (0.08) | -1.64 (0.08) | -1.55 (0.08)
  Change at Week 4 | -2.29 (0.09) | -2.31 (0.09) | -1.96 (0.09)
  Change at Week 8 | -2.46 (0.10) | -2.69 (0.10) | -2.27 (0.10)
  Change at Week 24 | -2.78 (0.13) | -2.88 (0.13) | -2.66 (0.13)
  Change at Week 32 | -2.66 (0.13) | -2.67 (0.13) | -2.55 (0.13)
  Change at Week 40 | -2.56 (0.13) | -2.57 (0.13) | -2.50 (0.13)
  Change at Week 48 | -2.56 (0.14) | -2.49 (0.13) | -2.45 (0.13)
  Change at Week 56 | -2.45 (0.14) | -2.36 (0.13) | -2.41 (0.14)
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Change at Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC physical function subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0150, ANCOVA; LS Mean Difference = -0.21, 95% CI 2-sided [-0.37 to -0.04], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 18, analysis 1]; Test type: Superiority; p = 0.3286, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-0.25 to 0.08], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: Tanezumab 2.5 mg vs NSAID; Change at Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC physical function subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0004, ANCOVA; LS Mean Difference = -0.32, 95% CI 2-sided [-0.50 to -0.15], Standard Error of Mean 0.09
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 18, analysis 3]; Test type: Superiority; p = 0.0001, ANCOVA; LS Mean Difference = -0.35, 95% CI 2-sided [-0.53 to -0.17], Standard Error of Mean 0.09
Statistical Analysis 5: Comparison: Tanezumab 2.5 mg vs NSAID; Change at Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC physical function subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0517, ANCOVA; LS Mean Difference = -0.18, 95% CI 2-sided [-0.37 to 0.00], Standard Error of Mean 0.09
Statistical Analysis 6: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 18, analysis 5]; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -0.42, 95% CI 2-sided [-0.61 to -0.23], Standard Error of Mean 0.09
Statistical Analysis 7: Comparison: Tanezumab 2.5 mg vs NSAID; Change at Week 24: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC physical function subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.3621, ANCOVA; LS Mean Difference = -0.12, 95% CI 2-sided [-0.37 to 0.13], Standard Error of Mean 0.13
Statistical Analysis 8: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 18, analysis 7]; Test type: Superiority; p = 0.0832, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-0.47 to 0.03], Standard Error of Mean 0.13
Statistical Analysis 9: Comparison: Tanezumab 2.5 mg vs NSAID; Change at Week 32: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC physical function subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.4072, ANCOVA; LS Mean Difference = -0.11, 95% CI 2-sided [-0.38 to 0.15], Standard Error of Mean 0.13
Statistical Analysis 10: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 18, analysis 9]; Test type: Superiority; p = 0.3404, ANCOVA; LS Mean Difference = -0.13, 95% CI 2-sided [-0.39 to 0.13], Standard Error of Mean 0.13
Statistical Analysis 11: Comparison: Tanezumab 2.5 mg vs NSAID; Change at Week 40: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC physical function subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.6344, ANCOVA; LS Mean Difference = -0.07, 95% CI 2-sided [-0.34 to 0.20], Standard Error of Mean 0.14
Statistical Analysis 12: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 18, analysis 11]; Test type: Superiority; p = 0.5756, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-0.35 to 0.19], Standard Error of Mean 0.14
Statistical Analysis 13: Comparison: Tanezumab 2.5 mg vs NSAID; Change at Week 48: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC physical function subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.4394, ANCOVA; LS Mean Difference = -0.11, 95% CI 2-sided [-0.38 to 0.16], Standard Error of Mean 0.14
Statistical Analysis 14: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 18, analysis 13]; Test type: Superiority; p = 0.7747, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.31 to 0.23], Standard Error of Mean 0.14
Statistical Analysis 15: Comparison: Tanezumab 2.5 mg vs NSAID; Change at Week 56: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC physical function subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.7305, ANCOVA; LS Mean Difference = -0.05, 95% CI 2-sided [-0.32 to 0.22], Standard Error of Mean 0.14
Statistical Analysis 16: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 18, analysis 15]; Test type: Superiority; p = 0.7330, ANCOVA; LS Mean Difference = 0.05, 95% CI 2-sided [-0.22 to 0.32], Standard Error of Mean 0.14

19. Secondary Outcome: Change From Baseline in WOMAC Physical Function Subscale at Week 64
Description: as for outcome 4
Time Frame: Baseline, Week 64
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
units on a scale
  Baseline: number analyzed (Participants) | 1000 | 995 | 994
  Baseline | 7.09 (1.07) | 7.08 (1.11) | 6.99 (1.09)
  Change at Week 64: number analyzed (Participants) | 437 | 419 | 445
  Change at Week 64 | -3.42 (2.40) | -3.12 (2.41) | -3.81 (2.12)

20. Secondary Outcome: Change From Baseline in Patient's Global Assessment (PGA) of Osteoarthritis at Weeks 2, 4, 8, 24, 32, 40, 48 and 56
Description: PGA of OA was assessed by asking a question from participants: "Considering all the ways your OA in your knee or hip (index joint) affects you, how are you doing today?" Participants responded on a scale ranging from 1-5, using IRT, where 1=very good (no symptom and no limitation of normal activities), 2= good (mild symptoms and no limitation of normal activities), 3= fair (moderate symptoms and limitation of some normal activities), 4= poor (severe symptoms and inability to carry out most normal activities), and 5= very poor (very severe symptoms and inability to carry out all normal activities). Higher scores indicated worsening of condition.
Time Frame: Baseline, Weeks 2, 4, 8, 24, 32, 40, 48 and 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
units on a scale
  Change at Week 2 | -0.67 (0.03) | -0.67 (0.03) | -0.63 (0.03)
  Change at Week 4 | -0.81 (0.03) | -0.84 (0.03) | -0.69 (0.03)
  Change at Week 8 | -0.77 (0.03) | -0.85 (0.03) | -0.76 (0.03)
  Change at Week 24 | -0.74 (0.05) | -0.79 (0.05) | -0.74 (0.05)
  Change at Week 32 | -0.72 (0.05) | -0.71 (0.05) | -0.72 (0.05)
  Change at Week 40 | -0.70 (0.05) | -0.69 (0.05) | -0.69 (0.05)
  Change at Week 48 | -0.70 (0.05) | -0.66 (0.05) | -0.67 (0.05)
  Change at Week 56 | -0.65 (0.05) | -0.60 (0.05) | -0.66 (0.05)
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Change at Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline PGA and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.2159, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.10 to 0.02], Standard Error of Mean 0.03
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.2049, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.10 to 0.02], Standard Error of Mean 0.03
Statistical Analysis 3: Comparison: Tanezumab 2.5 mg vs NSAID; Change at Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline PGA and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0002, ANCOVA; LS Mean Difference = -0.12, 95% CI 2-sided [-0.19 to -0.06], Standard Error of Mean 0.03
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 20, analysis 3]; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -0.15, 95% CI 2-sided [-0.21 to -0.08], Standard Error of Mean 0.03
Statistical Analysis 5: Comparison: Tanezumab 2.5 mg vs NSAID; Change at Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline PGA and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.7799, ANCOVA; LS Mean Difference = -0.01, 95% CI 2-sided [-0.08 to 0.06], Standard Error of Mean 0.03
Statistical Analysis 6: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 20, analysis 5]; Test type: Superiority; p = 0.0061, ANCOVA; LS Mean Difference = -0.09, 95% CI 2-sided [-0.16 to -0.03], Standard Error of Mean 0.03
Statistical Analysis 7: Comparison: Tanezumab 2.5 mg vs NSAID; Change at Week 24: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline PGA and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.9718, ANCOVA; LS Mean Difference = -0.00, 95% CI 2-sided [-0.10 to 0.10], Standard Error of Mean 0.05
Statistical Analysis 8: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 20, analysis 7]; Test type: Superiority; p = 0.3292, ANCOVA; LS Mean Difference = -0.05, 95% CI 2-sided [-0.14 to 0.05], Standard Error of Mean 0.05
Statistical Analysis 9: Comparison: Tanezumab 2.5 mg vs NSAID; Change at Week 32: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline PGA and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.9830, ANCOVA; LS Mean Difference = 0.00, 95% CI 2-sided [-0.10 to 0.10], Standard Error of Mean 0.05
Statistical Analysis 10: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 20, analysis 9]; Test type: Superiority; p = 0.9137, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-0.09 to 0.11], Standard Error of Mean 0.05
Statistical Analysis 11: Comparison: Tanezumab 2.5 mg vs NSAID; Change at Week 40: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline PGA and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.8784, ANCOVA; LS Mean Difference = -0.01, 95% CI 2-sided [-0.11 to 0.09], Standard Error of Mean 0.05
Statistical Analysis 12: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 20, analysis 11]; Test type: Superiority; p = 0.9995, ANCOVA; LS Mean Difference = 0.00, 95% CI 2-sided [-0.10 to 0.10], Standard Error of Mean 0.05
Statistical Analysis 13: Comparison: Tanezumab 2.5 mg vs NSAID; Change at Week 48: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline PGA and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.6648, ANCOVA; LS Mean Difference = -0.02, 95% CI 2-sided [-0.13 to 0.08], Standard Error of Mean 0.05
Statistical Analysis 14: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 20, analysis 13]; Test type: Superiority; p = 0.7280, ANCOVA; LS Mean Difference = 0.02, 95% CI 2-sided [-0.09 to 0.12], Standard Error of Mean 0.05
Statistical Analysis 15: Comparison: Tanezumab 2.5 mg vs NSAID; Change at Week 56: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline PGA and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.8856, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-0.09 to 0.11], Standard Error of Mean 0.05
Statistical Analysis 16: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 20, analysis 15]; Test type: Superiority; p = 0.2814, ANCOVA; LS Mean Difference = 0.06, 95% CI 2-sided [-0.05 to 0.16], Standard Error of Mean 0.05

21. Secondary Outcome: Change From Baseline in Patient's Global Assessment (PGA) of Osteoarthritis at Week 64
Description: as for outcome 20
Time Frame: Baseline, Week 64
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
units on a scale
  Baseline: number analyzed (Participants) | 1000 | 995 | 994
  Baseline | 3.49 (0.61) | 3.46 (0.60) | 3.44 (0.59)
  Change at Week 64: number analyzed (Participants) | 437 | 419 | 445
  Change at Week 64 | -0.79 (0.96) | -0.64 (0.98) | -0.95 (0.96)

22. Secondary Outcome: Percentage of Participants Meeting Outcome Measures in Arthritis Clinical Trials-Osteoarthritis Research Society International (OMERACT-OARSI) Responder Index at Weeks 2, 4, 8, 16, 24, 32, 40, 48, 56 and 64
Description: Participants were considered as OMERACT-OARSI responders: if the change (improvement) from baseline to week of interest was >=50 percent and >= 2 units in either WOMAC pain subscale or physical function subscale score; if change (improvement) from baseline to week of interest was >=20 percent and >=1 unit in at least 2 of the following: 1) WOMAC pain subscale score, 2) WOMAC physical function subscale score, 3) PGA of OA. WOMAC pain subscale assess amount of pain experienced (score: 0 [no pain] to 10 [extreme pain], higher score = more pain), WOMAC physical function subscale assess degree of difficulty experienced (score: 0 [no difficulty] to 10 [extreme difficulty], higher score = worse physical function) and PGA of OA (score: 1 [very good] to 5 [very poor], higher score = worse condition). Missing data was imputed using mixed baseline/last observation carried forward (BOCF/LOCF).
Time Frame: Weeks 2, 4, 8, 16, 24, 32, 40, 48, 56 and 64
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or matching placebo). "Number analyzed"=participants who were evaluable for this outcome measure at specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
percentage of participants
  Week 2: number analyzed (Participants) | 1001 | 996 | 996
  Week 2 | 46.7 | 43.7 | 44.8
  Week 4: number analyzed (Participants) | 1001 | 996 | 996
  Week 4 | 62.6 | 62.7 | 56.4
  Week 8: number analyzed (Participants) | 1001 | 996 | 996
  Week 8 | 67.5 | 70.3 | 64.4
  Week 16: number analyzed (Participants) | 1001 | 996 | 996
  Week 16 | 78.2 | 78.3 | 75.1
  Week 24: number analyzed (Participants) | 1001 | 996 | 995
  Week 24 | 62.4 | 64.8 | 61.3
  Week 32: number analyzed (Participants) | 1001 | 996 | 995
  Week 32 | 59.2 | 59.9 | 58.6
  Week 40: number analyzed (Participants) | 1001 | 996 | 995
  Week 40 | 58.4 | 58.7 | 58.2
  Week 48: number analyzed (Participants) | 1001 | 996 | 995
  Week 48 | 57.4 | 56.2 | 57.3
  Week 56: number analyzed (Participants) | 1001 | 996 | 995
  Week 56 | 56.5 | 54.5 | 56.0
  Week 64: number analyzed (Participants) | 437 | 420 | 446
  Week 64 | 79.2 | 75.2 | 86.5
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Week 2; Test type: Superiority; p = 0.4691, Regression, Logistic; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.89 to 1.28] — OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade, NSAID and treatment
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; Week 2; Test type: Superiority; p = 0.5451, Regression, Logistic; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.79 to 1.13] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 3: Comparison: Tanezumab 2.5 mg vs NSAID; Week 4; Test type: Superiority; p = 0.0059, Regression, Logistic; Odds Ratio (OR) = 1.29, 95% CI 2-sided [1.08 to 1.54] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs NSAID; Week 4; Test type: Superiority; p = 0.0057, Regression, Logistic; Odds Ratio (OR) = 1.29, 95% CI 2-sided [1.08 to 1.55] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 5: Comparison: Tanezumab 2.5 mg vs NSAID; Week 8; Test type: Superiority; p = 0.1584, Regression, Logistic; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.95 to 1.38] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 6: Comparison: Tanezumab 5 mg vs NSAID; Week 8; Test type: Superiority; p = 0.0060, Regression, Logistic; Odds Ratio (OR) = 1.30, 95% CI [1.08 to 1.58] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 7: Comparison: Tanezumab 2.5 mg vs NSAID; Week 16; Test type: Superiority; p = 0.1117, Regression, Logistic; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.96 to 1.46] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 8: Comparison: Tanezumab 5 mg vs NSAID; Week 16; Test type: Superiority; p = 0.1004, Regression, Logistic; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.97 to 1.47] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 9: Comparison: Tanezumab 2.5 mg vs NSAID; Week 24; Test type: Superiority; p = 0.6258, Regression, Logistic; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.87 to 1.25] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 10: Comparison: Tanezumab 5 mg vs NSAID; Week 24; Test type: Superiority; p = 0.1154, Regression, Logistic; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.96 to 1.39] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 11: Comparison: Tanezumab 2.5 mg vs NSAID; Week 32; Test type: Superiority; p = 0.8018, Regression, Logistic; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.86 to 1.22] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 12: Comparison: Tanezumab 5 mg vs NSAID; Week 32; Test type: Superiority; p = 0.5697, Regression, Logistic; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.88 to 1.26] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 13: Comparison: Tanezumab 2.5 mg vs NSAID; Week 40; Test type: Superiority; p = 0.9557, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.84 to 1.20] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 14: Comparison: Tanezumab 5 mg vs NSAID; Week 40; Test type: Superiority; p = 0.8553, Regression, Logistic; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.85 to 1.22] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 15: Comparison: Tanezumab 2.5 mg vs NSAID; Week 48; Test type: Superiority; p = 0.9901, Regression, Logistic; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.84 to 1.20] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 16: Comparison: Tanezumab 5 mg vs NSAID; Week 48; Test type: Superiority; p = 0.5870, Regression, Logistic; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.80 to 1.14] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 17: Comparison: Tanezumab 2.5 mg vs NSAID; Week 56; Test type: Superiority; p = 0.8302, Regression, Logistic; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.85 to 1.22] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 18: Comparison: Tanezumab 5 mg vs NSAID; Week 56; Test type: Superiority; p = 0.4823, Regression, Logistic; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.79 to 1.12] — [estimate comment as in outcome 22, analysis 1]

23. Secondary Outcome: Percentage of Participants Achieving Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Reduction >=30 Percent (%), >=50%, >=70% and >=90% Response at Weeks 2, 4, 8, 16, 24, 32, 40, 48, 56 and 64
Description: Percentage of participants with reduction in WOMAC pain intensity of >= 30%, 50%, 70% and 90% at Weeks 2, 4, 8, 16, 24, 32, 40, 48, 56 and 64 compared to baseline were classified as responders to WOMAC pain subscale and are reported here. WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA. The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to OA of index joint (knee or hip) during past 48 hours. It was calculated as the mean of scores from 5 individual questions scored on a NRS. Scores for each question and WOMAC Pain subscale score on NRS ranged from 0 (no pain) to 10 (extreme pain), where higher scores indicated higher pain. Missing data was imputed using mixed BOCF/LOCF.
Time Frame: Weeks 2, 4, 8, 16, 24, 32, 40, 48, 56 and 64
Population: as for outcome 22
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
percentage of participants
  Week 2: At least 30% reduction | 34.8 | 30.5 | 32.4
  Week 2: At least 50% reduction | 17.8 | 16.5 | 14.7
  Week 2: At least 70% reduction | 7.7 | 7.1 | 6.2
  Week 2: At least 90% reduction | 2.4 | 2.5 | 1.8
  Week 4: At least 30% reduction | 50.2 | 49.5 | 44.4
  Week 4: At least 50% reduction | 30.4 | 30.5 | 24.9
  Week 4: At least 70% reduction | 14.5 | 16.4 | 11.9
  Week 4: At least 90% reduction | 4.3 | 4.9 | 3.1
  Week 8: At least 30% reduction | 55.9 | 59.0 | 54.1
  Week 8: At least 50% reduction | 36.8 | 39.3 | 32.6
  Week 8: At least 70% reduction | 19.3 | 22.4 | 15.9
  Week 8: At least 90% reduction | 4.7 | 6.6 | 4.2
  Week 16: At least 30% reduction | 71.8 | 72.9 | 68.9
  Week 16: At least 50% reduction | 54.9 | 56.5 | 51.5
  Week 16: At least 70% reduction | 28.9 | 35.0 | 28.8
  Week 16: At least 90% reduction | 10.3 | 12.7 | 8.5
  Week 24: At least 30% reduction | 59.4 | 61.1 | 59.4
  Week 24: At least 50% reduction | 49.3 | 49.4 | 47.5
  Week 24: At least 70% reduction | 30.8 | 33.8 | 29.0
  Week 24: At least 90% reduction | 10.3 | 13.3 | 11.5
  Week 32: At least 30% reduction | 56.8 | 55.7 | 56.3
  Week 32: At least 50% reduction | 47.4 | 45.8 | 46.3
  Week 32: At least 70% reduction | 31.2 | 31.5 | 27.4
  Week 32: At least 90% reduction | 10.3 | 12.9 | 10.0
  Week 40: At least 30% reduction | 55.7 | 54.6 | 54.8
  Week 40: At least 50% reduction | 47.2 | 45.2 | 46.0
  Week 40: At least 70% reduction | 30.0 | 30.4 | 29.3
  Week 40: At least 90% reduction | 10.8 | 12.0 | 10.4
  Week 48: At least 30% reduction | 54.6 | 52.9 | 54.2
  Week 48: At least 50% reduction | 46.2 | 43.2 | 44.4
  Week 48: At least 70% reduction | 29.6 | 29.4 | 28.5
  Week 48: At least 90% reduction | 10.3 | 11.4 | 10.6
  Week 56: At least 30% reduction | 53.1 | 51.2 | 52.7
  Week 56: At least 50% reduction | 44.3 | 41.5 | 43.5
  Week 56: At least 70% reduction | 28.2 | 27.0 | 27.5
  Week 56: At least 90% reduction | 10.1 | 10.5 | 10.1
  Week 64: At least 30% reduction: number analyzed (Participants) | 437 | 419 | 445
  Week 64: At least 30% reduction | 73.0 | 69.0 | 81.3
  Week 64: At least 50% reduction: number analyzed (Participants) | 437 | 419 | 445
  Week 64: At least 50% reduction | 55.4 | 47.3 | 60.2
  Week 64: At least 70% reduction: number analyzed (Participants) | 437 | 419 | 445
  Week 64: At least 70% reduction | 31.1 | 24.3 | 34.2
  Week 64: At least 90% reduction: number analyzed (Participants) | 437 | 419 | 445
  Week 64: At least 90% reduction | 9.6 | 7.9 | 12.6
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Week 2: >=30% reduction; Test type: Superiority; p = 0.2938, Regression, Logistic; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.92 to 1.33] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; Week 2: >=30% reduction; Test type: Superiority; p = 0.3146, Regression, Logistic; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.75 to 1.10] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 3: Comparison: Tanezumab 2.5 mg vs NSAID; Week 2: >=50% reduction; Test type: Superiority; p = 0.0748, Regression, Logistic; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.98 to 1.58] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs NSAID; Week 2: >=50% reduction; Test type: Superiority; p = 0.3000, Regression, Logistic; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.89 to 1.45] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 5: Comparison: Tanezumab 2.5 mg vs NSAID; Week 2: >=70% reduction; Test type: Superiority; p = 0.2550, Regression, Logistic; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.86 to 1.74] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 6: Comparison: Tanezumab 5 mg vs NSAID; Week 2: >=70% reduction; Test type: Superiority; p = 0.4780, Regression, Logistic; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.80 to 1.62] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 7: Comparison: Tanezumab 2.5 mg vs NSAID; Week 2: >=90% reduction; Test type: Superiority; p = 0.4006, Regression, Logistic; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.70 to 2.42] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 8: Comparison: Tanezumab 5 mg vs NSAID; Week 2: >=90% reduction; Test type: Superiority; p = 0.3089, Regression, Logistic; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.74 to 2.54] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 9: Comparison: Tanezumab 2.5 mg vs NSAID; Week 4: >=30% reduction; Test type: Superiority; p = 0.0114, Regression, Logistic; Odds Ratio (OR) = 1.26, 95% CI 2-sided [1.05 to 1.50] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 10: Comparison: Tanezumab 5 mg vs NSAID; Week 4: >=30% reduction; Test type: Superiority; p = 0.0239, Regression, Logistic; Odds Ratio (OR) = 1.23, 95% CI 2-sided [1.03 to 1.47] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 11: Comparison: Tanezumab 2.5 mg vs NSAID; Week 4: >=50% reduction; Test type: Superiority; p = 0.0079, Regression, Logistic; Odds Ratio (OR) = 1.31, 95% CI 2-sided [1.07 to 1.60] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 12: Comparison: Tanezumab 5 mg vs NSAID; Week 4: >=50% reduction; Test type: Superiority; p = 0.0068, Regression, Logistic; Odds Ratio (OR) = 1.32, 95% CI 2-sided [1.08 to 1.60] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 13: Comparison: Tanezumab 2.5 mg vs NSAID; Week 4: >=70% reduction; Test type: Superiority; p = 0.1037, Regression, Logistic; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.96 to 1.62] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 14: Comparison: Tanezumab 5 mg vs NSAID; Week 4: >=70% reduction; Test type: Superiority; p = 0.0046, Regression, Logistic; Odds Ratio (OR) = 1.45, 95% CI 2-sided [1.12 to 1.88] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 15: Comparison: Tanezumab 2.5 mg vs NSAID; Week 4: >=90% reduction; Test type: Superiority; p = 0.1971, Regression, Logistic; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.85 to 2.19] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 16: Comparison: Tanezumab 5 mg vs NSAID; Week 4: >=90% reduction; Test type: Superiority; p = 0.0480, Regression, Logistic; Odds Ratio (OR) = 1.59, 95% CI 2-sided [1.00 to 2.52] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 17: Comparison: Tanezumab 2.5 mg vs NSAID; Week 8: >=30% reduction; Test type: Superiority; p = 0.4744, Regression, Logistic; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.89 to 1.28] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 18: Comparison: Tanezumab 5 mg vs NSAID; Week 8: >=30% reduction; Test type: Superiority; p = 0.0336, Regression, Logistic; Odds Ratio (OR) = 1.21, 95% CI 2-sided [1.02 to 1.45] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 19: Comparison: Tanezumab 2.5 mg vs NSAID; Week 8: >=50% reduction; Test type: Superiority; p = 0.0559, Regression, Logistic; Odds Ratio (OR) = 1.20, 95% CI 2-sided [1.00 to 1.44] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 20: Comparison: Tanezumab 5 mg vs NSAID; Week 8: >=50% reduction; Test type: Superiority; p = 0.0021, Regression, Logistic; Odds Ratio (OR) = 1.34, 95% CI 2-sided [1.11 to 1.61] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 21: Comparison: Tanezumab 2.5 mg vs NSAID; Week 8: >=70% reduction; Test type: Superiority; p = 0.0535, Regression, Logistic; Odds Ratio (OR) = 1.26, 95% CI 2-sided [1.00 to 1.59] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 22: Comparison: Tanezumab 5 mg vs NSAID; Week 8: >=70% reduction; Test type: Superiority; p = 0.0003, Regression, Logistic; Odds Ratio (OR) = 1.53, 95% CI 2-sided [1.22 to 1.92] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 23: Comparison: Tanezumab 2.5 mg vs NSAID; Week 8: >=90% reduction; Test type: Superiority; p = 0.6421, Regression, Logistic; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.72 to 1.70] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 24: Comparison: Tanezumab 5 mg vs NSAID; Week 8: >=90% reduction; Test type: Superiority; p = 0.0207, Regression, Logistic; Odds Ratio (OR) = 1.60, 95% CI 2-sided [1.07 to 2.38] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 25: Comparison: Tanezumab 2.5 mg vs NSAID; Week 16: >=30% reduction; Test type: Superiority; p = 0.1635, Regression, Logistic; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.95 to 1.39] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 26: Comparison: Tanezumab 5 mg vs NSAID; Week 16: >=30% reduction; Test type: Superiority; p = 0.0529, Regression, Logistic; Odds Ratio (OR) = 1.21, 95% CI 2-sided [1.00 to 1.47] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 27: Comparison: Tanezumab 2.5 mg vs NSAID; Week 16: >=50% reduction; Test type: Superiority — The two key secondary comparisons for 'Participants with >=50% reduction from baseline in WOMAC Pain at Week 16' (tanezumab 2.5 mg treatment group versus NSAID and tanezumab 5 mg treatment group versus NSAID) could not be considered significant since preceding tests in the graphical testing procedure were not significant; p = 0.1322, Regression, Logistic; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.96 to 1.37] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 28: Comparison: Tanezumab 5 mg vs NSAID; Week 16: >=50% reduction; Test type: Superiority — [test comment as in outcome 23, analysis 27]; p = 0.0262, Regression, Logistic; Odds Ratio (OR) = 1.22, 95% CI 2-sided [1.02 to 1.46] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 29: Comparison: Tanezumab 2.5 mg vs NSAID; Week 16: >=70% reduction; Test type: Superiority; p = 0.9805, Regression, Logistic; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.83 to 1.22] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 30: Comparison: Tanezumab 5 mg vs NSAID; Week 16: >=70% reduction; Test type: Superiority; p = 0.0033, Regression, Logistic; Odds Ratio (OR) = 1.33, 95% CI 2-sided [1.10 to 1.61] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 31: Comparison: Tanezumab 2.5 mg vs NSAID; Week 16: >=90% reduction; Test type: Superiority; p = 0.1590, Regression, Logistic; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.92 to 1.69] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 32: Comparison: Tanezumab 5 mg vs NSAID; Week 16: >=90% reduction; Test type: Superiority; p = 0.0024, Regression, Logistic; Odds Ratio (OR) = 1.57, 95% CI 2-sided [1.17 to 2.11] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 33: Comparison: Tanezumab 2.5 mg vs NSAID; Week 24: >=30% reduction; Test type: Superiority; p = 0.9932, Regression, Logistic; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.83 to 1.20] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 34: Comparison: Tanezumab 5 mg vs NSAID; Week 24: >=30% reduction; Test type: Superiority; p = 0.4374, Regression, Logistic; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.90 to 1.29] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 35: Comparison: Tanezumab 2.5 mg vs NSAID; Week 24: >=50% reduction; Test type: Superiority; p = 0.4406, Regression, Logistic; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.90 to 1.28] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 36: Comparison: Tanezumab 5 mg vs NSAID; Week 24: >=50% reduction; Test type: Superiority; p = 0.4078, Regression, Logistic; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.90 to 1.29] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 37: Comparison: Tanezumab 2.5 mg vs NSAID; Week 24: >=70% reduction; Test type: Superiority; p = 0.4071, Regression, Logistic; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.89 to 1.31] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 38: Comparison: Tanezumab 5 mg vs NSAID; Week 24: >=70% reduction; Test type: Superiority; p = 0.0248, Regression, Logistic; Odds Ratio (OR) = 1.24, 95% CI 2-sided [1.03 to 1.50] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 39: Comparison: Tanezumab 2.5 mg vs NSAID; Week 24: >=90% reduction; Test type: Superiority; p = 0.3641, Regression, Logistic; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.66 to 1.16] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 40: Comparison: Tanezumab 5 mg vs NSAID; Week 24: >=90% reduction; Test type: Superiority; p = 0.2497, Regression, Logistic; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.89 to 1.53] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 41: Comparison: Tanezumab 2.5 mg vs NSAID; Week 32: >=30% reduction; Test type: Superiority; p = 0.8682, Regression, Logistic; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.85 to 1.21] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 42: Comparison: Tanezumab 5 mg vs NSAID; Week 32: >=30% reduction; Test type: Superiority; p = 0.7317, Regression, Logistic; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.81 to 1.16] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 43: Comparison: Tanezumab 2.5 mg vs NSAID; Week 32: >=50% reduction; Test type: Superiority; p = 0.6493, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.87 to 1.24] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 44: Comparison: Tanezumab 5 mg vs NSAID; Week 32: >=50% reduction; Test type: Superiority; p = 0.7973, Regression, Logistic; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.82 to 1.17] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 45: Comparison: Tanezumab 2.5 mg vs NSAID; Week 32: >=70% reduction; Test type: Superiority; p = 0.0757, Regression, Logistic; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.98 to 1.45] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 46: Comparison: Tanezumab 5 mg vs NSAID; Week 32: >=70% reduction; Test type: Superiority; p = 0.0578, Regression, Logistic; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.99 to 1.47] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 47: Comparison: Tanezumab 2.5 mg vs NSAID; Week 32: >=90% reduction; Test type: Superiority; p = 0.9010, Regression, Logistic; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.76 to 1.37] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 48: Comparison: Tanezumab 5 mg vs NSAID; Week 32: >=90% reduction; Test type: Superiority; p = 0.0548, Regression, Logistic; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.99 to 1.74] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 49: Comparison: Tanezumab 2.5 mg vs NSAID; Week 40: >=30% reduction; Test type: Superiority; p = 0.7331, Regression, Logistic; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.86 to 1.23] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 50: Comparison: Tanezumab 5 mg vs NSAID; Week 40: >=30% reduction; Test type: Superiority; p = 0.8632, Regression, Logistic; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.82 to 1.18] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 51: Comparison: Tanezumab 2.5 mg vs NSAID; Week 40: >=50% reduction; Test type: Superiority; p = 0.6262, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.88 to 1.25] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 52: Comparison: Tanezumab 5 mg vs NSAID; Week 40: >=50% reduction; Test type: Superiority; p = 0.6817, Regression, Logistic; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.81 to 1.15] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 53: Comparison: Tanezumab 2.5 mg vs NSAID; Week 40: >=70% reduction; Test type: Superiority; p = 0.7990, Regression, Logistic; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.85 to 1.24] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 54: Comparison: Tanezumab 5 mg vs NSAID; Week 40: >=70% reduction; Test type: Superiority; p = 0.6786, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.86 to 1.26] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 55: Comparison: Tanezumab 2.5 mg vs NSAID; Week 40: >=90% reduction; Test type: Superiority; p = 0.8069, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.78 to 1.38] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 56: Comparison: Tanezumab 5 mg vs NSAID; Week 40: >=90% reduction; Test type: Superiority; p = 0.2951, Regression, Logistic; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.88 to 1.54] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 57: Comparison: Tanezumab 2.5 mg vs NSAID; Week 48: >=30% reduction; Test type: Superiority; p = 0.9093, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.85 to 1.21] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 58: Comparison: Tanezumab 5 mg vs NSAID; Week 48: >=30% reduction; Test type: Superiority; p = 0.5032, Regression, Logistic; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.79 to 1.12] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 59: Comparison: Tanezumab 2.5 mg vs NSAID; Week 48: >=50% reduction; Test type: Superiority; p = 0.4382, Regression, Logistic; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.90 to 1.28] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 60: Comparison: Tanezumab 5 mg vs NSAID; Week 48: >=50% reduction; Test type: Superiority; p = 0.5638, Regression, Logistic; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.79 to 1.13] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 61: Comparison: Tanezumab 2.5 mg vs NSAID; Week 48: >=70% reduction; Test type: Superiority; p = 0.6436, Regression, Logistic; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.86 to 1.27] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 62: Comparison: Tanezumab 5 mg vs NSAID; Week 48: >=70% reduction; Test type: Superiority; p = 0.7060, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.85 to 1.26] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 63: Comparison: Tanezumab 2.5 mg vs NSAID; Week 48: >=90% reduction; Test type: Superiority; p = 0.7729, Regression, Logistic; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.72 to 1.28] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 64: Comparison: Tanezumab 5 mg vs NSAID; Week 48: >=90% reduction; Test type: Superiority; p = 0.6405, Regression, Logistic; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.81 to 1.42] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 65: Comparison: Tanezumab 2.5 mg vs NSAID; Week 56: >=30% reduction; Test type: Superiority; p = 0.9046, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.85 to 1.21] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 66: Comparison: Tanezumab 5 mg vs NSAID; Week 56: >=30% reduction; Test type: Superiority; p = 0.4491, Regression, Logistic; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.78 to 1.11] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 67: Comparison: Tanezumab 2.5 mg vs NSAID; Week 56: >=50% reduction; Test type: Superiority; p = 0.7429, Regression, Logistic; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.86 to 1.23] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 68: Comparison: Tanezumab 5 mg vs NSAID; Week 56: >=50% reduction; Test type: Superiority; p = 0.3467, Regression, Logistic; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.77 to 1.10] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 69: Comparison: Tanezumab 2.5 mg vs NSAID; Week 56: >=70% reduction; Test type: Superiority; p = 0.7624, Regression, Logistic; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.85 to 1.26] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 70: Comparison: Tanezumab 5 mg vs NSAID; Week 56: >=70% reduction; Test type: Superiority; p = 0.7686, Regression, Logistic; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.80 to 1.18] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 71: Comparison: Tanezumab 2.5 mg vs NSAID; Week 56: >=90% reduction; Test type: Superiority; p = 0.9384, Regression, Logistic; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.74 to 1.33] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 72: Comparison: Tanezumab 5 mg vs NSAID; Week 56: >=90% reduction; Test type: Superiority; p = 0.8495, Regression, Logistic; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.77 to 1.38] — [estimate comment as in outcome 22, analysis 1]

24. Secondary Outcome: Percentage of Participants With Cumulative Percent Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale at Weeks 16, 24 and 56
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA. The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to OA of index joint during past 48 hours. It was calculated as the mean of scores from 5 individual questions scored on a NRS. Scores for each question and WOMAC Pain subscale score on NRS ranged from 0 (no pain) to 10 (extreme pain), where higher scores indicated higher pain. Percentage of participants with cumulative reduction (as percent) (greater than [>] 0% ; >= 10, 20, 30, 40, 50, 60, 70, 80 and 90%; = 100 %) in WOMAC pain subscale from Baseline to Weeks 16, 24 and 56 were reported, participants (%) are reported more than once in categories specified. Missing data was imputed using mixed BOCF/LOCF.
Time Frame: Baseline, Weeks 16, 24 and 56
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or matching placebo). Here 'Overall number of participants analyzed' = participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1000 | 995 | 994
percentage of participants
  Week 16: >0% | 89.5 | 87.6 | 87.1
  Week 16: >=10% | 85.0 | 82.8 | 82.8
  Week 16: >=20% | 78.1 | 78.3 | 75.8
  Week 16: >=30% | 71.8 | 72.9 | 68.9
  Week 16: >=40% | 63.7 | 63.5 | 59.9
  Week 16: >=50% | 54.9 | 56.5 | 51.5
  Week 16: >=60% | 40.9 | 44.8 | 38.8
  Week 16: >=70% | 28.9 | 35.0 | 28.8
  Week 16: >=80% | 19.4 | 23.9 | 18.8
  Week 16: >=90% | 10.3 | 12.7 | 8.5
  Week 16: =100% | 4.4 | 3.9 | 3.3
  Week 24: >0% | 66.7 | 68.2 | 64.8
  Week 24: >=10% | 64.9 | 66.4 | 63.4
  Week 24: >=20% | 62.2 | 65.2 | 62.1
  Week 24: >=30% | 59.4 | 61.1 | 59.4
  Week 24: >=40% | 55.2 | 55.7 | 54.7
  Week 24: >=50% | 49.3 | 49.4 | 47.5
  Week 24: >=60% | 40.7 | 41.2 | 38.1
  Week 24: >=70% | 30.8 | 33.8 | 29.0
  Week 24: >=80% | 20.6 | 24.0 | 20.2
  Week 24: >=90% | 10.3 | 13.3 | 11.5
  Week 24: =100% | 3.9 | 4.5 | 3.4
  Week 56: >0% | 60.8 | 59.1 | 59.7
  Week 56: >=10% | 59.1 | 57.0 | 58.1
  Week 56: >=20% | 55.9 | 54.8 | 56.3
  Week 56: >=30% | 53.1 | 51.2 | 52.7
  Week 56: >=40% | 48.6 | 46.8 | 48.6
  Week 56: >=50% | 44.3 | 41.5 | 43.5
  Week 56: >=60% | 37.0 | 33.8 | 36.3
  Week 56: >=70% | 28.2 | 27.0 | 27.5
  Week 56: >=80% | 18.9 | 19.1 | 18.6
  Week 56: >=90% | 10.1 | 10.5 | 10.1
  Week 56: =100% | 4.5 | 5.3 | 4.1

25. Secondary Outcome: Percentage of Participants Achieving Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale Reduction of >=30%, >=50%, >=70% and >=90% Response at Weeks 2, 4, 8, 16, 24, 32, 40, 48, 56 and 64
Description: Percentage of participants with reduction in WOMAC physical function of >=(30%,50%,70%,90%) at Weeks 2,4,8,16,24,32,40,48,56 and 64 compared to baseline were classified as responders to WOMAC physical function subscale. WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA. Physical function:Participant's ability to move around and perform usual activities of daily living. WOMAC physical function subscale17-item questionnaire used to assess the degree of difficulty experienced due to OA in index joint (knee/hip) during past 48 hours, calculated as mean of the scores from 17 individual questions scored on a NRS. Scores for each question and WOMAC physical subscale on NRS ranged from 0 (no difficulty) to 10 (extreme difficulty), where higher scores indicated extreme difficulty/worse physical function. Missing data was imputed using mixed BOCF/LOCF.
Time Frame: Weeks 2, 4, 8, 16, 24, 32, 40, 48, 56 and 64
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either Tanezumab or matching placebo). "Overall number of participants analyzed" = participants who were evaluable for this outcome measure. "Number analyzed"=participants who were evaluable for this outcome measure at specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1000 | 995 | 994
percentage of participants
  Week 2: At least 30% reduction | 35.8 | 32.1 | 31.7
  Week 2: At least 50% reduction | 20.0 | 17.0 | 15.4
  Week 2: At least 70% reduction | 8.3 | 8.2 | 5.8
  Week 2: At least 90% reduction | 2.1 | 3.2 | 1.7
  Week 4: At least 30% reduction | 49.0 | 49.1 | 43.2
  Week 4: At least 50% reduction | 31.1 | 31.3 | 23.1
  Week 4: At least 70% reduction | 15.5 | 15.8 | 11.2
  Week 4: At least 90% reduction | 4.6 | 5.4 | 2.6
  Week 8: At least 30% reduction | 56.0 | 59.5 | 55.0
  Week 8: At least 50% reduction | 36.6 | 40.0 | 31.4
  Week 8: At least 70% reduction | 18.7 | 21.3 | 14.1
  Week 8: At least 90% reduction | 5.8 | 7.1 | 4.4
  Week 16: At least 30% reduction | 71.6 | 71.8 | 68.1
  Week 16: At least 50% reduction | 53.1 | 55.8 | 50.1
  Week 16: At least 70% reduction | 29.9 | 34.3 | 27.9
  Week 16: At least 90% reduction | 10.7 | 13.4 | 9.7
  Week 24: At least 30% reduction | 59.5 | 61.3 | 59.0
  Week 24: At least 50% reduction | 49.9 | 48.2 | 46.8
  Week 24: At least 70% reduction | 30.4 | 32.7 | 27.8
  Week 24: At least 90% reduction | 11.0 | 13.0 | 9.8
  Week 32: At least 30% reduction | 56.7 | 56.6 | 55.9
  Week 32: At least 50% reduction | 47.2 | 45.7 | 44.7
  Week 32: At least 70% reduction | 29.7 | 30.2 | 26.8
  Week 32: At least 90% reduction | 11.0 | 13.1 | 9.4
  Week 40: At least 30% reduction | 55.5 | 55.5 | 54.9
  Week 40: At least 50% reduction | 45.5 | 45.0 | 45.0
  Week 40: At least 70% reduction | 29.5 | 29.1 | 27.6
  Week 40: At least 90% reduction | 10.3 | 13.2 | 9.5
  Week 48: At least 30% reduction | 54.5 | 53.3 | 54.6
  Week 48: At least 50% reduction | 45.3 | 43.5 | 43.4
  Week 48: At least 70% reduction | 29.1 | 27.9 | 26.1
  Week 48: At least 90% reduction | 10.2 | 12.0 | 9.4
  Week 56: At least 30% reduction | 52.0 | 51.1 | 52.9
  Week 56: At least 50% reduction | 44.1 | 41.3 | 42.5
  Week 56: At least 70% reduction | 26.9 | 26.4 | 26.0
  Week 56: At least 90% reduction | 9.3 | 10.5 | 9.0
  Week 64: At least 30% reduction: number analyzed (Participants) | 437 | 419 | 445
  Week 64: At least 30% reduction | 71.4 | 68.0 | 78.2
  Week 64: At least 50% reduction: number analyzed (Participants) | 437 | 419 | 445
  Week 64: At least 50% reduction | 52.9 | 44.6 | 58.9
  Week 64: At least 70% reduction: number analyzed (Participants) | 437 | 419 | 445
  Week 64: At least 70% reduction | 31.4 | 22.9 | 33.9
  Week 64: At least 90% reduction: number analyzed (Participants) | 437 | 419 | 445
  Week 64: At least 90% reduction | 9.4 | 7.9 | 13.3
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Week 2: >=30% reduction; Test type: Superiority; p = 0.0651, Regression, Logistic; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.99 to 1.44] — OR and 95% CI estimated from logistic regression model.Logistic regression model included baseline WOMAC physical function subscale,baseline diary average pain,classification variables index joint,highest Kellgren-Lawrence grade,NSAID and treatment
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; Week 2: >=30% reduction; Test type: Superiority; p = 0.9032, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.84 to 1.22] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Tanezumab 2.5 mg vs NSAID; Week 2: >=50% reduction; Test type: Superiority; p = 0.0100, Regression, Logistic; Odds Ratio (OR) = 1.36, 95% CI 2-sided [1.08 to 1.72] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs NSAID; Week 2: >=50% reduction; Test type: Superiority; p = 0.3728, Regression, Logistic; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.88 to 1.42] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 5: Comparison: Tanezumab 2.5 mg vs NSAID; Week 2: >=70% reduction; Test type: Superiority; p = 0.0434, Regression, Logistic; Odds Ratio (OR) = 1.44, 95% CI 2-sided [1.01 to 2.04] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 6: Comparison: Tanezumab 5 mg vs NSAID; Week 2: >=70% reduction; Test type: Superiority; p = 0.0425, Regression, Logistic; Odds Ratio (OR) = 1.44, 95% CI 2-sided [1.01 to 2.04] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 7: Comparison: Tanezumab 2.5 mg vs NSAID; Week 2: >=90% reduction; Test type: Superiority; p = 0.5442, Regression, Logistic; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.64 to 2.34] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 8: Comparison: Tanezumab 5 mg vs NSAID; Week 2: >=90% reduction; Test type: Superiority; p = 0.0349, Regression, Logistic; Odds Ratio (OR) = 1.90, 95% CI 2-sided [1.05 to 3.45] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 9: Comparison: Tanezumab 2.5 mg vs NSAID; Week 4: >=30% reduction; Test type: Superiority; p = 0.0108, Regression, Logistic; Odds Ratio (OR) = 1.26, 95% CI 2-sided [1.05 to 1.51] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 10: Comparison: Tanezumab 5 mg vs NSAID; Week 4: >=30% reduction; Test type: Superiority; p = 0.0080, Regression, Logistic; Odds Ratio (OR) = 1.27, 95% CI 2-sided [1.07 to 1.52] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 11: Comparison: Tanezumab 2.5 mg vs NSAID; Week 4: >=50% reduction; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.50, 95% CI 2-sided [1.22 to 1.83] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 12: Comparison: Tanezumab 5 mg vs NSAID; Week 4: >=50% reduction; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.51, 95% CI 2-sided [1.24 to 1.85] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 13: Comparison: Tanezumab 2.5 mg vs NSAID; Week 4: >=70% reduction; Test type: Superiority; p = 0.0060, Regression, Logistic; Odds Ratio (OR) = 1.45, 95% CI 2-sided [1.11 to 1.88] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 14: Comparison: Tanezumab 5 mg vs NSAID; Week 4: >=70% reduction; Test type: Superiority; p = 0.0031, Regression, Logistic; Odds Ratio (OR) = 1.49, 95% CI 2-sided [1.14 to 1.93] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 15: Comparison: Tanezumab 2.5 mg vs NSAID; Week 4: >=90% reduction; Test type: Superiority; p = 0.0235, Regression, Logistic; Odds Ratio (OR) = 1.76, 95% CI 2-sided [1.08 to 2.88] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 16: Comparison: Tanezumab 5 mg vs NSAID; Week 4: >=90% reduction; Test type: Superiority; p = 0.0021, Regression, Logistic; Odds Ratio (OR) = 2.12, 95% CI 2-sided [1.31 to 3.42] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 17: Comparison: Tanezumab 2.5 mg vs NSAID; Week 8: >=30% reduction; Test type: Superiority; p = 0.7613, Regression, Logistic; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.86 to 1.23] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 18: Comparison: Tanezumab 5 mg vs NSAID; Week 8: >=30% reduction; Test type: Superiority; p = 0.0548, Regression, Logistic; Odds Ratio (OR) = 1.19, 95% CI 2-sided [1.00 to 1.43] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 19: Comparison: Tanezumab 2.5 mg vs NSAID; Week 8: >=50% reduction; Test type: Superiority; p = 0.0196, Regression, Logistic; Odds Ratio (OR) = 1.25, 95% CI 2-sided [1.04 to 1.51] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 20: Comparison: Tanezumab 5 mg vs NSAID; Week 8: >=50% reduction; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.45, 95% CI 2-sided [1.20 to 1.75] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 21: Comparison: Tanezumab 2.5 mg vs NSAID; Week 8: >=70% reduction; Test type: Superiority; p = 0.0077, Regression, Logistic; Odds Ratio (OR) = 1.39, 95% CI [1.09 to 1.77] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 22: Comparison: Tanezumab 5 mg vs NSAID; Week 8: >=70% reduction; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.65, 95% CI 2-sided [1.30 to 2.09] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 23: Comparison: Tanezumab 2.5 mg vs NSAID; Week 8: >=90% reduction; Test type: Superiority; p = 0.1942, Regression, Logistic; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.87 to 1.96] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 24: Comparison: Tanezumab 5 mg vs NSAID; Week 8: >=90% reduction; Test type: Superiority; p = 0.0122, Regression, Logistic; Odds Ratio (OR) = 1.64, 95% CI 2-sided [1.11 to 2.43] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 25: Comparison: Tanezumab 2.5 mg vs NSAID; Week 16: >=30% reduction; Test type: Superiority; p = 0.0977, Regression, Logistic; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.97 to 1.43] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 26: Comparison: Tanezumab 5 mg vs NSAID; Week 16: >=30% reduction; Test type: Superiority; p = 0.0806, Regression, Logistic; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.98 to 1.44] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 27: Comparison: Tanezumab 2.5 mg vs NSAID; Week 16: >=50% reduction; Test type: Superiority; p = 0.2097, Regression, Logistic; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.94 to 1.34] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 28: Comparison: Tanezumab 5 mg vs NSAID; Week 16: >=50% reduction; Test type: Superiority; p = 0.0135, Regression, Logistic; Odds Ratio (OR) = 1.25, 95% CI 2-sided [1.05 to 1.49] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 29: Comparison: Tanezumab 2.5 mg vs NSAID; Week 16: >=70% reduction; Test type: Superiority; p = 0.3571, Regression, Logistic; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.90 to 1.33] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 30: Comparison: Tanezumab 5 mg vs NSAID; Week 16: >=70% reduction; Test type: Superiority; p = 0.0025, Regression, Logistic; Odds Ratio (OR) = 1.34, 95% CI 2-sided [1.11 to 1.63] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 31: Comparison: Tanezumab 2.5 mg vs NSAID; Week 16: >=90% reduction; Test type: Superiority; p = 0.4658, Regression, Logistic; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.83 to 1.49] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 32: Comparison: Tanezumab 5 mg vs NSAID; Week 16: >=90% reduction; Test type: Superiority; p = 0.0108, Regression, Logistic; Odds Ratio (OR) = 1.44, 95% CI 2-sided [1.09 to 1.90] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 33: Comparison: Tanezumab 2.5 mg vs NSAID; Week 24: >=30% reduction; Test type: Superiority; p = 0.8393, Regression, Logistic; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.85 to 1.22] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 34: Comparison: Tanezumab 5 mg vs NSAID; Week 24: >=30% reduction; Test type: Superiority; p = 0.2977, Regression, Logistic; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.92 to 1.32] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 35: Comparison: Tanezumab 2.5 mg vs NSAID; Week 24: >=50% reduction; Test type: Superiority; p = 0.1944, Regression, Logistic; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.94 to 1.34] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 36: Comparison: Tanezumab 5 mg vs NSAID; Week 24: >=50% reduction; Test type: Superiority; p = 0.5714, Regression, Logistic; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.88 to 1.26] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 37: Comparison: Tanezumab 2.5 mg vs NSAID; Week 24: >=70% reduction; Test type: Superiority; p = 0.2472, Regression, Logistic; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.92 to 1.36] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 38: Comparison: Tanezumab 5 mg vs NSAID; Week 24: >=70% reduction; Test type: Superiority; p = 0.0235, Regression, Logistic; Odds Ratio (OR) = 1.25, 95% CI 2-sided [1.03 to 1.51] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 39: Comparison: Tanezumab 2.5 mg vs NSAID; Week 24: >=90% reduction; Test type: Superiority; p = 0.4074, Regression, Logistic; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.85 to 1.51] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 40: Comparison: Tanezumab 5 mg vs NSAID; Week 24: >=90% reduction; Test type: Superiority; p = 0.0296, Regression, Logistic; Odds Ratio (OR) = 1.37, 95% CI 2-sided [1.03 to 1.81] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 41: Comparison: Tanezumab 2.5 mg vs NSAID; Week 32: >=30% reduction; Test type: Superiority; p = 0.7607, Regression, Logistic; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.86 to 1.23] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 42: Comparison: Tanezumab 5 mg vs NSAID; Week 32: >=30% reduction; Test type: Superiority; p = 0.7979, Regression, Logistic; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.86 to 1.22] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 43: Comparison: Tanezumab 2.5 mg vs NSAID; Week 32: >=50% reduction; Test type: Superiority; p = 0.2964, Regression, Logistic; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.92 to 1.31] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 44: Comparison: Tanezumab 5 mg vs NSAID; Week 32: >=50% reduction; Test type: Superiority; p = 0.6950, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.87 to 1.24] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 45: Comparison: Tanezumab 2.5 mg vs NSAID; Week 32: >=70% reduction; Test type: Superiority; p = 0.1985, Regression, Logistic; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.93 to 1.38] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 46: Comparison: Tanezumab 5 mg vs NSAID; Week 32: >=70% reduction; Test type: Superiority; p = 0.1239, Regression, Logistic; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.96 to 1.42] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 47: Comparison: Tanezumab 2.5 mg vs NSAID; Week 32: >=90% reduction; Test type: Superiority; p = 0.2762, Regression, Logistic; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.88 to 1.58] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 48: Comparison: Tanezumab 5 mg vs NSAID; Week 32: >=90% reduction; Test type: Superiority; p = 0.0121, Regression, Logistic; Odds Ratio (OR) = 1.44, 95% CI 2-sided [1.08 to 1.91] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 49: Comparison: Tanezumab 2.5 mg vs NSAID; Week 40: >=30% reduction; Test type: Superiority; p = 0.8443, Regression, Logistic; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.85 to 1.22] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 50: Comparison: Tanezumab 5 mg vs NSAID; Week 40: >=30% reduction; Test type: Superiority; p = 0.8472, Regression, Logistic; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.85 to 1.22] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 51: Comparison: Tanezumab 2.5 mg vs NSAID; Week 40: >=50% reduction; Test type: Superiority; p = 0.8980, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.85 to 1.21] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 52: Comparison: Tanezumab 5 mg vs NSAID; Week 40: >=50% reduction; Test type: Superiority; p = 0.9385, Regression, Logistic; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.83 to 1.19] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 53: Comparison: Tanezumab 2.5 mg vs NSAID; Week 40: >=70% reduction; Test type: Superiority; p = 0.4261, Regression, Logistic; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.89 to 1.32] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 54: Comparison: Tanezumab 5 mg vs NSAID; Week 40: >=70% reduction; Test type: Superiority; p = 0.5250, Regression, Logistic; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.88 to 1.30] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 55: Comparison: Tanezumab 2.5 mg vs NSAID; Week 40: >=90% reduction; Test type: Superiority; p = 0.6273, Regression, Logistic; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.80 to 1.45] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 56: Comparison: Tanezumab 5 mg vs NSAID; Week 40: >=90% reduction; Test type: Superiority; p = 0.0132, Regression, Logistic; Odds Ratio (OR) = 1.43, 95% CI 2-sided [1.08 to 1.90] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 57: Comparison: Tanezumab 2.5 mg vs NSAID; Week 48: >=30% reduction; Test type: Superiority; p = 0.9095, Regression, Logistic; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.83 to 1.18] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 58: Comparison: Tanezumab 5 mg vs NSAID; Week 48: >=30% reduction; Test type: Superiority; p = 0.5098, Regression, Logistic; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.79 to 1.12] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 59: Comparison: Tanezumab 2.5 mg vs NSAID; Week 48: >=50% reduction; Test type: Superiority; p = 0.4488, Regression, Logistic; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.90 to 1.28] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 60: Comparison: Tanezumab 5 mg vs NSAID; Week 48: >=50% reduction; Test type: Superiority; p = 0.9757, Regression, Logistic; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.83 to 1.19] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 61: Comparison: Tanezumab 2.5 mg vs NSAID; Week 48: >=70% reduction; Test type: Superiority; p = 0.1843, Regression, Logistic; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.94 to 1.39] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 62: Comparison: Tanezumab 5 mg vs NSAID; Week 48: >=70% reduction; Test type: Superiority; p = 0.4356, Regression, Logistic; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.89 to 1.32] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 63: Comparison: Tanezumab 2.5 mg vs NSAID; Week 48: >=90% reduction; Test type: Superiority; p = 0.6342, Regression, Logistic; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.80 to 1.45] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 64: Comparison: Tanezumab 5 mg vs NSAID; Week 48: >=90% reduction; Test type: Superiority; p = 0.0810, Regression, Logistic; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.97 to 1.73] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 65: Comparison: Tanezumab 2.5 mg vs NSAID; Week 56: >=30% reduction; Test type: Superiority; p = 0.6527, Regression, Logistic; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.80 to 1.15] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 66: Comparison: Tanezumab 5 mg vs NSAID; Week 56: >=30% reduction; Test type: Superiority; p = 0.3857, Regression, Logistic; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.77 to 1.10] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 67: Comparison: Tanezumab 2.5 mg vs NSAID; Week 56: >=50% reduction; Test type: Superiority; p = 0.5280, Regression, Logistic; Odds Ratio, log = 1.06, 95% CI 2-sided [0.89 to 1.27] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 68: Comparison: Tanezumab 5 mg vs NSAID; Week 56: >=50% reduction; Test type: Superiority; p = 0.5355, Regression, Logistic; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.79 to 1.13] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 69: Comparison: Tanezumab 2.5 mg vs NSAID; Week 56: >=70% reduction; Test type: Superiority; p = 0.7732, Regression, Logistic; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.84 to 1.26] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 70: Comparison: Tanezumab 5 mg vs NSAID; Week 56: >=70% reduction; Test type: Superiority; p = 0.9397, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.82 to 1.23] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 71: Comparison: Tanezumab 2.5 mg vs NSAID; Week 56: >=90% reduction; Test type: Superiority; p = 0.9044, Regression, Logistic; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.75 to 1.39] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 72: Comparison: Tanezumab 5 mg vs NSAID; Week 56: >=90% reduction; Test type: Superiority; p = 0.3193, Regression, Logistic; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.86 to 1.57] — [estimate comment as in outcome 25, analysis 1]

26. Secondary Outcome: Percentage of Participants With Cumulative Percent Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale at Weeks 16, 24 and 56
Description: Percentage of participants with cumulative reduction (as percent) (> 0 %; >= 10%, 20%, 30%, 40%, 50%, 60%, 70%, 80% and 90%; =100%) in WOMAC physical function subscale from baseline to Weeks 16, 24 and 56 were reported. WOMAC:Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA. Physical function: participant's ability to move around and perform usual activities of daily living. WOMAC physical function subscale:17-item questionnaire to assess the degree of difficulty experienced due to OA in index joint (knee or hip) during past 48 hours, calculated as mean of the scores from 17 individual questions scored on a NRS. Scores for each question and WOMAC Pain subscale on NRS ranged from 0 (no difficulty) to 10 (extreme difficulty), higher scores indicate extreme difficulty/worse physical function. Missing data was imputed using mixed BOCF/LOCF.
Time Frame: Baseline, Weeks 16, 24 and 56
Population: as for outcome 24
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1000 | 995 | 994
percentage of participants
  Week 16: >0% | 90.0 | 88.8 | 87.4
  Week 16: >=10% | 85.0 | 83.9 | 81.4
  Week 16: >=20% | 78.4 | 77.3 | 73.7
  Week 16: >=30% | 71.6 | 71.8 | 68.1
  Week 16: >=40% | 63.7 | 64.1 | 61.0
  Week 16: >=50% | 53.1 | 55.8 | 50.1
  Week 16: >=60% | 41.4 | 44.7 | 39.8
  Week 16: >=70% | 29.9 | 34.3 | 27.9
  Week 16: >=80% | 20.8 | 24.4 | 17.9
  Week 16: >=90% | 10.7 | 13.4 | 9.7
  Week 16: =100% | 2.9 | 3.3 | 2.0
  Week 24: >0% | 66.7 | 68.6 | 65.0
  Week 24: >=10% | 65.0 | 66.6 | 63.3
  Week 24: >=20% | 62.6 | 64.2 | 60.8
  Week 24: >=30% | 59.5 | 61.3 | 59.0
  Week 24: >=40% | 54.9 | 56.0 | 53.9
  Week 24: >=50% | 49.9 | 48.2 | 46.8
  Week 24: >=60% | 41.3 | 42.0 | 37.7
  Week 24: >=70% | 30.4 | 32.7 | 27.8
  Week 24: >=80% | 19.9 | 22.6 | 18.9
  Week 24: >=90% | 11.0 | 13.0 | 9.8
  Week 24: =100% | 3.0 | 3.2 | 2.7
  Week 56: >0% | 61.1 | 59.5 | 60.1
  Week 56: >=10% | 59.3 | 57.3 | 57.8
  Week 56: >=20% | 56.1 | 54.3 | 55.4
  Week 56: >=30% | 52.0 | 51.1 | 52.9
  Week 56: >=40% | 48.5 | 46.3 | 48.9
  Week 56: >=50% | 44.1 | 41.3 | 42.5
  Week 56: >=60% | 36.7 | 34.6 | 34.8
  Week 56: >=70% | 26.9 | 26.4 | 26.0
  Week 56: >=80% | 17.1 | 17.1 | 17.4
  Week 56: >=90% | 9.3 | 10.5 | 9.0
  Week 56: =100% | 2.9 | 3.6 | 3.3

27. Secondary Outcome: Percentage of Participants Achieving Improvement of >=2 Points in Patient's Global Assessment (PGA) of Osteoarthritis at Weeks 2, 4, 8, 16, 24, 32, 40, 48, 56 and 64
Description: PGA of OA was assessed by asking a question from participants: "Considering all the ways your OA in your knee or hip affects you, how are you doing today?" Participants responded on a scale ranging from 1-5, where, 1=very good (no symptom and no limitation of normal activities), 2= good (mild symptoms and no limitation of normal activities), 3= fair (moderate symptoms and limitation of some normal activities), 4= poor (severe symptoms and inability to carry out most normal activities), and 5 = very poor (very severe symptoms and inability to carry out all normal activities). Higher scores indicated worse condition. Percentage of participants with improvement of at least 2 points from baseline in PGA of OA were reported. Missing data was imputed using mixed BOCF/LOCF.
Time Frame: Weeks 2, 4, 8, 16, 24, 32, 40, 48, 56 and 64
Population: as for outcome 25
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1000 | 995 | 994
percentage of participants
  Week 2 | 14.6 | 15.6 | 11.6
  Week 4 | 21.4 | 22.4 | 15.9
  Week 8 | 21.9 | 23.7 | 19.0
  Week 16 | 29.1 | 30.3 | 28.2
  Week 24 | 23.4 | 24.8 | 23.7
  Week 32 | 23.7 | 22.3 | 23.6
  Week 40 | 21.7 | 21.7 | 21.0
  Week 48 | 22.0 | 21.7 | 21.1
  Week 56 | 21.0 | 19.7 | 20.8
  Week 64: number analyzed (Participants) | 437 | 419 | 445
  Week 64 | 21.1 | 17.4 | 25.8
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Week 2: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline PGA of OA scale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade, NSAID and treatment; Test type: Superiority; p = 0.1772, Regression, Logistic; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.91 to 1.62]
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 27, analysis 1]; Test type: Superiority; p = 0.0154, Regression, Logistic; Odds Ratio (OR) = 1.42, 95% CI 2-sided [1.07 to 1.89]
Statistical Analysis 3: Comparison: Tanezumab 2.5 mg vs NSAID; Week 4: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline PGA of OA scale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade, NSAID and treatment; Test type: Superiority; p = 0.0105, Regression, Logistic; Odds Ratio (OR) = 1.40, 95% CI 2-sided [1.08 to 1.81]
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 27, analysis 3]; Test type: Superiority; p = 0.0002, Regression, Logistic; Odds Ratio (OR) = 1.63, 95% CI 2-sided [1.26 to 2.10]
Statistical Analysis 5: Comparison: Tanezumab 2.5 mg vs NSAID; Week 8: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline PGA of OA scale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade, NSAID and treatment; Test type: Superiority; p = 0.4007, Regression, Logistic; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.87 to 1.43]
Statistical Analysis 6: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 27, analysis 5]; Test type: Superiority; p = 0.0116, Regression, Logistic; Odds Ratio (OR) = 1.37, 95% CI 2-sided [1.07 to 1.75]
Statistical Analysis 7: Comparison: Tanezumab 2.5 mg vs NSAID; Week 16: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline PGA of OA scale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade, NSAID and treatment; Test type: Superiority; p = 0.6279, Regression, Logistic; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.76 to 1.18]
Statistical Analysis 8: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 27, analysis 7]; Test type: Superiority; p = 0.4674, Regression, Logistic; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.87 to 1.35]
Statistical Analysis 9: Comparison: Tanezumab 2.5 mg vs NSAID; Week 24: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline PGA of OA scale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade, NSAID and treatment; Test type: Superiority; p = 0.3135, Regression, Logistic; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.71 to 1.12]
Statistical Analysis 10: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 27, analysis 9]; Test type: Superiority; p = 0.7581, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.83 to 1.30]
Statistical Analysis 11: Comparison: Tanezumab 2.5 mg vs NSAID; Week 32: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline PGA of OA scale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade, NSAID and treatment; Test type: Superiority; p = 0.4504, Regression, Logistic; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.73 to 1.15]
Statistical Analysis 12: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 27, analysis 11]; Test type: Superiority; p = 0.2629, Regression, Logistic; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.70 to 1.10]
Statistical Analysis 13: Comparison: Tanezumab 2.5 mg vs NSAID; Week 40: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline PGA of OA scale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade, NSAID and treatment; Test type: Superiority; p = 0.6763, Regression, Logistic; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.75 to 1.20]
Statistical Analysis 14: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 27, analysis 13]; Test type: Superiority; p = 0.9456, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.80 to 1.27]
Statistical Analysis 15: Comparison: Tanezumab 2.5 mg vs NSAID; Week 48: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline PGA of OA scale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade, NSAID and treatment; Test type: Superiority; p = 0.7520, Regression, Logistic; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.76 to 1.22]
Statistical Analysis 16: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 27, analysis 15]; Test type: Superiority; p = 0.9981, Regression, Logistic; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.79 to 1.26]
Statistical Analysis 17: Comparison: Tanezumab 2.5 mg vs NSAID; Week 56: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline PGA of OA scale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade, NSAID and treatment; Test type: Superiority; p = 0.5284, Regression, Logistic; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.74 to 1.17]
Statistical Analysis 18: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 27, analysis 17]; Test type: Superiority; p = 0.3220, Regression, Logistic; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.70 to 1.12]

28. Secondary Outcome: Change From Baseline in Average Pain Score in the Index Joint at Weeks 1, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24, 32, 40, 48 and 56
Description: Participants assessed their average pain in the index hip/knee in the past 24 hours using NRS, with a scale ranging from 0 (no pain) to 10 (worst possible pain). Higher scores indicated higher pain. Data for Weeks 20 through 56 represents averages of the values reported during the 4-week interval up to and including the given week. Change from baseline was calculated using the difference between each post-baseline weekly mean and the baseline mean score.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24, 32, 40, 48 and 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
units on a scale
  Change at Week 1 | -0.47 (0.05) | -0.56 (0.05) | -0.56 (0.05)
  Change at Week 2 | -1.02 (0.07) | -0.97 (0.07) | -0.91 (0.07)
  Change at Week 3 | -1.40 (0.08) | -1.30 (0.08) | -1.23 (0.08)
  Change at Week 4 | -1.62 (0.09) | -1.65 (0.09) | -1.32 (0.09)
  Change at Week 6 | -1.85 (0.09) | -1.97 (0.09) | -1.49 (0.09)
  Change at Week 8 | -1.83 (0.10) | -2.04 (0.10) | -1.59 (0.10)
  Change at Week 10 | -2.35 (0.10) | -2.46 (0.10) | -1.98 (0.10)
  Change at Week 12 | -2.48 (0.10) | -2.55 (0.10) | -2.10 (0.10)
  Change at Week 16 | -2.41 (0.10) | -2.52 (0.10) | -2.17 (0.11)
  Change at Week 20 | -2.56 (0.11) | -2.60 (0.11) | -2.27 (0.11)
  Change at Week 24 | -2.35 (0.13) | -2.41 (0.12) | -2.11 (0.12)
  Change at Week 32 | -2.27 (0.13) | -2.26 (0.13) | -2.06 (0.13)
  Change at Week 40 | -2.25 (0.13) | -2.20 (0.13) | -2.07 (0.13)
  Change at Week 48 | -2.20 (0.13) | -2.10 (0.13) | -2.03 (0.13)
  Change at Week 56 | -2.17 (0.13) | -2.03 (0.13) | -2.04 (0.13)
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Week 1: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline pain in the index joint as covariate, and study site as a random effect; Test type: Superiority; p = 0.1120, ANCOVA; LS Mean Difference = 0.09, 95% CI 2-sided [-0.02 to 0.20], Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 28, analysis 1]; Test type: Superiority; p = 0.9686, ANCOVA; LS Mean Difference = 0.00, 95% CI 2-sided [-0.11 to 0.11], Standard Error of Mean 0.06
Statistical Analysis 3: Comparison: Tanezumab 2.5 mg vs NSAID; Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline pain in the index joint as covariate, and study site as a random effect; Test type: Superiority; p = 0.1589, ANCOVA; LS Mean Difference = -0.11, 95% CI 2-sided [-0.25 to 0.04], Standard Error of Mean 0.08
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 28, analysis 3]; Test type: Superiority; p = 0.4720, ANCOVA; LS Mean Difference = -0.05, 95% CI 2-sided [-0.20 to 0.09], Standard Error of Mean 0.08
Statistical Analysis 5: Comparison: Tanezumab 2.5 mg vs NSAID; Week 3: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline pain in the index joint as covariate, and study site as a random effect; Test type: Superiority; p = 0.0320, ANCOVA; LS Mean Difference = -0.17, 95% CI 2-sided [-0.33 to -0.01], Standard Error of Mean 0.08
Statistical Analysis 6: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 28, analysis 5]; Test type: Superiority; p = 0.3336, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-0.24 to 0.08], Standard Error of Mean 0.08
Statistical Analysis 7: Comparison: Tanezumab 2.5 mg vs NSAID; Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline pain in the index joint as covariate, and study site as a random effect; Test type: Superiority; p = 0.0005, ANCOVA; LS Mean Difference = -0.30, 95% CI 2-sided [-0.47 to -0.13], Standard Error of Mean 0.09
Statistical Analysis 8: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 28, analysis 7]; Test type: Superiority; p = 0.0001, ANCOVA; LS Mean Difference = -0.33, 95% CI 2-sided [-0.50 to -0.16], Standard Error of Mean 0.09
Statistical Analysis 9: Comparison: Tanezumab 2.5 mg vs NSAID; Week 6: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline pain in the index joint as covariate, and study site as a random effect; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -0.37, 95% CI 2-sided [-0.55 to -0.18], Standard Error of Mean 0.09
Statistical Analysis 10: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 28, analysis 9]; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -0.48, 95% CI 2-sided [-0.66 to -0.30], Standard Error of Mean 0.09
Statistical Analysis 11: Comparison: Tanezumab 2.5 mg vs NSAID; Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline pain in the index joint as covariate, and study site as a random effect; Test type: Superiority; p = 0.0115, ANCOVA; LS Mean Difference = -0.24, 95% CI 2-sided [-0.42 to -0.05], Standard Error of Mean 0.09
Statistical Analysis 12: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 28, analysis 11]; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -0.45, 95% CI 2-sided [-0.63 to -0.26], Standard Error of Mean 0.09
Statistical Analysis 13: Comparison: Tanezumab 2.5 mg vs NSAID; Week 10: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline pain in the index joint as covariate, and study site as a random effect; Test type: Superiority; p = 0.0002, ANCOVA; LS Mean Difference = -0.36, 95% CI 2-sided [-0.56 to -0.17], Standard Error of Mean 0.10
Statistical Analysis 14: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 28, analysis 13]; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -0.48, 95% CI 2-sided [-0.67 to -0.28], Standard Error of Mean 0.10
Statistical Analysis 15: Comparison: Tanezumab 2.5 mg vs NSAID; Week 12: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline pain in the index joint as covariate, and study site as a random effect; Test type: Superiority; p = 0.0002, ANCOVA; LS Mean Difference = -0.37, 95% CI 2-sided [-0.57 to -0.18], Standard Error of Mean 0.10
Statistical Analysis 16: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 28, analysis 15]; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -0.45, 95% CI 2-sided [-0.64 to -0.25], Standard Error of Mean 0.10
Statistical Analysis 17: Comparison: Tanezumab 2.5 mg vs NSAID; Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline pain in the index joint as covariate, and study site as a random effect; Test type: Superiority; p = 0.0238, ANCOVA; LS Mean Difference = -0.24, 95% CI 2-sided [-0.44 to -0.03], Standard Error of Mean 0.10
Statistical Analysis 18: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 28, analysis 17]; Test type: Superiority; p = 0.0011, ANCOVA; LS Mean Difference = -0.34, 95% CI 2-sided [-0.55 to -0.14], Standard Error of Mean 0.11
Statistical Analysis 19: Comparison: Tanezumab 2.5 mg vs NSAID; Week 20: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline pain in the index joint as covariate, and study site as a random effect; Test type: Superiority; p = 0.0064, ANCOVA; LS Mean Difference = -0.30, 95% CI 2-sided [-0.51 to -0.08], Standard Error of Mean 0.11
Statistical Analysis 20: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 28, analysis 19]; Test type: Superiority; p = 0.0025, ANCOVA; LS Mean Difference = -0.33, 95% CI 2-sided [-0.54 to -0.12], Standard Error of Mean 0.11
Statistical Analysis 21: Comparison: Tanezumab 2.5 mg vs NSAID; Week 24: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline pain in the index joint as covariate, and study site as a random effect; Test type: Superiority; p = 0.0589, ANCOVA; LS Mean Difference = -0.23, 95% CI 2-sided [-0.48 to 0.01], Standard Error of Mean 0.12
Statistical Analysis 22: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 28, analysis 21]; Test type: Superiority; p = 0.0180, ANCOVA; LS Mean Difference = -0.29, 95% CI 2-sided [-0.53 to -0.05], Standard Error of Mean 0.12
Statistical Analysis 23: Comparison: Tanezumab 2.5 mg vs NSAID; Week 32: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline pain in the index joint as covariate, and study site as a random effect; Test type: Superiority; p = 0.0944, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-0.47 to 0.04], Standard Error of Mean 0.13
Statistical Analysis 24: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 28, analysis 23]; Test type: Superiority; p = 0.1198, ANCOVA; LS Mean Difference = -0.20, 95% CI 2-sided [-0.45 to 0.05], Standard Error of Mean 0.13
Statistical Analysis 25: Comparison: Tanezumab 2.5 mg vs NSAID; Week 40: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline pain in the index joint as covariate, and study site as a random effect; Test type: Superiority; p = 0.1837, ANCOVA; LS Mean Difference = -0.17, 95% CI 2-sided [-0.43 to 0.08], Standard Error of Mean 0.13
Statistical Analysis 26: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 28, analysis 25]; Test type: Superiority; p = 0.3170, ANCOVA; LS Mean Difference = -0.13, 95% CI 2-sided [-0.39 to 0.13], Standard Error of Mean 0.13
Statistical Analysis 27: Comparison: Tanezumab 2.5 mg vs NSAID; Week 48: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline pain in the index joint as covariate, and study site as a random effect; Test type: Superiority; p = 0.1873, ANCOVA; LS Mean Difference = -0.17, 95% CI 2-sided [-0.43 to 0.08], Standard Error of Mean 0.13
Statistical Analysis 28: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 28, analysis 27]; Test type: Superiority; p = 0.5719, ANCOVA; LS Mean Difference = -0.07, 95% CI 2-sided [-0.33 to 0.18], Standard Error of Mean 0.13
Statistical Analysis 29: Comparison: Tanezumab 2.5 mg vs NSAID; Week 56: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline pain in the index joint as covariate, and study site as a random effect; Test type: Superiority; p = 0.3571, ANCOVA; LS Mean Difference = -0.12, 95% CI 2-sided [-0.39 to 0.14], Standard Error of Mean 0.13
Statistical Analysis 30: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 28, analysis 29]; Test type: Superiority; p = 0.9072, ANCOVA; LS Mean Difference = 0.02, 95% CI 2-sided [-0.25 to 0.28], Standard Error of Mean 0.14

29. Secondary Outcome: Change From Baseline in Average Pain Score in the Index Joint at Week 64
Description: Participants assessed their average pain in the index hip/knee in the past 24 hours using NRS, with a scale ranging from 0 (no pain) to 10 (worst possible pain). Higher scores indicated higher pain. Data represents averages of the values reported during the 4-week interval up to and including Week 64. Change from baseline was calculated using the difference between each post-baseline weekly mean and the baseline mean score.
Time Frame: Baseline, Week 64
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
units on a scale
  Baseline: number analyzed (Participants) | 995 | 992 | 990
  Baseline | 6.76 (1.59) | 6.77 (1.58) | 6.76 (1.54)
  Change at Week 64: number analyzed (Participants) | 436 | 416 | 434
  Change at Week 64 | -3.01 (2.60) | -2.81 (2.71) | -3.24 (2.55)

30. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale at Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA. Stiffness was defined as a sensation of decreased ease of movement in the index joint (knee or hip). The WOMAC stiffness subscale is a 2-item questionnaire used to assess the amount of stiffness experienced due to OA in the index joint (knee or hip) during the past 48 hours. It was calculated as the mean of scores from 2 individual questions scored on NRS. Scores for each question and WOMAC stiffness subscale score on NRS ranged from 0 (no stiffness) to 10 (extreme stiffness), where higher scores indicated higher stiffness.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
units on a scale
  Change at Week 2 | -1.79 (0.09) | -1.70 (0.09) | -1.48 (0.09)
  Change at Week 4 | -2.32 (0.10) | -2.43 (0.10) | -1.95 (0.10)
  Change at Week 8 | -2.46 (0.10) | -2.79 (0.10) | -2.16 (0.10)
  Change at Week 16 | -3.32 (0.11) | -3.54 (0.11) | -3.10 (0.11)
  Change at Week 24 | -2.77 (0.13) | -2.95 (0.13) | -2.63 (0.13)
  Change at Week 32 | -2.68 (0.13) | -2.74 (0.13) | -2.52 (0.13)
  Change at Week 40 | -2.58 (0.14) | -2.64 (0.14) | -2.46 (0.14)
  Change at Week 48 | -2.60 (0.14) | -2.54 (0.13) | -2.44 (0.14)
  Change at Week 56 | -2.46 (0.14) | -2.46 (0.14) | -2.42 (0.14)
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC stiffness subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0004, ANCOVA; LS Mean Difference = -0.31, 95% CI 2-sided [-0.49 to -0.14], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 30, analysis 1]; Test type: Superiority; p = 0.0134, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-0.40 to -0.05], Standard Error of Mean 0.09
Statistical Analysis 3: Comparison: Tanezumab 2.5 mg vs NSAID; Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC stiffness subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -0.38, 95% CI 2-sided [-0.56 to -0.19], Standard Error of Mean 0.10
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 30, analysis 3]; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -0.48, 95% CI 2-sided [-0.67 to -0.29], Standard Error of Mean 0.10
Statistical Analysis 5: Comparison: Tanezumab 2.5 mg vs NSAID; Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC stiffness subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0031, ANCOVA; LS Mean Difference = -0.29, 95% CI 2-sided [-0.49 to -0.10], Standard Error of Mean 0.10
Statistical Analysis 6: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 30, analysis 5]; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -0.63, 95% CI 2-sided [-0.82 to -0.43], Standard Error of Mean 0.10
Statistical Analysis 7: Comparison: Tanezumab 2.5 mg vs NSAID; Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC stiffness subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0425, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-0.43 to -0.01], Standard Error of Mean 0.11
Statistical Analysis 8: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 30, analysis 7]; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -0.44, 95% CI 2-sided [-0.65 to -0.23], Standard Error of Mean 0.11
Statistical Analysis 9: Comparison: Tanezumab 2.5 mg vs NSAID; Week 24: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC stiffness subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.2980, ANCOVA; LS Mean Difference = -0.14, 95% CI 2-sided [-0.40 to 0.12], Standard Error of Mean 0.13
Statistical Analysis 10: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 30, analysis 9]; Test type: Superiority; p = 0.0179, ANCOVA; LS Mean Difference = -0.32, 95% CI 2-sided [-0.58 to -0.05], Standard Error of Mean 0.13
Statistical Analysis 11: Comparison: Tanezumab 2.5 mg vs NSAID; Week 32: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC stiffness subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.2328, ANCOVA; LS Mean Difference = -0.16, 95% CI 2-sided [-0.42 to 0.10], Standard Error of Mean 0.13
Statistical Analysis 12: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 30, analysis 11]; Test type: Superiority; p = 0.1019, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-0.49 to 0.04], Standard Error of Mean 0.14
Statistical Analysis 13: Comparison: Tanezumab 2.5 mg vs NSAID; Week 40: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC stiffness subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.4002, ANCOVA; LS Mean Difference = -0.12, 95% CI 2-sided [-0.38 to 0.15], Standard Error of Mean 0.14
Statistical Analysis 14: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 30, analysis 13]; Test type: Superiority; p = 0.2149, ANCOVA; LS Mean Difference = -0.17, 95% CI 2-sided [-0.45 to 0.10], Standard Error of Mean 0.14
Statistical Analysis 15: Comparison: Tanezumab 2.5 mg vs NSAID; Week 48: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC stiffness subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.2442, ANCOVA; LS Mean Difference = -0.16, 95% CI 2-sided [-0.43 to 0.11], Standard Error of Mean 0.14
Statistical Analysis 16: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 30, analysis 15]; Test type: Superiority; p = 0.4609, ANCOVA; LS Mean Difference = -0.10, 95% CI 2-sided [-0.37 to 0.17], Standard Error of Mean 0.14
Statistical Analysis 17: Comparison: Tanezumab 2.5 mg vs NSAID; Week 56: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC stiffness subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.8129, ANCOVA; LS Mean Difference = -0.03, 95% CI 2-sided [-0.31 to 0.24], Standard Error of Mean 0.14
Statistical Analysis 18: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 30, analysis 17]; Test type: Superiority; p = 0.7883, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.32 to 0.24], Standard Error of Mean 0.14

31. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale at Week 64
Description: as for outcome 30
Time Frame: Baseline, Week 64
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
units on a scale
  Baseline: number analyzed (Participants) | 1000 | 995 | 994
  Baseline | 7.15 (1.42) | 7.20 (1.40) | 7.09 (1.42)
  Change at Week 64: number analyzed (Participants) | 437 | 419 | 445
  Change at Week 64 | -3.31 (2.72) | -3.04 (2.64) | -3.66 (2.36)

32. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Average Score at Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA of index joint (knee or hip). WOMAC pain subscale assess amount of pain experienced (score: 0 [no pain] to 10 [extreme pain], higher score = more pain), WOMAC physical function subscale assess degree of difficulty experienced (score: 0 [no difficulty] to 10 [extreme difficulty], higher score = worse physical function) and WOMAC stiffness subscale assess the amount of stiffness experienced (score: 0 [no stiffness] to 10 [extreme stiffness], higher score = higher stiffness). WOMAC average score was the mean of WOMAC pain, physical function and stiffness subscale scores and ranges from 0 to 10, where higher scores indicated worse response.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
units on a scale
  Change at Week 2 | -1.73 (0.08) | -1.61 (0.08) | -1.52 (0.08)
  Change at Week 4 | -2.28 (0.09) | -2.34 (0.09) | -1.95 (0.09)
  Change at Week 8 | -2.44 (0.10) | -2.71 (0.10) | -2.23 (0.10)
  Change at Week 16 | -3.26 (0.11) | -3.41 (0.11) | -3.07 (0.11)
  Change at Week 24 | -2.74 (0.13) | -2.88 (0.13) | -2.64 (0.13)
  Change at Week 32 | -2.65 (0.13) | -2.69 (0.13) | -2.54 (0.13)
  Change at Week 40 | -2.57 (0.13) | -2.58 (0.13) | -2.49 (0.13)
  Change at Week 48 | -2.56 (0.13) | -2.48 (0.13) | -2.44 (0.13)
  Change at Week 56 | -2.45 (0.13) | -2.38 (0.13) | -2.40 (0.13)
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC average score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0119, ANCOVA; LS Mean Difference = -0.21, 95% CI 2-sided [-0.37 to -0.05], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 32, analysis 1]; Test type: Superiority; p = 0.3073, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-0.24 to 0.08], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: Tanezumab 2.5 mg vs NSAID; Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC average score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0002, ANCOVA; LS Mean Difference = -0.33, 95% CI 2-sided [-0.50 to -0.15], Standard Error of Mean 0.09
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 32, analysis 3]; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -0.39, 95% CI 2-sided [-0.56 to -0.22], Standard Error of Mean 0.09
Statistical Analysis 5: Comparison: Tanezumab 2.5 mg vs NSAID; Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC average score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0251, ANCOVA; LS Mean Difference = -0.21, 95% CI 2-sided [-0.39 to -0.03], Standard Error of Mean 0.09
Statistical Analysis 6: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 32, analysis 5]; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -0.48, 95% CI 2-sided [-0.66 to -0.30], Standard Error of Mean 0.09
Statistical Analysis 7: Comparison: Tanezumab 2.5 mg vs NSAID; Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC average score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0625, ANCOVA; LS Mean Difference = -0.19, 95% CI 2-sided [-0.39 to 0.01], Standard Error of Mean 0.10
Statistical Analysis 8: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 32, analysis 7]; Test type: Superiority; p = 0.0010, ANCOVA; LS Mean Difference = -0.34, 95% CI 2-sided [-0.54 to -0.14], Standard Error of Mean 0.10
Statistical Analysis 9: Comparison: Tanezumab 2.5 mg vs NSAID; Week 24: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC average score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.4005, ANCOVA; LS Mean Difference = -0.11, 95% CI 2-sided [-0.36 to 0.14], Standard Error of Mean 0.13
Statistical Analysis 10: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 32, analysis 9]; Test type: Superiority; p = 0.0530, ANCOVA; LS Mean Difference = -0.25, 95% CI 2-sided [-0.50 to 0.00], Standard Error of Mean 0.13
Statistical Analysis 11: Comparison: Tanezumab 2.5 mg vs NSAID; Week 32: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC average score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.4074, ANCOVA; LS Mean Difference = -0.11, 95% CI 2-sided [-0.37 to 0.15], Standard Error of Mean 0.13
Statistical Analysis 12: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 32, analysis 11]; Test type: Superiority; p = 0.2629, ANCOVA; LS Mean Difference = -0.15, 95% CI 2-sided [-0.41 to 0.11], Standard Error of Mean 0.13
Statistical Analysis 13: Comparison: Tanezumab 2.5 mg vs NSAID; Week 40: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC average score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.5582, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-0.34 to 0.18], Standard Error of Mean 0.13
Statistical Analysis 14: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 32, analysis 13]; Test type: Superiority; p = 0.4907, ANCOVA; LS Mean Difference = -0.09, 95% CI 2-sided [-0.35 to 0.17], Standard Error of Mean 0.13
Statistical Analysis 15: Comparison: Tanezumab 2.5 mg vs NSAID; Week 48: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC average score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.4043, ANCOVA; LS Mean Difference = -0.11, 95% CI 2-sided [-0.38 to 0.15], Standard Error of Mean 0.14
Statistical Analysis 16: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 32, analysis 15]; Test type: Superiority; p = 0.7663, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.31 to 0.23], Standard Error of Mean 0.14
Statistical Analysis 17: Comparison: Tanezumab 2.5 mg vs NSAID; Week 56: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC average score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.7415, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.31 to 0.22], Standard Error of Mean 0.14
Statistical Analysis 18: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 32, analysis 17]; Test type: Superiority; p = 0.8688, ANCOVA; LS Mean Difference = 0.02, 95% CI 2-sided [-0.24 to 0.29], Standard Error of Mean 0.13

33. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Average Score at Week 64
Description: as for outcome 32
Time Frame: Baseline, Week 64
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
units on a scale
  Baseline: number analyzed (Participants) | 1000 | 995 | 994
  Baseline | 7.09 (1.08) | 7.10 (1.10) | 7.01 (1.08)
  Change at Week 64: number analyzed (Participants) | 437 | 419 | 445
  Change at Week 64 | -3.40 (2.40) | -3.09 (2.37) | -3.77 (2.06)

34. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Item: Pain When Walking on a Flat Surface at Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA in index joint (knee or hip). Participants answered a question: "How much pain have you had when walking on a flat surface?". Participants responded about the amount of pain they experienced when walking on a flat surface by using a NRS of 0 (no pain) to 10 (extreme pain), where higher scores indicated higher pain.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
units on a scale
  Change at Week 2 | -1.54 (0.08) | -1.39 (0.08) | -1.46 (0.08)
  Change at Week 4 | -2.14 (0.10) | -2.15 (0.10) | -1.91 (0.10)
  Change at Week 8 | -2.26 (0.10) | -2.47 (0.10) | -2.22 (0.10)
  Change at Week 16 | -3.01 (0.11) | -3.13 (0.11) | -2.95 (0.11)
  Change at Week 24 | -2.64 (0.13) | -2.76 (0.13) | -2.60 (0.13)
  Change at Week 32 | -2.54 (0.13) | -2.54 (0.13) | -2.52 (0.14)
  Change at Week 40 | -2.48 (0.14) | -2.42 (0.14) | -2.48 (0.14)
  Change at Week 48 | -2.45 (0.14) | -2.34 (0.14) | -2.42 (0.14)
  Change at Week 56 | -2.37 (0.14) | -2.21 (0.14) | -2.39 (0.14)
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC pain when walking on a flat surface and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.3622, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-0.25 to 0.09], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 34, analysis 1]; Test type: Superiority; p = 0.3894, ANCOVA; LS Mean Difference = 0.07, 95% CI 2-sided [-0.09 to 0.24], Standard Error of Mean 0.09
Statistical Analysis 3: Comparison: Tanezumab 2.5 mg vs NSAID; Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC pain when walking on a flat surface and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0137, ANCOVA; LS Mean Difference = -0.23, 95% CI 2-sided [-0.42 to -0.05], Standard Error of Mean 0.09
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 34, analysis 3]; Test type: Superiority; p = 0.0106, ANCOVA; LS Mean Difference = -0.24, 95% CI 2-sided [-0.43 to -0.06], Standard Error of Mean 0.09
Statistical Analysis 5: Comparison: Tanezumab 2.5 mg vs NSAID; Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC pain when walking on a flat surface and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.7179, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.23 to 0.16], Standard Error of Mean 0.10
Statistical Analysis 6: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 34, analysis 5]; Test type: Superiority; p = 0.0120, ANCOVA; LS Mean Difference = -0.25, 95% CI 2-sided [-0.44 to -0.05], Standard Error of Mean 0.10
Statistical Analysis 7: Comparison: Tanezumab 2.5 mg vs NSAID; Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC pain when walking on a flat surface and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.5372, ANCOVA; LS Mean Difference = -0.07, 95% CI 2-sided [-0.28 to 0.15], Standard Error of Mean 0.11
Statistical Analysis 8: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 34, analysis 7]; Test type: Superiority; p = 0.0899, ANCOVA; LS Mean Difference = -0.18, 95% CI 2-sided [-0.40 to 0.03], Standard Error of Mean 0.11
Statistical Analysis 9: Comparison: Tanezumab 2.5 mg vs NSAID; Week 24: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC pain when walking on a flat surface and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.7646, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.30 to 0.22], Standard Error of Mean 0.13
Statistical Analysis 10: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 34, analysis 9]; Test type: Superiority; p = 0.2547, ANCOVA; LS Mean Difference = -0.15, 95% CI 2-sided [-0.41 to 0.11], Standard Error of Mean 0.13
Statistical Analysis 11: Comparison: Tanezumab 2.5 mg vs NSAID; Week 32: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC pain when walking on a flat surface and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.8806, ANCOVA; LS Mean Difference = -0.02, 95% CI 2-sided [-0.29 to 0.25], Standard Error of Mean 0.14
Statistical Analysis 12: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 34, analysis 11]; Test type: Superiority; p = 0.8416, ANCOVA; LS Mean Difference = -0.03, 95% CI 2-sided [-0.30 to 0.24], Standard Error of Mean 0.14
Statistical Analysis 13: Comparison: Tanezumab 2.5 mg vs NSAID; Week 40: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC pain when walking on a flat surface and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.9981, ANCOVA; LS Mean Difference = -0.00, 95% CI 2-sided [-0.28 to 0.28], Standard Error of Mean 0.14
Statistical Analysis 14: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 34, analysis 13]; Test type: Superiority; p = 0.6485, ANCOVA; LS Mean Difference = 0.06, 95% CI 2-sided [-0.21 to 0.34], Standard Error of Mean 0.14
Statistical Analysis 15: Comparison: Tanezumab 2.5 mg vs NSAID; Week 48: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC pain when walking on a flat surface and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.8317, ANCOVA; LS Mean Difference = -0.03, 95% CI 2-sided [-0.30 to 0.24], Standard Error of Mean 0.14
Statistical Analysis 16: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 34, analysis 15]; Test type: Superiority; p = 0.5819, ANCOVA; LS Mean Difference = 0.08, 95% CI 2-sided [-0.19 to 0.35], Standard Error of Mean 0.14
Statistical Analysis 17: Comparison: Tanezumab 2.5 mg vs NSAID; Week 56: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC pain when walking on a flat surface and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.8538, ANCOVA; LS Mean Difference = 0.03, 95% CI 2-sided [-0.26 to 0.31], Standard Error of Mean 0.14
Statistical Analysis 18: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 34, analysis 17]; Test type: Superiority; p = 0.1981, ANCOVA; LS Mean Difference = 0.19, 95% CI 2-sided [-0.10 to 0.47], Standard Error of Mean 0.15

35. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Item: Pain When Walking on a Flat Surface at Week 64
Description: as for outcome 34
Time Frame: Baseline, Week 64
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
units on a scale
  Baseline: number analyzed (Participants) | 1000 | 995 | 994
  Baseline | 6.86 (1.33) | 6.90 (1.34) | 6.86 (1.30)
  Change at Week 64: number analyzed (Participants) | 437 | 419 | 445
  Change at Week 64 | -3.20 (2.78) | -2.69 (2.58) | -3.67 (2.32)

36. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Item: Pain When Going Up or Down Stairs at Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA in index joint (knee or hip). Participants answered a question: "How much pain have you had when going up or down the stairs?" Participants responded about the amount of pain they experienced when going up or down stairs by using a NRS of 0 (no pain) to 10 (extreme pain), where higher scores indicated higher pain.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
units on a scale
  Change at Week 2 | -1.81 (0.08) | -1.66 (0.08) | -1.66 (0.09)
  Change at Week 4 | -2.34 (0.10) | -2.43 (0.10) | -2.08 (0.10)
  Change at Week 8 | -2.48 (0.10) | -2.81 (0.10) | -2.40 (0.10)
  Change at Week 16 | -3.34 (0.11) | -3.50 (0.11) | -3.18 (0.12)
  Change at Week 24 | -2.89 (0.13) | -3.03 (0.13) | -2.83 (0.14)
  Change at Week 32 | -2.76 (0.14) | -2.84 (0.14) | -2.74 (0.14)
  Change at Week 40 | -2.69 (0.14) | -2.74 (0.14) | -2.70 (0.14)
  Change at Week 48 | -2.70 (0.14) | -2.63 (0.14) | -2.67 (0.14)
  Change at Week 56 | -2.55 (0.14) | -2.47 (0.14) | -2.55 (0.14)
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC pain when going up or down stairs and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0846, ANCOVA; LS Mean Difference = -0.15, 95% CI 2-sided [-0.33 to 0.02], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 36, analysis 1]; Test type: Superiority; p = 0.9749, ANCOVA; LS Mean Difference = -0.00, 95% CI 2-sided [-0.18 to 0.17], Standard Error of Mean 0.09
Statistical Analysis 3: Comparison: Tanezumab 2.5 mg vs NSAID; Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC pain when going up or down stairs and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0076, ANCOVA; LS Mean Difference = -0.26, 95% CI 2-sided [-0.45 to -0.07], Standard Error of Mean 0.10
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 36, analysis 3]; Test type: Superiority; p = 0.0003, ANCOVA; LS Mean Difference = -0.35, 95% CI 2-sided [-0.54 to -0.16], Standard Error of Mean 0.10
Statistical Analysis 5: Comparison: Tanezumab 2.5 mg vs NSAID; Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC pain when going up or down stairs and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.4402, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-0.27 to 0.12], Standard Error of Mean 0.10
Statistical Analysis 6: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 36, analysis 5]; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -0.41, 95% CI 2-sided [-0.61 to -0.21], Standard Error of Mean 0.10
Statistical Analysis 7: Comparison: Tanezumab 2.5 mg vs NSAID; Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC pain when going up or down stairs and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.1543, ANCOVA; LS Mean Difference = -0.16, 95% CI 2-sided [-0.38 to 0.06], Standard Error of Mean 0.11
Statistical Analysis 8: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 36, analysis 7]; Test type: Superiority; p = 0.0053, ANCOVA; LS Mean Difference = -0.31, 95% CI 2-sided [-0.53 to -0.09], Standard Error of Mean 0.11
Statistical Analysis 9: Comparison: Tanezumab 2.5 mg vs NSAID; Week 24: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC pain when going up or down stairs and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.6445, ANCOVA; LS Mean Difference = -0.06, 95% CI 2-sided [-0.33 to 0.20], Standard Error of Mean 0.14
Statistical Analysis 10: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 36, analysis 9]; Test type: Superiority; p = 0.1439, ANCOVA; LS Mean Difference = -0.20, 95% CI 2-sided [-0.47 to 0.07], Standard Error of Mean 0.14
Statistical Analysis 11: Comparison: Tanezumab 2.5 mg vs NSAID; Week 32: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC pain when going up or down stairs and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.8402, ANCOVA; LS Mean Difference = -0.03, 95% CI 2-sided [-0.30 to 0.25], Standard Error of Mean 0.14
Statistical Analysis 12: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 36, analysis 11]; Test type: Superiority; p = 0.4439, ANCOVA; LS Mean Difference = -0.11, 95% CI 2-sided [-0.38 to 0.17], Standard Error of Mean 0.14
Statistical Analysis 13: Comparison: Tanezumab 2.5 mg vs NSAID; Week 40: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC pain when going up or down stairs and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.9376, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-0.27 to 0.29], Standard Error of Mean 0.14
Statistical Analysis 14: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 36, analysis 13]; Test type: Superiority; p = 0.7614, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.33 to 0.24], Standard Error of Mean 0.14
Statistical Analysis 15: Comparison: Tanezumab 2.5 mg vs NSAID; Week 48: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC pain when going up or down stairs and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.8081, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.32 to 0.25], Standard Error of Mean 0.15
Statistical Analysis 16: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 36, analysis 15]; Test type: Superiority; p = 0.8078, ANCOVA; LS Mean Difference = 0.04, 95% CI 2-sided [-0.25 to 0.33], Standard Error of Mean 0.15
Statistical Analysis 17: Comparison: Tanezumab 2.5 mg vs NSAID; Week 56: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WOMAC pain when going up or down stairs and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.9705, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-0.28 to 0.29], Standard Error of Mean 0.15
Statistical Analysis 18: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 36, analysis 17]; Test type: Superiority; p = 0.5785, ANCOVA; LS Mean Difference = 0.08, 95% CI 2-sided [-0.21 to 0.38], Standard Error of Mean 0.15

37. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Item: Pain When Going Up or Down Stairs at Week 64
Description: as for outcome 36
Time Frame: Baseline, Week 64
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
units on a scale
  Baseline: number analyzed (Participants) | 1000 | 995 | 994
  Baseline | 7.89 (1.24) | 7.88 (1.29) | 7.83 (1.19)
  Change at Week 64: number analyzed (Participants) | 437 | 419 | 445
  Change at Week 64 | -3.28 (2.67) | -2.97 (2.69) | -3.70 (2.50)

38. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment Questionnaire for Osteoarthritis (WPAI:OA) Scores at Weeks 16, 24 and 56
Description: WPAI is 6-question participant rated questionnaire to determine the impact of OA on absenteeism, presenteeism, work productivity, and daily activity impairment for a period of 7 days prior to a visit. It yields 4 sub-scores: work time missed (absenteeism), impairment while working (presenteeism), overall work impairment (work productivity) and activity impairment (daily activity impairment). These sub-scores are expressed as an impairment percentage (range from 0 to 100), with higher numbers indicating greater impairment and less productivity.
Time Frame: Weeks 16, 24 and 56
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
units on a scale
  Change at Week 16: Percent Work Time Missed: number analyzed (Participants) | 350 | 339 | 338
  Change at Week 16: Percent Work Time Missed | -2.33 (0.62) | -3.35 (0.64) | -2.92 (0.63)
  Change at Week 16:Percent Impairment While Working: number analyzed (Participants) | 343 | 336 | 336
  Change at Week 16:Percent Impairment While Working | -28.07 (1.58) | -26.94 (1.61) | -26.59 (1.60)
  Change at Week 16: Percent Overall Work Impairment: number analyzed (Participants) | 343 | 336 | 336
  Change at Week 16: Percent Overall Work Impairment | -28.67 (1.62) | -27.51 (1.65) | -27.04 (1.63)
  Change at Week 16: Percent Activity Impairment: number analyzed (Participants) | 932 | 941 | 930
  Change at Week 16: Percent Activity Impairment | -30.59 (1.04) | -31.36 (1.04) | -29.38 (1.05)
  Change at Week 24: Percent Work Time Missed: number analyzed (Participants) | 300 | 286 | 282
  Change at Week 24: Percent Work Time Missed | -2.70 (0.80) | -2.19 (0.81) | -2.73 (0.81)
  Change at Week 24:Percent Impairment While Working: number analyzed (Participants) | 297 | 282 | 279
  Change at Week 24:Percent Impairment While Working | -25.34 (1.73) | -26.66 (1.74) | -25.15 (1.74)
  Change at Week 24: Percent Overall Work Impairment: number analyzed (Participants) | 297 | 282 | 279
  Change at Week 24: Percent Overall Work Impairment | -26.05 (1.78) | -27.33 (1.80) | -25.90 (1.80)
  Change at Week 24: Percent Activity Impairment: number analyzed (Participants) | 822 | 821 | 820
  Change at Week 24: Percent Activity Impairment | -29.88 (1.13) | -30.53 (1.13) | -29.76 (1.14)
  Change at Week 56: Percent Work Time Missed: number analyzed (Participants) | 163 | 178 | 152
  Change at Week 56: Percent Work Time Missed | -0.12 (1.56) | -1.84 (1.47) | -0.81 (1.53)
  Change at Week 56:Percent Impairment While Working: number analyzed (Participants) | 162 | 174 | 152
  Change at Week 56:Percent Impairment While Working | -31.49 (2.22) | -29.92 (2.12) | -34.59 (2.17)
  Change at Week 56: Percent Overall Work Impairment: number analyzed (Participants) | 162 | 174 | 152
  Change at Week 56: Percent Overall Work Impairment | -31.21 (2.39) | -29.29 (2.28) | -34.26 (2.34)
  Change at Week 56: Percent Activity Impairment: number analyzed (Participants) | 480 | 486 | 477
  Change at Week 56: Percent Activity Impairment | -34.47 (1.42) | -32.91 (1.39) | -36.17 (1.41)
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Week 16: Percent Work Time Missed: ANCOVA model included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WPAI score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.4303, ANCOVA; LS Mean Difference = 0.58, 95% CI 2-sided [-0.87 to 2.04], Standard Error of Mean 0.74
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 38, analysis 1]; Test type: Superiority; p = 0.5656, ANCOVA; LS Mean Difference = -0.43, 95% CI 2-sided [-1.90 to 1.04], Standard Error of Mean 0.75
Statistical Analysis 3: Comparison: Tanezumab 2.5 mg vs NSAID; Week 24: Percent Work Time Missed: ANCOVA model included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WPAI score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.9760, ANCOVA; LS Mean Difference = 0.03, 95% CI 2-sided [-1.78 to 1.83], Standard Error of Mean 0.92
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 38, analysis 3]; Test type: Superiority; p = 0.5678, ANCOVA; LS Mean Difference = 0.53, 95% CI 2-sided [-1.30 to 2.36], Standard Error of Mean 0.93
Statistical Analysis 5: Comparison: Tanezumab 2.5 mg vs NSAID; Week 56: Percent Work Time Missed: ANCOVA model included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WPAI score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.6974, ANCOVA; LS Mean Difference = 0.68, 95% CI 2-sided [-2.77 to 4.14], Standard Error of Mean 1.76
Statistical Analysis 6: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 38, analysis 5]; Test type: Superiority; p = 0.1261, ANCOVA; LS Mean Difference = 2.64, 95% CI 2-sided [-0.75 to 6.04], Standard Error of Mean 1.72
Statistical Analysis 7: Comparison: Tanezumab 2.5 mg vs NSAID; Week 16: Percent Impairment While Working: ANCOVA model included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WPAI score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.4060, ANCOVA; LS Mean Difference = -1.48, 95% CI 2-sided [-4.96 to 2.01], Standard Error of Mean 1.78
Statistical Analysis 8: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 38, analysis 7]; Test type: Superiority; p = 0.8480, ANCOVA; LS Mean Difference = -0.34, 95% CI 2-sided [-3.84 to 3.15], Standard Error of Mean 1.78
Statistical Analysis 9: Comparison: Tanezumab 2.5 mg vs NSAID; Week 24: Percent Impairment While Working: ANCOVA model included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WPAI score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.9230, ANCOVA; LS Mean Difference = -0.19, 95% CI 2-sided [-4.00 to 3.63], Standard Error of Mean 1.94
Statistical Analysis 10: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 38, analysis 9]; Test type: Superiority; p = 0.4421, ANCOVA; LS Mean Difference = -1.51, 95% CI 2-sided [-5.36 to 2.34], Standard Error of Mean 1.96
Statistical Analysis 11: Comparison: Tanezumab 2.5 mg vs NSAID; Week 56: Percent Impairment While Working: ANCOVA model included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WPAI score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.2049, ANCOVA; LS Mean Difference = 3.10, 95% CI 2-sided [-1.70 to 7.91], Standard Error of Mean 2.44
Statistical Analysis 12: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 38, analysis 11]; Test type: Superiority; p = 0.0527, ANCOVA; LS Mean Difference = 4.68, 95% CI 2-sided [-0.05 to 9.41], Standard Error of Mean 2.40
Statistical Analysis 13: Comparison: Tanezumab 2.5 mg vs NSAID; Week 16: Percent Overall Work Impairment: ANCOVA model included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WPAI score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.3699, ANCOVA; LS Mean Difference = -1.63, 95% CI 2-sided [-5.21 to 1.94], Standard Error of Mean 1.82
Statistical Analysis 14: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 38, analysis 13]; Test type: Superiority; p = 0.7945, ANCOVA; LS Mean Difference = -0.48, 95% CI 2-sided [-4.06 to 3.11], Standard Error of Mean 1.83
Statistical Analysis 15: Comparison: Tanezumab 2.5 mg vs NSAID; Week 24: Percent Overall Work Impairment: ANCOVA model included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WPAI score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.9410, ANCOVA; LS Mean Difference = -0.15, 95% CI 2-sided [-4.13 to 3.83], Standard Error of Mean 2.03
Statistical Analysis 16: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 38, analysis 15]; Test type: Superiority; p = 0.4860, ANCOVA; LS Mean Difference = -1.43, 95% CI 2-sided [-5.44 to 2.59], Standard Error of Mean 2.05
Statistical Analysis 17: Comparison: Tanezumab 2.5 mg vs NSAID; Week 56: Percent Overall Work Impairment: ANCOVA model included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WPAI score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.2448, ANCOVA; LS Mean Difference = 3.05, 95% CI 2-sided [-2.10 to 8.20], Standard Error of Mean 2.62
Statistical Analysis 18: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 38, analysis 17]; Test type: Superiority; p = 0.0551, ANCOVA; LS Mean Difference = 4.96, 95% CI 2-sided [-0.11 to 10.04], Standard Error of Mean 2.58
Statistical Analysis 19: Comparison: Tanezumab 2.5 mg vs NSAID; Week 16: Percent Activity Impairment: ANCOVA model included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WPAI score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.2470, ANCOVA; LS Mean Difference = -1.21, 95% CI 2-sided [-3.26 to 0.84], Standard Error of Mean 1.05
Statistical Analysis 20: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 38, analysis 19]; Test type: Superiority; p = 0.0570, ANCOVA; LS Mean Difference = -1.98, 95% CI 2-sided [-4.01 to 0.06], Standard Error of Mean 1.04
Statistical Analysis 21: Comparison: Tanezumab 2.5 mg vs NSAID; Week 24: Percent Activity Impairment: ANCOVA model included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WPAI score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.9170, ANCOVA; LS Mean Difference = -0.12, 95% CI 2-sided [-2.36 to 2.12], Standard Error of Mean 1.14
Statistical Analysis 22: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 38, analysis 21]; Test type: Superiority; p = 0.4991, ANCOVA; LS Mean Difference = -0.77, 95% CI 2-sided [-3.00 to 1.46], Standard Error of Mean 1.14
Statistical Analysis 23: Comparison: Tanezumab 2.5 mg vs NSAID; Week 56: Percent Activity Impairment: ANCOVA model included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline WPAI score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.2377, ANCOVA; LS Mean Difference = 1.70, 95% CI 2-sided [-1.12 to 4.52], Standard Error of Mean 1.44
Statistical Analysis 24: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 38, analysis 23]; Test type: Superiority; p = 0.0238, ANCOVA; LS Mean Difference = 3.26, 95% CI 2-sided [0.43 to 6.08], Standard Error of Mean 1.44

39. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment Questionnaire for Osteoarthritis (WPAI:OA) Scores at Week 64
Description: as for outcome 38
Time Frame: Baseline, Week 64
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
units on a scale
  Baseline: Percent Work Time Missed: number analyzed (Participants) | 438 | 417 | 420
  Baseline: Percent Work Time Missed | 6.1 (15.81) | 6.0 (15.56) | 5.2 (14.54)
  Baseline: Percent Impairment While Working: number analyzed (Participants) | 434 | 413 | 417
  Baseline: Percent Impairment While Working | 60.5 (20.39) | 58.3 (20.78) | 59.3 (18.97)
  Baseline: Percent Overall Work Impairment: number analyzed (Participants) | 434 | 413 | 417
  Baseline: Percent Overall Work Impairment | 62.1 (21.02) | 60.0 (21.37) | 60.6 (19.78)
  Baseline: Percent Activity Impairment: number analyzed (Participants) | 1000 | 995 | 994
  Baseline: Percent Activity Impairment | 68.3 (14.93) | 67.9 (15.83) | 66.7 (15.35)
  Change at Week 64: Percent Work Time Missed: number analyzed (Participants) | 149 | 137 | 142
  Change at Week 64: Percent Work Time Missed | -1.8 (19.35) | 4.1 (21.88) | -2.1 (16.65)
  Change at Week 64:Percent Impairment While Working: number analyzed (Participants) | 146 | 135 | 141
  Change at Week 64:Percent Impairment While Working | -24.2 (27.69) | -20.7 (29.13) | -26.5 (26.24)
  Change at Week 64: Percent Overall Work Impairment: number analyzed (Participants) | 146 | 135 | 141
  Change at Week 64: Percent Overall Work Impairment | -24.5 (28.77) | -19.2 (30.54) | -27.0 (27.22)
  Change at Week 64: Percent Activity Impairment: number analyzed (Participants) | 450 | 427 | 453
  Change at Week 64: Percent Activity Impairment | -28.7 (26.68) | -24.1 (27.80) | -32.1 (24.51)

40. Secondary Outcome: Number of Participants With Responses to European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L): Mobility Domain
Description: Number of participants with mobility domain responses of EQ-5D-5L were provided. EQ-5D-5L is a standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score. EQ-5D-5L consists of two components: a health state profile and an optional visual analogue scale (VAS). EQ-5D health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. Higher scores indicated greater levels of problems across the five dimensions.
Time Frame: Baseline, Weeks 8, 16, 24, 40, 56 and 64
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or matching placebo). Here, "Number analyzed" signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
Participants
  Baseline: number analyzed (Participants) | 1000 | 995 | 994
  Baseline: No problem in walking | 26 | 20 | 23
  Baseline: Slight problem in walking | 203 | 192 | 194
  Baseline: Moderate problem in walking | 567 | 579 | 588
  Baseline: Severe problem in walking | 204 | 202 | 189
  Baseline: Unable to walk | 0 | 2 | 0
  Week 8: number analyzed (Participants) | 956 | 966 | 956
  Week 8: No problem in walking | 223 | 241 | 216
  Week 8: Slight problem in walking | 374 | 411 | 392
  Week 8: Moderate problem in walking | 318 | 266 | 301
  Week 8: Severe problem in walking | 41 | 48 | 44
  Week 8: Unable to walk | 0 | 0 | 3
  Week 16: number analyzed (Participants) | 913 | 920 | 915
  Week 16: No problem in walking | 299 | 319 | 292
  Week 16: Slight problem in walking | 388 | 371 | 412
  Week 16: Moderate problem in walking | 199 | 196 | 185
  Week 16: Severe problem in walking | 27 | 34 | 26
  Week 16: Unable to walk | 0 | 0 | 0
  Week 24: number analyzed (Participants) | 817 | 816 | 813
  Week 24: No problem in walking | 259 | 261 | 260
  Week 24: Slight problem in walking | 308 | 310 | 337
  Week 24: Moderate problem in walking | 216 | 200 | 186
  Week 24: Severe problem in walking | 34 | 43 | 29
  Week 24: Unable to walk | 0 | 2 | 1
  Week 40: number analyzed (Participants) | 561 | 553 | 535
  Week 40: No problem in walking | 217 | 211 | 218
  Week 40: Slight problem in walking | 215 | 209 | 217
  Week 40: Moderate problem in walking | 110 | 106 | 91
  Week 40: Severe problem in walking | 19 | 27 | 9
  Week 40: Unable to walk | 0 | 0 | 0
  Week 56: number analyzed (Participants) | 458 | 458 | 459
  Week 56: No problem in walking | 157 | 147 | 170
  Week 56: Slight problem in walking | 205 | 166 | 189
  Week 56: Moderate problem in walking | 77 | 120 | 91
  Week 56: Severe problem in walking | 19 | 24 | 9
  Week 56: Unable to walk | 0 | 1 | 0
  Week 64: number analyzed (Participants) | 450 | 428 | 454
  Week 64: No problem in walking | 98 | 66 | 107
  Week 64: Slight problem in walking | 156 | 156 | 205
  Week 64: Moderate problem in walking | 150 | 151 | 121
  Week 64: Severe problem in walking | 45 | 54 | 21
  Week 64: Unable to walk | 1 | 1 | 0

41. Secondary Outcome: Number of Participants With Responses to European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L): Self-Care Domain
Description: Number of participants with self-care domain responses of EQ-5D-5L were provided. EQ-5D-5L is a standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score. EQ-5D-5L consists of two components: a health state profile and an optional visual analogue scale (VAS). EQ-5D health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. Higher scores indicated greater levels of problems across the five dimensions.
Time Frame: Baseline, Weeks 8, 16, 24, 40, 56 and 64
Population: as for outcome 40
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
Participants
  Baseline: number analyzed (Participants) | 1000 | 995 | 994
  Baseline: No problems washing or dressing | 251 | 242 | 270
  Baseline: Slight problems washing or dressing | 315 | 295 | 319
  Baseline: Moderate problems washing or dressing | 361 | 389 | 350
  Baseline: Severe problems washing or dressing | 73 | 69 | 55
  Baseline: Unable to wash or dress | 0 | 0 | 0
  Week 8: number analyzed (Participants) | 956 | 966 | 956
  Week 8: No problems washing or dressing | 551 | 569 | 542
  Week 8: Slight problems washing or dressing | 270 | 261 | 276
  Week 8: Moderate problems washing or dressing | 126 | 128 | 134
  Week 8: Severe problems washing or dressing | 8 | 8 | 3
  Week 8: Unable to wash or dress | 1 | 0 | 1
  Week 16: number analyzed (Participants) | 913 | 920 | 915
  Week 16: No problems washing or dressing | 610 | 597 | 583
  Week 16: Slight problems washing or dressing | 216 | 231 | 246
  Week 16: Moderate problems washing or dressing | 81 | 87 | 77
  Week 16: Severe problems washing or dressing | 6 | 5 | 9
  Week 16: Unable to wash or dress | 0 | 0 | 0
  Week 24: number analyzed (Participants) | 817 | 816 | 813
  Week 24: No problems washing or dressing | 504 | 504 | 527
  Week 24: Slight problems washing or dressing | 214 | 200 | 192
  Week 24: Moderate problems washing or dressing | 91 | 102 | 86
  Week 24: Severe problems washing or dressing | 7 | 9 | 8
  Week 24: Unable to wash or dress | 1 | 1 | 0
  Week 40: number analyzed (Participants) | 561 | 553 | 535
  Week 40: No problems washing or dressing | 377 | 359 | 371
  Week 40: Slight problems washing or dressing | 140 | 136 | 125
  Week 40: Moderate problems washing or dressing | 42 | 54 | 38
  Week 40: Severe problems washing or dressing | 1 | 4 | 1
  Week 40: Unable to wash or dress | 1 | 0 | 0
  Week 56: number analyzed (Participants) | 458 | 458 | 459
  Week 56: No problems washing or dressing | 305 | 294 | 291
  Week 56: Slight problems washing or dressing | 107 | 115 | 122
  Week 56: Moderate problems washing or dressing | 42 | 47 | 40
  Week 56: Severe problems washing or dressing | 3 | 2 | 5
  Week 56: Unable to wash or dress | 1 | 0 | 1
  Week 64: number analyzed (Participants) | 450 | 428 | 454
  Week 64: No problems washing or dressing | 233 | 192 | 264
  Week 64: Slight problems washing or dressing | 142 | 136 | 131
  Week 64: Moderate problems washing or dressing | 66 | 89 | 57
  Week 64: Severe problems washing or dressing | 8 | 11 | 2
  Week 64: Unable to wash or dress | 1 | 0 | 0

42. Secondary Outcome: Number of Participants With Responses to European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L): Usual Activities Domain
Description: Number of participants with usual activities domain responses of EQ-5D-5L were provided. EQ-5D-5L is a standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score. EQ-5D-5L consists of two components: a health state profile and an optional visual analogue scale (VAS). EQ-5D health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. Higher scores indicated greater levels of problems across the five dimensions.
Time Frame: Baseline, Weeks 8, 16, 24, 40, 56 and 64
Population: as for outcome 40
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
Participants
  Baseline: number analyzed (Participants) | 1000 | 995 | 994
  Baseline: No problems doing usual activities | 22 | 24 | 38
  Baseline: Slight problems doing usual activities | 229 | 218 | 225
  Baseline: Moderate problems doing usual activities | 538 | 551 | 561
  Baseline: Severe problems doing usual activities | 208 | 201 | 169
  Baseline: Unable to do usual activities | 3 | 1 | 1
  Week 8: number analyzed (Participants) | 956 | 966 | 956
  Week 8: No problems doing usual activities | 229 | 266 | 221
  Week 8: Slight problems doing usual activities | 402 | 411 | 426
  Week 8: Moderate problems doing usual activities | 292 | 256 | 274
  Week 8: Severe problems doing usual activities | 33 | 31 | 35
  Week 8: Unable to do usual activities | 0 | 2 | 0
  Week 16: number analyzed (Participants) | 913 | 920 | 915
  Week 16: No problems doing usual activities | 302 | 333 | 310
  Week 16: Slight problems doing usual activities | 402 | 382 | 408
  Week 16: Moderate problems doing usual activities | 184 | 182 | 172
  Week 16: Severe problems doing usual activities | 24 | 21 | 24
  Week 16: Unable to do usual activities | 1 | 2 | 1
  Week 24: number analyzed (Participants) | 817 | 816 | 813
  Week 24: No problems doing usual activities | 262 | 290 | 273
  Week 24: Slight problems doing usual activities | 353 | 315 | 344
  Week 24: Moderate problems doing usual activities | 174 | 182 | 166
  Week 24: Severe problems doing usual activities | 27 | 27 | 29
  Week 24: Unable to do usual activities | 1 | 2 | 1
  Week 40: number analyzed (Participants) | 561 | 553 | 535
  Week 40: No problems doing usual activities | 225 | 221 | 218
  Week 40: Slight problems doing usual activities | 239 | 213 | 233
  Week 40: Moderate problems doing usual activities | 85 | 97 | 74
  Week 40: Severe problems doing usual activities | 12 | 20 | 10
  Week 40: Unable to do usual activities | 0 | 2 | 0
  Week 56: number analyzed (Participants) | 458 | 458 | 459
  Week 56: No problems doing usual activities | 155 | 170 | 182
  Week 56: Slight problems doing usual activities | 211 | 179 | 199
  Week 56: Moderate problems doing usual activities | 79 | 86 | 69
  Week 56: Severe problems doing usual activities | 13 | 22 | 9
  Week 56: Unable to do usual activities | 0 | 1 | 0
  Week 64: number analyzed (Participants) | 450 | 428 | 454
  Week 64: No problems doing usual activities | 101 | 69 | 129
  Week 64: Slight problems doing usual activities | 173 | 163 | 197
  Week 64: Moderate problems doing usual activities | 138 | 155 | 115
  Week 64: Severe problems doing usual activities | 37 | 37 | 12
  Week 64: Unable to do usual activities | 1 | 4 | 1

43. Secondary Outcome: Number of Participants With Responses to European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L): Pain/Discomfort Domain
Description: Number of participants with pain/discomfort domain responses of EQ-5D-5L were provided. EQ-5D-5L is a standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score. EQ-5D-5L consists of two components: a health state profile and an optional visual analogue scale (VAS). EQ-5D health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. Higher scores indicated greater levels of problems across the five dimensions.
Time Frame: Baseline, Weeks 8, 16, 24, 40, 56 and 64
Population: as for outcome 40
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
Participants
  Baseline: number analyzed (Participants) | 1000 | 995 | 994
  Baseline: No pain or discomfort | 6 | 4 | 5
  Baseline: Slight pain or discomfort | 81 | 75 | 86
  Baseline: Moderate pain or discomfort | 548 | 574 | 588
  Baseline: Severe pain or discomfort | 334 | 314 | 295
  Baseline: Extreme pain or discomfort | 31 | 28 | 20
  Week 8: number analyzed (Participants) | 956 | 966 | 956
  Week 8: No pain or discomfort | 82 | 102 | 83
  Week 8: Slight pain or discomfort | 433 | 465 | 434
  Week 8: Moderate pain or discomfort | 369 | 327 | 365
  Week 8: Severe pain or discomfort | 68 | 68 | 71
  Week 8: Extreme pain or discomfort | 4 | 4 | 3
  Week 16: number analyzed (Participants) | 913 | 920 | 915
  Week 16: No pain or discomfort | 128 | 163 | 131
  Week 16: Slight pain or discomfort | 508 | 482 | 515
  Week 16: Moderate pain or discomfort | 235 | 225 | 217
  Week 16: Severe pain or discomfort | 39 | 44 | 46
  Week 16: Extreme pain or discomfort | 3 | 6 | 6
  Week 24: number analyzed (Participants) | 817 | 816 | 813
  Week 24: No pain or discomfort | 117 | 148 | 130
  Week 24: Slight pain or discomfort | 413 | 384 | 413
  Week 24: Moderate pain or discomfort | 213 | 218 | 215
  Week 24: Severe pain or discomfort | 70 | 62 | 51
  Week 24: Extreme pain or discomfort | 4 | 4 | 4
  Week 40: number analyzed (Participants) | 561 | 553 | 535
  Week 40: No pain or discomfort | 97 | 122 | 110
  Week 40: Slight pain or discomfort | 298 | 264 | 308
  Week 40: Moderate pain or discomfort | 139 | 130 | 104
  Week 40: Severe pain or discomfort | 25 | 30 | 13
  Week 40: Extreme pain or discomfort | 2 | 7 | 0
  Week 56: number analyzed (Participants) | 458 | 458 | 459
  Week 56: No pain or discomfort | 76 | 90 | 85
  Week 56: Slight pain or discomfort | 248 | 211 | 259
  Week 56: Moderate pain or discomfort | 111 | 128 | 103
  Week 56: Severe pain or discomfort | 23 | 26 | 9
  Week 56: Extreme pain or discomfort | 0 | 3 | 3
  Week 64: number analyzed (Participants) | 450 | 428 | 454
  Week 64: No pain or discomfort | 45 | 35 | 62
  Week 64: Slight pain or discomfort | 169 | 115 | 191
  Week 64: Moderate pain or discomfort | 165 | 191 | 171
  Week 64: Severe pain or discomfort | 66 | 76 | 29
  Week 64: Extreme pain or discomfort | 5 | 11 | 1

44. Secondary Outcome: Number of Participants With Responses to European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L): Anxiety/ Depression Domain
Description: Number of participants with anxiety/ depression domain responses of EQ-5D-5L were provided. EQ-5D-5L is a standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score. EQ-5D-5L consists of two components: a health state profile and an optional visual analogue scale (VAS). EQ-5D health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. Higher scores indicated greater levels of problems across the five dimensions.
Time Frame: Baseline, Weeks 8, 16, 24, 40, 56 and 64
Population: as for outcome 40
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
Participants
  Baseline: number analyzed (Participants) | 1000 | 995 | 994
  Baseline: Not anxious or depressed | 560 | 570 | 585
  Baseline: Slightly anxious or depressed | 252 | 235 | 236
  Baseline: Moderately anxious or depressed | 155 | 151 | 144
  Baseline: Severely anxious or depressed | 28 | 37 | 26
  Baseline: Extremely anxious or depressed | 5 | 2 | 3
  Week 8: number analyzed (Participants) | 956 | 966 | 956
  Week 8: Not anxious or depressed | 693 | 703 | 664
  Week 8: Slightly anxious or depressed | 189 | 180 | 206
  Week 8: Moderately anxious or depressed | 64 | 71 | 75
  Week 8: Severely anxious or depressed | 9 | 7 | 9
  Week 8: Extremely anxious or depressed | 1 | 5 | 2
  Week 16: number analyzed (Participants) | 913 | 920 | 915
  Week 16: Not anxious or depressed | 680 | 701 | 701
  Week 16: Slightly anxious or depressed | 170 | 147 | 151
  Week 16: Moderately anxious or depressed | 53 | 62 | 53
  Week 16: Severely anxious or depressed | 8 | 6 | 8
  Week 16: Extremely anxious or depressed | 2 | 4 | 2
  Week 24: number analyzed (Participants) | 817 | 816 | 813
  Week 24: Not anxious or depressed | 611 | 606 | 599
  Week 24: Slightly anxious or depressed | 147 | 131 | 144
  Week 24: Moderately anxious or depressed | 52 | 66 | 58
  Week 24: Severely anxious or depressed | 7 | 10 | 11
  Week 24: Extremely anxious or depressed | 0 | 3 | 1
  Week 40: number analyzed (Participants) | 561 | 553 | 535
  Week 40: Not anxious or depressed | 442 | 429 | 400
  Week 40: Slightly anxious or depressed | 92 | 82 | 107
  Week 40: Moderately anxious or depressed | 24 | 35 | 21
  Week 40: Severely anxious or depressed | 3 | 6 | 7
  Week 40: Extremely anxious or depressed | 0 | 1 | 0
  Week 56: number analyzed (Participants) | 458 | 458 | 459
  Week 56: Not anxious or depressed | 351 | 330 | 338
  Week 56: Slightly anxious or depressed | 88 | 90 | 86
  Week 56: Moderately anxious or depressed | 18 | 33 | 34
  Week 56: Severely anxious or depressed | 0 | 3 | 1
  Week 56: Extremely anxious or depressed | 1 | 2 | 0
  Week 64: number analyzed (Participants) | 450 | 428 | 454
  Week 64: Not anxious or depressed | 308 | 275 | 315
  Week 64: Slightly anxious or depressed | 104 | 96 | 100
  Week 64: Moderately anxious or depressed | 29 | 46 | 34
  Week 64: Severely anxious or depressed | 8 | 9 | 5
  Week 64: Extremely anxious or depressed | 1 | 2 | 0

45. Secondary Outcome: European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) Overall Health Utility Score/Index Value
Description: EQ-5D-5L: standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score. EQ-5D-5L consists of two components: a health state profile and an optional VAS. EQ-5D health state profile comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. Responses from the five domains were used to calculate a single utility index (the Overall health utility score) where values are less than or equal to (<=) 1. The Overall health utility score for a participant with no problems in all 5 items is 1 for all countries (except for Zimbabwe where it is 0.9), and is reduced where a participant reports greater levels of problems across the five dimensions.
Time Frame: Baseline, Weeks 8, 16, 24, 40, 56 and 64
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
units on a scale
  Baseline: number analyzed (Participants) | 992 | 985 | 980
  Baseline | 0.61 (0.14) | 0.61 (0.14) | 0.62 (0.13)
  Week 8: number analyzed (Participants) | 948 | 957 | 942
  Week 8 | 0.74 (0.12) | 0.75 (0.13) | 0.74 (0.13)
  Week 16: number analyzed (Participants) | 905 | 912 | 901
  Week 16 | 0.77 (0.12) | 0.78 (0.13) | 0.77 (0.13)
  Week 24: number analyzed (Participants) | 809 | 808 | 799
  Week 24 | 0.76 (0.14) | 0.76 (0.15) | 0.77 (0.14)
  Week 40: number analyzed (Participants) | 554 | 545 | 523
  Week 40 | 0.79 (0.13) | 0.78 (0.15) | 0.80 (0.12)
  Week 56: number analyzed (Participants) | 453 | 452 | 449
  Week 56 | 0.78 (0.12) | 0.77 (0.15) | 0.79 (0.12)
  Week 64: number analyzed (Participants) | 444 | 421 | 445
  Week 64 | 0.72 (0.15) | 0.69 (0.16) | 0.75 (0.13)

46. Secondary Outcome: Treatment Satisfaction Questionnaire Medicine Version II (TSQM v.II) Score With Effectiveness, Side Effects, Convenience, and Overall Satisfaction Responses
Description: TSQM v.II is a self-administered 11-item validated scale that quantified participant's level of satisfaction with study medication (scored on a 7-point Likert scale [1= extremely dissatisfied, 2=very dissatisfied, 3=dissatisfied, 4=somewhat satisfied, 5=satisfied, 6=very satisfied, 7=extremely satisfied]) and dissatisfaction with side effects (3 questions scored on 5 point Likert scale [1= extremely dissatisfied, 2=very dissatisfied, 3=somewhat dissatisfied, 4=slightly dissatisfied, 5=not at all dissatisfied] and 1 question on 2 point scale [0 =No, 1=Yes]). Participants were asked to assess their level of satisfaction taking all things into account. The 11 questions of the TSQM were used to calculate the 4 endpoints of effectiveness, side Effects, convenience and global satisfaction, each scored on a 0-100 scale with 100 being the best level of satisfaction.
Time Frame: Weeks 16 and 56
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either Tanezumab or matching placebo). Here 'Overall number of participants analyzed'=participants evaluable for this outcome measure. Here, "Number analyzed" =participants who were evaluable at specified time point for each arm, respectively.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 939 | 954 | 936
units on a scale
  Week 16: Effectiveness | 64.26 (1.03) | 66.27 (1.02) | 61.61 (1.03)
  Week 16: Side Effects: number analyzed (Participants) | 86 | 94 | 84
  Week 16: Side Effects | 68.61 (3.20) | 73.32 (3.09) | 71.03 (3.15)
  Week 16: Convenience | 75.50 (0.80) | 75.78 (0.79) | 73.70 (0.80)
  Week 16: Global Satisfaction | 70.32 (0.99) | 70.69 (0.98) | 67.13 (0.99)
  Week 56: Effectiveness: number analyzed (Participants) | 498 | 487 | 489
  Week 56: Effectiveness | 69.79 (1.38) | 67.91 (1.36) | 67.64 (1.38)
  Week 56: Side Effects: number analyzed (Participants) | 30 | 38 | 24
  Week 56: Side Effects | 78.62 (5.28) | 62.00 (4.88) | 71.34 (5.14)
  Week 56: Convenience: number analyzed (Participants) | 498 | 487 | 489
  Week 56: Convenience | 78.03 (1.12) | 77.67 (1.10) | 76.18 (1.11)
  Week 56: Global Satisfaction: number analyzed (Participants) | 498 | 487 | 489
  Week 56: Global Satisfaction | 75.31 (1.27) | 73.37 (1.25) | 73.37 (1.26)
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; TSQM Effectiveness; Week 16: ANCOVA model included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0142, ANCOVA; LS Mean Difference = 2.66, 95% CI 2-sided [0.53 to 4.78], Standard Error of Mean 1.08
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 46, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = 4.67, 95% CI 2-sided [2.56 to 6.78], Standard Error of Mean 1.08
Statistical Analysis 3: Comparison: Tanezumab 2.5 mg vs NSAID; TSQM Effectiveness; Week 56: ANCOVA model included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.1371, ANCOVA; LS Mean Difference = 2.15, 95% CI 2-sided [-0.69 to 4.99], Standard Error of Mean 1.45
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 46, analysis 3]; Test type: Superiority; p = 0.8524, ANCOVA; LS Mean Difference = 0.27, 95% CI 2-sided [-2.60 to 3.14], Standard Error of Mean 1.46
Statistical Analysis 5: Comparison: Tanezumab 2.5 mg vs NSAID; TSQM Side Effects; Week 16: ANCOVA model included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.5253, ANCOVA; LS Mean Difference = -2.42, 95% CI 2-sided [-9.93 to 5.09], Standard Error of Mean 3.80
Statistical Analysis 6: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 46, analysis 5]; Test type: Superiority; p = 0.5381, ANCOVA; LS Mean Difference = 2.29, 95% CI 2-sided [-5.04 to 9.62], Standard Error of Mean 3.71
Statistical Analysis 7: Comparison: Tanezumab 2.5 mg vs NSAID; TSQM Side Effects; Week 56: ANCOVA model included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.2694, ANCOVA; LS Mean Difference = 7.27, 95% CI 2-sided [-5.99 to 20.54], Standard Error of Mean 6.44
Statistical Analysis 8: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 46, analysis 7]; Test type: Superiority; p = 0.1349, ANCOVA; LS Mean Difference = -9.34, 95% CI 2-sided [-21.80 to 3.11], Standard Error of Mean 6.05
Statistical Analysis 9: Comparison: Tanezumab 2.5 mg vs NSAID; TSQM Convenience; Week 16: ANCOVA model included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0264, ANCOVA; LS Mean Difference = 1.80, 95% CI 2-sided [0.21 to 3.38], Standard Error of Mean 0.81
Statistical Analysis 10: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 46, analysis 9]; Test type: Superiority; p = 0.0098, ANCOVA; LS Mean Difference = 2.07, 95% CI 2-sided [0.50 to 3.65], Standard Error of Mean 0.80
Statistical Analysis 11: Comparison: Tanezumab 2.5 mg vs NSAID; TSQM Convenience; Week 56: ANCOVA model included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0937, ANCOVA; LS Mean Difference = 1.85, 95% CI 2-sided [-0.31 to 4.01], Standard Error of Mean 1.10
Statistical Analysis 12: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 46, analysis 11]; Test type: Superiority; p = 0.1838, ANCOVA; LS Mean Difference = 1.48, 95% CI 2-sided [-0.70 to 3.67], Standard Error of Mean 1.11
Statistical Analysis 13: Comparison: Tanezumab 2.5 mg vs NSAID; TSQM Global Satisfaction; Week 16: ANCOVA model included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0025, ANCOVA; LS Mean Difference = 3.18, 95% CI 2-sided [1.12 to 5.25], Standard Error of Mean 1.05
Statistical Analysis 14: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 46, analysis 13]; Test type: Superiority; p = 0.0007, ANCOVA; LS Mean Difference = 3.55, 95% CI 2-sided [1.51 to 5.60], Standard Error of Mean 1.04
Statistical Analysis 15: Comparison: Tanezumab 2.5 mg vs NSAID; TSQM Global Satisfaction; Week 56: ANCOVA model included treatment, randomization stratification variables (index joint, highest Kellgren-Lawrence grade and NSAID) as fixed effects, baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.1373, ANCOVA; LS Mean Difference = 1.94, 95% CI 2-sided [-0.62 to 4.51], Standard Error of Mean 1.31
Statistical Analysis 16: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 46, analysis 15]; Test type: Superiority; p = 0.9960, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-2.59 to 2.60], Standard Error of Mean 1.32

47. Secondary Outcome: Patient-Reported Treatment Impact Assessment- Modified (mPRTI) Score at Weeks 16 and 56: Participant Global Preference Assessment- What is The Current or Most Recent Treatment You Were Receiving for Osteoarthritis Pain Before Enrolling?
Description: The mPRTI is a self-administered questionnaire containing participant's global preference assessment (to assess previous treatment and preference to continue using the investigational product) and participant's willingness to use drug again assessment. To assess current or most recent treatment, participants responded for, 1=injectable prescription medicines, 2=prescription medicines taken by mouth, 3=surgery, 4=prescription medicines and surgery and 5=no treatment. Number of participants who responded for the specified question were reported.
Time Frame: Weeks 16 and 56
Population: as for outcome 40
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
Participants
  Week 16: number analyzed (Participants) | 939 | 954 | 936
  Week 16: Injectable prescription medicines | 99 | 98 | 82
  Week 16: Prescription medicines taken by mouth | 611 | 633 | 647
  Week 16: Surgery | 7 | 7 | 9
  Week 16: Prescription medicines and surgery | 33 | 28 | 27
  Week 16: No treatment | 189 | 188 | 171
  Week 56: number analyzed (Participants) | 498 | 487 | 489
  Week 56: Injectable prescription medicines | 44 | 47 | 40
  Week 56: Prescription medicines taken by mouth | 307 | 296 | 324
  Week 56: Surgery | 8 | 4 | 2
  Week 56: Prescription medicines and surgery | 20 | 18 | 20
  Week 56: No treatment | 119 | 122 | 103

48. Secondary Outcome: Patient Reported Treatment Impact Assessment-Modified (mPRTI) Score at Weeks 16 and 56: Participant Global Preference Assessment- Overall, do You Prefer the Drug That You Received in This Study to Previous Treatment?
Description: The mPRTI is a self-administered questionnaire containing participant global preference assessment (to assess previous treatment and preference to continue using the investigational product) and participant willingness to use drug again assessment. To assess preference to continue using the investigational product, participants responded using IRT on a 5 point Likert scale from 1-5, where, 1= yes, I definitely prefer the drug that I am receiving now, 2= I have a slight preference for the drug that I am receiving now, 3= I have no preference either way, 4= I have a slight preference for my previous treatment, 5= No, I definitely prefer my previous treatment. Higher scores indicate lesser preference to use the investigational product. Number of participants who responded for the specified question were reported.
Time Frame: Weeks 16 and 56
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either Tanezumab or matching placebo). Here, "Number analyzed" = participants who were evaluable at specified time point for each arm, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
Participants
  Week 16: number analyzed (Participants) | 939 | 954 | 936
  Week 16: Yes, definitely prefer the study drug | 577 | 597 | 531
  Week 16: Slight preference for the study drug | 141 | 169 | 158
  Week 16: No preference either way | 149 | 114 | 164
  Week 16: Slight preference for my previous treatment | 28 | 34 | 36
  Week 16: No, definitely prefer my previous treatment | 44 | 40 | 47
  Week 56: number analyzed (Participants) | 498 | 487 | 489
  Week 56: Yes, definitely prefer the study drug | 342 | 323 | 302
  Week 56: Slight preference for the study drug | 70 | 75 | 89
  Week 56: No preference either way | 61 | 65 | 71
  Week 56: Slight preference for my previous treatment | 16 | 16 | 13
  Week 56: No, definitely prefer my previous treatment | 9 | 8 | 14
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Week 16: Cochran-Mantel-Haenszel test for row mean scores differ, stratified by the combinations of the three stratification factors (index joint, highest Kellgren-Lawrence grade and NSAID); Test type: Superiority; p = 0.0823, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 48, analysis 1]; Test type: Superiority; p = 0.0049, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Tanezumab 2.5 mg vs NSAID; Week 56: Cochran-Mantel-Haenszel test for row mean scores differ, stratified by the combinations of the three stratification factors (index joint, highest Kellgren-Lawrence grade and NSAID); Test type: Superiority; p = 0.0718, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 48, analysis 3]; Test type: Superiority; p = 0.1947, Cochran-Mantel-Haenszel

49. Secondary Outcome: Patient Reported Treatment Impact Assessment-Modified (mPRTI) Score at Weeks 16 and 56: Participant Willingness to Use Drug Again Assessment- Willing to Use the Same Drug That You Have Received in This Study for Your Osteoarthritis Pain?
Description: The mPRTI is a self-administered questionnaire containing participant global preference assessment (to assess previous treatment and preference to continue using the investigational product) and participant willingness to use drug again assessment. To assess participant willingness to use drug again, participants responded using IRT on a 5 point likert scale from 1-5, where, 1= yes, I would definitely want to use the same drug again, 2= I might want to use the same drug again, 3= I am not sure, 4= I might not want to use the same drug again, 5= no, I definitely would not want to use the same drug again. Higher scores indicate lesser willingness to use the investigational product. Number of participants who responded for the specified question were reported.
Time Frame: Weeks 16 and 56
Population: as for outcome 48
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
Participants
  Week 16: number analyzed (Participants) | 939 | 954 | 936
  Week 16: Yes, definitely want to use the same drug again | 627 | 641 | 560
  Week 16: Might want to use the same drug again | 138 | 154 | 169
  Week 16: I am not sure | 108 | 96 | 134
  Week 16: Might not want to use the same drug again | 19 | 21 | 23
  Week 16: No:definitely wouldn't want to use same drug again | 47 | 42 | 50
  Week 56: number analyzed (Participants) | 498 | 487 | 489
  Week 56: Yes, definitely want to use the same drug again | 352 | 341 | 310
  Week 56: Might want to use the same drug again | 78 | 75 | 97
  Week 56: I am not sure | 54 | 46 | 58
  Week 56: Might not want to use the same drug again | 4 | 11 | 12
  Week 56: No:definitely wouldn't want to use same drug again | 10 | 14 | 12
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; [analysis description as in outcome 48, analysis 1]; Test type: Superiority; p = 0.0229, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 48, analysis 1]; Test type: Superiority; p = 0.0029, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Tanezumab 2.5 mg vs NSAID; [analysis description as in outcome 48, analysis 3]; Test type: Superiority; p = 0.0266, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 48, analysis 3]; Test type: Superiority; p = 0.1835, Cochran-Mantel-Haenszel

50. Secondary Outcome: Number of Participants Who Withdrew Due to Lack of Efficacy
Description: Number of participants who withdrew from treatment due to lack of efficacy have been reported here.
Time Frame: Baseline up to Week 56
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
Participants | 60 | 63 | 91
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline diary average pain, baseline WOMAC pain score, classification variables index joint, highest Kellgren-Lawrence grade, NSAID and treatment; Test type: Superiority; p = 0.0076, Regression, Logistic; Odds Ratio (OR) = 0.63, 95% CI 2-sided [0.45 to 0.88]
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 50, analysis 1]; Test type: Superiority; p = 0.0187, Regression, Logistic; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.48 to 0.94]

51. Secondary Outcome: Time to Discontinuation Due to Lack of Efficacy
Description: Time to discontinuation due to lack of efficacy was defined as the time interval from the date of first study drug administration up to the date of discontinuation of participant from treatment due to lack of efficacy.
Time Frame: Baseline up to Week 56
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or matching placebo). Here, 'Overall number of participants analyzed' signifies participants who discontinued from the study due to lack of efficacy.
Measure: Median (Full Range); unit: days
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 60 | 63 | 91
days | NA [7 to NA] — Due to the Kaplan-Meier estimate not reaching the level for discontinuation due to lack of efficacy, median and upper limit could not be calculated. | NA [14 to NA] — Due to the Kaplan-Meier estimate not reaching the level for discontinuation due to lack of efficacy, median and upper limit could not be calculated. | NA [14 to NA] — Due to the Kaplan-Meier estimate not reaching the level for discontinuation due to lack of efficacy, median and upper limit could not be calculated.
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Missing data for the selected percentile(s) was due to the Kaplan-Meier estimate not reaching the level for discontinuation due to lack of efficacy; Test type: Superiority; p = 0.0074, Log Rank
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 51, analysis 1]; Test type: Superiority; p = 0.0162, Log Rank

52. Secondary Outcome: Number of Participants Who Took Rescue Medication During Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56
Description: In case of inadequate pain relief, acetaminophen/paracetamol up to 3000 mg per day and up to 3 days in a week between baseline and Week 16, and 3000 mg per day and up to 7 days per week between Week 16 and 64 could be taken as rescue medication. Number of participants with any use of rescue medication during the particular study week were summarized.
Time Frame: Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
Participants
  Week 2: number analyzed (Participants) | 998 | 994 | 993
  Week 2 | 567 | 548 | 527
  Week 4: number analyzed (Participants) | 1002 | 995 | 995
  Week 4 | 481 | 437 | 469
  Week 8 | 433 | 377 | 418
  Week 16 | 353 | 330 | 352
  Week 24 | 372 | 358 | 384
  Week 32 | 391 | 380 | 390
  Week 40 | 391 | 388 | 388
  Week 48 | 391 | 393 | 389
  Week 56 | 391 | 408 | 397
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Week 2: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade, NSAID and treatment; Test type: Superiority; p = 0.1136, Regression, Logistic; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.97 to 1.38]
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 52, analysis 1]; Test type: Superiority; p = 0.3910, Regression, Logistic; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.90 to 1.29]
Statistical Analysis 3: Comparison: Tanezumab 2.5 mg vs NSAID; Week 4: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade, NSAID and treatment; Test type: Superiority; p = 0.7691, Regression, Logistic; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.86 to 1.22]
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 52, analysis 3]; Test type: Superiority; p = 0.1430, Regression, Logistic; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.73 to 1.05]
Statistical Analysis 5: Comparison: Tanezumab 2.5 mg vs NSAID; Week 8: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade, NSAID and treatment; Test type: Superiority; p = 0.6454, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.87 to 1.25]
Statistical Analysis 6: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 52, analysis 5]; Test type: Superiority; p = 0.0561, Regression, Logistic; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.70 to 1.00]
Statistical Analysis 7: Comparison: Tanezumab 2.5 mg vs NSAID; Week 16: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade, NSAID and treatment; Test type: Superiority; p = 0.9056, Regression, Logistic; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.82 to 1.19]
Statistical Analysis 8: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 52, analysis 7]; Test type: Superiority; p = 0.2919, Regression, Logistic; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.75 to 1.09]
Statistical Analysis 9: Comparison: Tanezumab 2.5 mg vs NSAID; Week 24: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade, NSAID and treatment; Test type: Superiority; p = 0.4976, Regression, Logistic; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.78 to 1.13]
Statistical Analysis 10: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 52, analysis 9]; Test type: Superiority; p = 0.2425, Regression, Logistic; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.75 to 1.08]
Statistical Analysis 11: Comparison: Tanezumab 2.5 mg vs NSAID; Week 32: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade, NSAID and treatment; Test type: Superiority; p = 0.9242, Regression, Logistic; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.83 to 1.19]
Statistical Analysis 12: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 52, analysis 11]; Test type: Superiority; p = 0.6621, Regression, Logistic; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.80 to 1.15]
Statistical Analysis 13: Comparison: Tanezumab 2.5 mg vs NSAID; Week 40: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade, NSAID and treatment; Test type: Superiority; p = 0.9977, Regression, Logistic; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.83 to 1.20]
Statistical Analysis 14: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 52, analysis 13]; Test type: Superiority; p = 0.9762, Regression, Logistic; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.84 to 1.20]
Statistical Analysis 15: Comparison: Tanezumab 2.5 mg vs NSAID; Week 48: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade, NSAID and treatment; Test type: Superiority; p = 0.9718, Regression, Logistic; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.83 to 1.19]
Statistical Analysis 16: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 52, analysis 15]; Test type: Superiority; p = 0.8219, Regression, Logistic; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.85 to 1.22]
Statistical Analysis 17: Comparison: Tanezumab 2.5 mg vs NSAID; Week 56: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade, NSAID and treatment; Test type: Superiority; p = 0.6936, Regression, Logistic; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.80 to 1.16]
Statistical Analysis 18: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 52, analysis 17]; Test type: Superiority; p = 0.5769, Regression, Logistic; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.88 to 1.26]

53. Secondary Outcome: Number of Participants Who Took Rescue Medication During Week 64
Description: In case of inadequate pain relief, after Week 16, acetaminophen/paracetamol up to 3000 mg per day up to 7 days in a week could be taken as rescue medication and use was reported weekly via diary. Number of participants with any use of rescue medication during Week 64 were summarized.
Time Frame: Week 64
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 437 | 417 | 437
Participants | 251 | 268 | 215

54. Secondary Outcome: Number of Days of Rescue Medication Used During Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56
Description: In case of inadequate pain relief during the treatment period, acetaminophen/paracetamol up to 3000 mg per day and up to 3 days in a week between baseline and Week 16, and 3000 mg per day and up to 7 days per week between Week 16 and 64 could be taken as rescue medication. Number of days the participants used the rescue medication during the particular study weeks were summarized.
Time Frame: Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
days
  Week 2 | 2.31 (0.13) | 2.29 (0.13) | 2.26 (0.13)
  Week 4 | 1.80 (0.12) | 1.70 (0.11) | 1.86 (0.12)
  Week 8 | 1.65 (0.12) | 1.42 (0.11) | 1.65 (0.12)
  Week 16 | 1.29 (0.11) | 1.25 (0.10) | 1.39 (0.11)
  Week 24 | 1.56 (0.12) | 1.56 (0.13) | 1.65 (0.13)
  Week 32 | 1.67 (0.13) | 1.66 (0.13) | 1.78 (0.13)
  Week 40 | 1.70 (0.13) | 1.71 (0.13) | 1.76 (0.13)
  Week 48 | 1.68 (0.13) | 1.76 (0.14) | 1.74 (0.13)
  Week 56 | 1.73 (0.13) | 1.85 (0.14) | 1.74 (0.13)
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Week 2: Analysis was performed using negative binomial model with model terms of baseline WOMAC Pain subscale score, baseline diary average pain score, index joint, Kellgren Lawrence grade, NSAID and treatment group; Test type: Superiority; p = 0.7746, Negative binomial model; LS Mean Ratio = 1.02, 95% CI 2-sided [0.89 to 1.16], Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 54, analysis 1]; Test type: Superiority; p = 0.8441, Negative binomial model; LS Mean Ratio = 1.01, 95% CI 2-sided [0.89 to 1.16], Standard Error of Mean 0.07
Statistical Analysis 3: Comparison: Tanezumab 2.5 mg vs NSAID; Week 4: Analysis was performed using negative binomial model with model terms of baseline WOMAC Pain subscale score, baseline diary average pain score, index joint, Kellgren Lawrence grade, NSAID and treatment group; Test type: Superiority; p = 0.6580, Negative binomial model; LS Mean Ratio = 0.97, 95% CI 2-sided [0.83 to 1.13], Standard Error of Mean 0.08
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 54, analysis 3]; Test type: Superiority; p = 0.2279, Negative binomial model; LS Mean Ratio = 0.91, 95% CI 2-sided [0.78 to 1.06], Standard Error of Mean 0.07
Statistical Analysis 5: Comparison: Tanezumab 2.5 mg vs NSAID; Week 8: Analysis was performed using negative binomial model with model terms of baseline WOMAC Pain subscale score, baseline diary average pain score, index joint, Kellgren Lawrence grade, NSAID and treatment group; Test type: Superiority; p = 0.9986, Negative binomial model; LS Mean Ratio = 1.00, 95% CI 2-sided [0.84 to 1.18], Standard Error of Mean 0.09
Statistical Analysis 6: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 54, analysis 5]; Test type: Superiority; p = 0.0771, Negative binomial model; LS Mean Ratio = 0.86, 95% CI 2-sided [0.72 to 1.02], Standard Error of Mean 0.07
Statistical Analysis 7: Comparison: Tanezumab 2.5 mg vs NSAID; Week 16: Analysis was performed using negative binomial model with model terms of baseline WOMAC Pain subscale score, baseline diary average pain score, index joint, Kellgren Lawrence grade, NSAID and treatment group; Test type: Superiority; p = 0.4485, Negative binomial model; LS Mean Ratio = 0.93, 95% CI 2-sided [0.77 to 1.13], Standard Error of Mean 0.09
Statistical Analysis 8: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 54, analysis 7]; Test type: Superiority; p = 0.2817, Negative binomial model; LS Mean Ratio = 0.90, 95% CI 2-sided [0.74 to 1.09], Standard Error of Mean 0.09
Statistical Analysis 9: Comparison: Tanezumab 2.5 mg vs NSAID; Week 24: Analysis was performed using negative binomial model with model terms of baseline WOMAC Pain subscale score, baseline diary average pain score, index joint, Kellgren Lawrence grade, NSAID and treatment group; Test type: Superiority; p = 0.5426, Negative binomial model; LS Mean Ratio = 0.94, 95% CI 2-sided [0.79 to 1.13], Standard Error of Mean 0.09
Statistical Analysis 10: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 54, analysis 9]; Test type: Superiority; p = 0.5385, Negative binomial model; LS Mean Ratio = 0.94, 95% CI 2-sided [0.79 to 1.13], Standard Error of Mean 0.09
Statistical Analysis 11: Comparison: Tanezumab 2.5 mg vs NSAID; Week 32: Analysis was performed using negative binomial model with model terms of baseline WOMAC Pain subscale score, baseline diary average pain score, index joint, Kellgren Lawrence grade, NSAID and treatment group; Test type: Superiority; p = 0.5041, Negative binomial model; LS Mean Ratio = 0.94, 95% CI 2-sided [0.79 to 1.12], Standard Error of Mean 0.09
Statistical Analysis 12: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 54, analysis 11]; Test type: Superiority; p = 0.4410, Negative binomial model; LS Mean Ratio = 0.93, 95% CI 2-sided [0.78 to 1.11], Standard Error of Mean 0.08
Statistical Analysis 13: Comparison: Tanezumab 2.5 mg vs NSAID; Week 40: Analysis was performed using negative binomial model with model terms of baseline WOMAC Pain subscale score, baseline diary average pain score, index joint, Kellgren Lawrence grade, NSAID and treatment group; Test type: Superiority; p = 0.7426, Negative binomial model; LS Mean Ratio = 0.97, 95% CI 2-sided [0.81 to 1.16], Standard Error of Mean 0.09
Statistical Analysis 14: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 54, analysis 13]; Test type: Superiority; p = 0.7469, Negative binomial model; LS Mean Ratio = 0.97, 95% CI 2-sided [0.81 to 1.16], Standard Error of Mean 0.09
Statistical Analysis 15: Comparison: Tanezumab 2.5 mg vs NSAID; Week 48: Analysis was performed using negative binomial model with model terms of baseline WOMAC Pain subscale score, baseline diary average pain score, index joint, Kellgren Lawrence grade, NSAID and treatment group; Test type: Superiority; p = 0.6784, Negative binomial model; LS Mean Ratio = 0.96, 95% CI 2-sided [0.81 to 1.15], Standard Error of Mean 0.09
Statistical Analysis 16: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 54, analysis 15]; Test type: Superiority; p = 0.8822, Negative binomial model; LS Mean Ratio = 1.01, 95% CI 2-sided [0.85 to 1.21], Standard Error of Mean 0.09
Statistical Analysis 17: Comparison: Tanezumab 2.5 mg vs NSAID; Week 56: Analysis was performed using negative binomial model with model terms of baseline WOMAC Pain subscale score, baseline diary average pain score, index joint, Kellgren Lawrence grade, NSAID and treatment group; Test type: Superiority; p = 0.9119, Negative binomial model; LS Mean Ratio = 0.99, 95% CI 2-sided [0.83 to 1.18], Standard Error of Mean 0.09
Statistical Analysis 18: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 54, analysis 17]; Test type: Superiority; p = 0.5148, Negative binomial model; LS Mean Ratio = 1.06, 95% CI 2-sided [0.89 to 1.26], Standard Error of Mean 0.09

55. Secondary Outcome: Number of Days of Rescue Medication Used During Week 64
Description: In case of inadequate pain relief, after week 16, acetaminophen/paracetamol up to 3000 mg per day up to 7 days in a week could be taken as rescue medication and use was reported weekly via diary. Number of days the participants used the rescue medication during Week 64 were summarized.
Time Frame: Week 64
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or matching placebo). Here 'Overall number of participants analyzed' = participants who took rescue medication.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 437 | 417 | 437
days | 2.0 (2.38) | 2.3 (2.46) | 1.7 (2.26)

56. Secondary Outcome: Amount of Rescue Medication Used During Weeks 2, 4, 8 and 16
Description: In case of inadequate pain relief, acetaminophen/paracetamol up to 3000 mg per day up to 3 days in a week could be taken as rescue medication. The total dosage of acetaminophen in milligrams used during the specified week were summarized.
Time Frame: Weeks 2, 4, 8 and 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: milligrams
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
milligrams
  Week 2 | 2880.3 (353.05) | 2898.7 (358.72) | 3310.5 (410.42)
  Week 4 | 2107.8 (302.24) | 1946.5 (277.29) | 2814.1 (401.29)
  Week 8 | 1995.6 (322.53) | 1628.8 (258.90) | 2839.7 (446.00)
  Week 16 | 1696.4 (307.80) | 1581.6 (284.12) | 2320.0 (413.14)
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; [analysis description as in outcome 54, analysis 1]; Test type: Superiority; p = 0.3348, Negative binomial model; LS Mean Ratio = 0.87, 95% CI 2-sided [0.66 to 1.15], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 54, analysis 1]; Test type: Superiority; p = 0.3595, Negative binomial model; LS Mean Ratio = 0.88, 95% CI 2-sided [0.66 to 1.16], Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: Tanezumab 2.5 mg vs NSAID; [analysis description as in outcome 54, analysis 3]; Test type: Superiority; p = 0.0854, Negative binomial model; LS Mean Ratio = 0.75, 95% CI 2-sided [0.54 to 1.04], Standard Error of Mean 0.13
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 54, analysis 3]; Test type: Superiority; p = 0.0281, Negative binomial model; LS Mean Ratio = 0.69, 95% CI 2-sided [0.50 to 0.96], Standard Error of Mean 0.12
Statistical Analysis 5: Comparison: Tanezumab 2.5 mg vs NSAID; [analysis description as in outcome 54, analysis 5]; Test type: Superiority; p = 0.0595, Negative binomial model; LS Mean Ratio = 0.70, 95% CI 2-sided [0.49 to 1.01], Standard Error of Mean 0.13
Statistical Analysis 6: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 54, analysis 5]; Test type: Superiority; p = 0.0030, Negative binomial model; LS Mean Ratio = 0.57, 95% CI 2-sided [0.40 to 0.83], Standard Error of Mean 0.11
Statistical Analysis 7: Comparison: Tanezumab 2.5 mg vs NSAID; [analysis description as in outcome 54, analysis 7]; Test type: Superiority; p = 0.1389, Negative binomial model; LS Mean Ratio = 0.73, 95% CI 2-sided [0.48 to 1.11], Standard Error of Mean 0.15
Statistical Analysis 8: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 54, analysis 7]; Test type: Superiority; p = 0.0709, Negative binomial model; LS Mean Ratio = 0.68, 95% CI 2-sided [0.45 to 1.03], Standard Error of Mean 0.14

57. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Visits of Services Directly Related to Osteoarthritis
Description: OA HCRU assessed healthcare usage during the last 3 months (for Baseline and Week 80) and past 8 weeks (for Week 64). Visits of services directly related to OA evaluated were: visits to primary care physician, neurologist, rheumatologist, physician assistant or nurse practitioner, pain specialist, orthopedist, physical therapist, chiropractor, alternative medicine or therapy, podiatrist, nutritionist/dietitian, radiologist, home healthcare services and other practitioner.
Time Frame: Baseline, Weeks 64 and 80
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or matching placebo). Here, "Number analyzed" signifies those participants who were evaluable at specified time point for this outcome measure for each arm, respectively.
Measure: Median (Full Range); unit: visits
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
visits
  Baseline: Primary Care Physician: number analyzed (Participants) | 442 | 433 | 436
  Baseline: Primary Care Physician | 1.0 [1.0 to 100.0] | 1.0 [1.0 to 101.0] | 1.0 [1.0 to 150.0]
  Baseline: Neurologist: number analyzed (Participants) | 10 | 15 | 12
  Baseline: Neurologist | 1.0 [1.0 to 120.0] | 1.0 [1.0 to 90.0] | 1.0 [1.0 to 10.0]
  Baseline: Rheumatologist: number analyzed (Participants) | 83 | 108 | 114
  Baseline: Rheumatologist | 1.0 [1.0 to 15.0] | 2.0 [1.0 to 111.0] | 2.0 [1.0 to 6.0]
  Baseline:Physician Assistant or Nurse Practitioner: number analyzed (Participants) | 35 | 38 | 30
  Baseline:Physician Assistant or Nurse Practitioner | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 122.0] | 1.0 [1.0 to 120.0]
  Baseline: Pain Specialist: number analyzed (Participants) | 42 | 51 | 41
  Baseline: Pain Specialist | 1.0 [1.0 to 100.0] | 2.0 [1.0 to 111.0] | 1.0 [1.0 to 23.0]
  Baseline: Orthopedist: number analyzed (Participants) | 171 | 189 | 160
  Baseline: Orthopedist | 2.0 [1.0 to 18.0] | 1.0 [1.0 to 190.0] | 2.0 [1.0 to 100.0]
  Baseline: Physical Therapist: number analyzed (Participants) | 57 | 62 | 51
  Baseline: Physical Therapist | 4.0 [1.0 to 100.0] | 3.0 [1.0 to 111.0] | 3.0 [1.0 to 32.0]
  Baseline: Chiropractor: number analyzed (Participants) | 48 | 33 | 43
  Baseline: Chiropractor | 3.0 [1.0 to 190.0] | 3.0 [1.0 to 30.0] | 3.0 [1.0 to 24.0]
  Baseline: Alternative Medicine or Therapy: number analyzed (Participants) | 33 | 50 | 52
  Baseline: Alternative Medicine or Therapy | 2.0 [1.0 to 24.0] | 2.0 [1.0 to 111.0] | 2.0 [1.0 to 80.0]
  Baseline: Podiatrist: number analyzed (Participants) | 10 | 20 | 13
  Baseline: Podiatrist | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 91.0] | 1.0 [1.0 to 2.0]
  Baseline: Nutritionist/Dietitian: number analyzed (Participants) | 8 | 11 | 14
  Baseline: Nutritionist/Dietitian | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 4.0]
  Baseline: Radiologist: number analyzed (Participants) | 139 | 152 | 138
  Baseline: Radiologist | 1.0 [1.0 to 100.0] | 1.0 [1.0 to 111.0] | 1.0 [1.0 to 5.0]
  Baseline: Home Healthcare Services: number analyzed (Participants) | 7 | 5 | 7
  Baseline: Home Healthcare Services | 2.0 [1.0 to 24.0] | 1.0 [1.0 to 111.0] | 3.0 [1.0 to 91.0]
  Baseline: Other Practitioner: number analyzed (Participants) | 82 | 98 | 91
  Baseline: Other Practitioner | 2.0 [1.0 to 190.0] | 2.0 [1.0 to 111.0] | 2.0 [1.0 to 111.0]
  Week 64: Primary Care Physician: number analyzed (Participants) | 231 | 264 | 223
  Week 64: Primary Care Physician | 1.0 [1.0 to 190.0] | 1.0 [1.0 to 101.0] | 1.0 [1.0 to 120.0]
  Week 64: Neurologist: number analyzed (Participants) | 17 | 20 | 13
  Week 64: Neurologist | 1.0 [1.0 to 110.0] | 1.0 [1.0 to 4.0] | 1.0 [1.0 to 83.0]
  Week 64: Rheumatologist: number analyzed (Participants) | 27 | 32 | 35
  Week 64: Rheumatologist | 1.0 [1.0 to 4.0] | 1.0 [1.0 to 4.0] | 1.0 [1.0 to 3.0]
  Week 64: Physician Assistant Or Nurse Practitioner: number analyzed (Participants) | 30 | 36 | 27
  Week 64: Physician Assistant Or Nurse Practitioner | 1.0 [1.0 to 10.0] | 1.0 [1.0 to 100.0] | 2.0 [1.0 to 101.0]
  Week 64: Pain Specialist: number analyzed (Participants) | 37 | 43 | 29
  Week 64: Pain Specialist | 1.0 [1.0 to 190.0] | 1.0 [1.0 to 144.0] | 1.0 [1.0 to 180.0]
  Week 64: Orthopedist: number analyzed (Participants) | 146 | 163 | 121
  Week 64: Orthopedist | 1.0 [1.0 to 190.0] | 1.0 [1.0 to 30.0] | 1.0 [1.0 to 100.0]
  Week 64: Physical Therapist: number analyzed (Participants) | 69 | 50 | 37
  Week 64: Physical Therapist | 4.0 [1.0 to 180.0] | 4.5 [1.0 to 111.0] | 3.0 [1.0 to 100.0]
  Week 64: Chiropractor: number analyzed (Participants) | 32 | 25 | 22
  Week 64: Chiropractor | 3.0 [1.0 to 21.0] | 2.0 [1.0 to 30.0] | 3.0 [1.0 to 111.0]
  Week 64: Alternative Medicine or Therapy: number analyzed (Participants) | 33 | 45 | 46
  Week 64: Alternative Medicine or Therapy | 1.0 [1.0 to 11.0] | 2.0 [1.0 to 10.0] | 2.0 [1.0 to 190.0]
  Week 64: Podiatrist: number analyzed (Participants) | 11 | 18 | 12
  Week 64: Podiatrist | 1.0 [1.0 to 5.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0]
  Week 64: Nutritionist/Dietitian: number analyzed (Participants) | 9 | 8 | 6
  Week 64: Nutritionist/Dietitian | 2.0 [1.0 to 8.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 3.0]
  Week 64: Radiologist: number analyzed (Participants) | 63 | 79 | 58
  Week 64: Radiologist | 1.0 [1.0 to 100.0] | 1.0 [1.0 to 30.0] | 1.0 [1.0 to 100.0]
  Week 64: Home Healthcare Services: number analyzed (Participants) | 5 | 9 | 6
  Week 64: Home Healthcare Services | 4.0 [1.0 to 9.0] | 4.0 [1.0 to 16.0] | 5.0 [2.0 to 90.0]
  Week 64: Other Practitioner: number analyzed (Participants) | 74 | 106 | 80
  Week 64: Other Practitioner | 1.0 [1.0 to 190.0] | 1.0 [1.0 to 190.0] | 1.0 [1.0 to 111.0]
  Week 80: Primary Care Physician: number analyzed (Participants) | 134 | 118 | 110
  Week 80: Primary Care Physician | 1.0 [1.0 to 102.0] | 1.0 [1.0 to 111.0] | 1.0 [1.0 to 101.0]
  Week 80: Neurologist: number analyzed (Participants) | 7 | 6 | 3
  Week 80: Neurologist | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 2.0]
  Week 80: Rheumatologist: number analyzed (Participants) | 16 | 33 | 15
  Week 80: Rheumatologist | 1.0 [1.0 to 100.0] | 1.0 [1.0 to 111.0] | 1.0 [1.0 to 101.0]
  Week 80: Physician Assistant or Nurse Practitioner: number analyzed (Participants) | 25 | 10 | 9
  Week 80: Physician Assistant or Nurse Practitioner | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 4.0] | 1.0 [1.0 to 90.0]
  Week 80: Pain Specialist: number analyzed (Participants) | 16 | 19 | 15
  Week 80: Pain Specialist | 1.5 [1.0 to 4.0] | 2.0 [1.0 to 111.0] | 1.0 [1.0 to 190.0]
  Week 80: Orthopedist: number analyzed (Participants) | 86 | 79 | 44
  Week 80: Orthopedist | 1.5 [1.0 to 101.0] | 1.0 [1.0 to 101.0] | 1.0 [1.0 to 100.0]
  Week 80: Physical Therapist: number analyzed (Participants) | 28 | 32 | 19
  Week 80: Physical Therapist | 8.0 [1.0 to 30.0] | 5.5 [1.0 to 21.0] | 3.0 [1.0 to 21.0]
  Week 80: Chiropractor: number analyzed (Participants) | 20 | 18 | 11
  Week 80: Chiropractor | 3.0 [1.0 to 111.0] | 4.5 [1.0 to 61.0] | 3.0 [1.0 to 120.0]
  Week 80: Alternative Medicine or Therapy: number analyzed (Participants) | 12 | 15 | 18
  Week 80: Alternative Medicine or Therapy | 3.5 [1.0 to 90.0] | 1.0 [1.0 to 90.0] | 2.0 [1.0 to 90.0]
  Week 80: Podiatrist: number analyzed (Participants) | 12 | 6 | 5
  Week 80: Podiatrist | 1.0 [1.0 to 90.0] | 1.0 [1.0 to 111.0] | 3.0 [1.0 to 101.0]
  Week 80: Nutritionist/Dietitian: number analyzed (Participants) | 5 | 2 | 4
  Week 80: Nutritionist/Dietitian | 1.0 [1.0 to 100.0] | 1.5 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Week 80: Radiologist: number analyzed (Participants) | 39 | 36 | 36
  Week 80: Radiologist | 1.0 [1.0 to 100.0] | 1.0 [1.0 to 4.0] | 1.0 [1.0 to 101.0]
  Week 80: Home Healthcare Services: number analyzed (Participants) | 4 | 3 | 2
  Week 80: Home Healthcare Services | 2.5 [1.0 to 140.0] | 4.0 [1.0 to 18.0] | 1.0 [1.0 to 1.0]
  Week 80: Other Practitioner: number analyzed (Participants) | 40 | 36 | 24
  Week 80: Other Practitioner | 1.0 [1.0 to 190.0] | 1.0 [1.0 to 100.0] | 1.0 [1.0 to 100.0]

58. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Participants Who Visited the Emergency Room Due to Osteoarthritis
Description: OA HCRU assessed healthcare usage during the last 3 months (for Baseline and Week 80) and past 8 weeks (for Week 64). Domain evaluated was number of participants who visited the emergency room due to OA.
Time Frame: Baseline, Weeks 64 and 80
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
Participants
  Baseline: number analyzed (Participants) | 1001 | 997 | 995
  Baseline | 15 | 23 | 11
  Week 64: number analyzed (Participants) | 773 | 782 | 799
  Week 64 | 10 | 15 | 5
  Week 80: number analyzed (Participants) | 432 | 396 | 424
  Week 80 | 4 | 5 | 2

59. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Visits to the Emergency Room Due to Osteoarthritis
Description: Osteoarthritis HCRU assessed healthcare usage during the last 3 months (for Baseline and Week 80) and past 8 weeks (for Week 64). Domain evaluated was number of visits to the emergency room due to OA.
Time Frame: Baseline, Weeks 64 and 80
Population: as for outcome 46
Measure: Median (Full Range); unit: visits
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 15 | 23 | 11
visits
  Baseline | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 222.0] | 1.0 [1.0 to 6.0]
  Week 64: number analyzed (Participants) | 10 | 15 | 5
  Week 64 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0]
  Week 80: number analyzed (Participants) | 4 | 5 | 2
  Week 80 | 1.0 [1.0 to 2.0] | 3.0 [1.0 to 11.0] | 1.0 [1.0 to 1.0]

60. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Participants Hospitalized Due to Osteoarthritis
Description: OA HCRU assessed healthcare usage during the last 3 months (for Baseline and Week 80) and past 8 weeks (for Week 64). Domain evaluated was number of participants who were hospitalized due to OA.
Time Frame: Baseline, Weeks 64 and 80
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
Participants
  Baseline: number analyzed (Participants) | 1001 | 997 | 995
  Baseline | 11 | 6 | 1
  Week 64: number analyzed (Participants) | 773 | 782 | 799
  Week 64 | 5 | 11 | 6
  Week 80: number analyzed (Participants) | 432 | 396 | 424
  Week 80 | 8 | 12 | 0

61. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Nights Stayed in the Hospital Due to Osteoarthritis
Description: OA HCRU assessed healthcare usage during the last 3 months (for Baseline and Week 80) and past 8 weeks (for Week 64). Domain evaluated was number of nights stayed in the hospital due to OA.
Time Frame: Baseline, Weeks 64 and 80
Population: as for outcome 46
Measure: Median (Full Range); unit: nights
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 11 | 12 | 6
nights
  Baseline: number analyzed (Participants) | 11 | 6 | 1
  Baseline | 12.0 [1.0 to 15.0] | 9.0 [1.0 to 14.0] | 11.0 [11.0 to 11.0]
  Week 64: number analyzed (Participants) | 5 | 11 | 6
  Week 64 | 2.0 [1.0 to 20.0] | 2.0 [1.0 to 40.0] | 2.0 [1.0 to 4.0]
  Week 80: number analyzed (Participants) | 8 | 12 | 0
  Week 80 | 2.0 [1.0 to 26.0] | 2.0 [1.0 to 21.0] |

62. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Participants Who Used Any Aids/Devices for Doing Things Due to Osteoarthritis
Description: OA HCRU assessed healthcare usage during the last 3 months (for Baseline and Week 80) and past 8 weeks (for Week 64). Domain evaluated was number of participants who used any aids/devices for doing things. Aids such as walking aid, wheelchair, device or utensil for dress/bathe/eat and any other aids/devices.
Time Frame: Baseline, Weeks 64 and 80
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
Participants
  Baseline: Walking Aid Use: number analyzed (Participants) | 1001 | 997 | 995
  Baseline: Walking Aid Use: Never | 852 | 838 | 851
  Baseline: Walking Aid Use: Rarely | 27 | 18 | 24
  Baseline: Walking Aid Use: Sometimes | 71 | 69 | 75
  Baseline: Walking Aid Use: Often | 32 | 43 | 26
  Baseline: Walking Aid Use: Always | 19 | 29 | 19
  Baseline: Wheelchair Use: number analyzed (Participants) | 1001 | 997 | 995
  Baseline: Wheelchair Use: Never | 992 | 989 | 988
  Baseline: Wheelchair Use: Rarely | 2 | 2 | 1
  Baseline: Wheelchair Use: Sometimes | 4 | 6 | 5
  Baseline: Wheelchair Use: Often | 3 | 0 | 1
  Baseline: Wheelchair Use: Always | 0 | 0 | 0
  Baseline: Device/Utensil to Dress Bathe Eat: number analyzed (Participants) | 1001 | 997 | 995
  Baseline: Device/Utensil to Dress Bathe Eat: Never | 970 | 976 | 977
  Baseline: Device/Utensil to Dress Bathe Eat: Rarely | 2 | 1 | 0
  Baseline: Device/Utensil to Dress Bathe Eat: Sometimes | 7 | 6 | 6
  Baseline: Device/Utensil to Dress Bathe Eat: Often | 16 | 9 | 7
  Baseline: Device/Utensil to Dress Bathe Eat: Always | 6 | 5 | 5
  Baseline: Other Aids Or Devices: number analyzed (Participants) | 1001 | 997 | 995
  Baseline: Other Aids Or Devices: Never | 932 | 935 | 921
  Baseline: Other Aids Or Devices: Rarely | 8 | 7 | 9
  Baseline: Other Aids Or Devices: Sometimes | 27 | 22 | 41
  Baseline: Other Aids Or Devices: Often | 27 | 22 | 14
  Baseline: Other Aids Or Devices: Always | 7 | 11 | 10
  Week 64: Walking Aid Use: number analyzed (Participants) | 773 | 782 | 799
  Week 64: Walking Aid Use: Never | 662 | 662 | 714
  Week 64: Walking Aid Use: Rarely | 21 | 9 | 12
  Week 64: Walking Aid Use: Sometimes | 48 | 47 | 37
  Week 64: Walking Aid Use: Often | 20 | 30 | 17
  Week 64: Walking Aid Use: Always | 22 | 34 | 19
  Week 64: Wheelchair Use: number analyzed (Participants) | 773 | 782 | 799
  Week 64: Wheelchair Use: Never | 765 | 776 | 794
  Week 64: Wheelchair Use: Rarely | 2 | 1 | 2
  Week 64: Wheelchair Use: Sometimes | 4 | 2 | 3
  Week 64: Wheelchair Use: Often | 2 | 1 | 0
  Week 64: Wheelchair Use: Always | 0 | 2 | 0
  Week 64: Device/Utensil to Dress Bathe Eat: number analyzed (Participants) | 773 | 782 | 799
  Week 64: Device/Utensil to Dress Bathe Eat: Never | 760 | 768 | 792
  Week 64: Device/Utensil to Dress Bathe Eat: Rarely | 2 | 1 | 1
  Week 64: Device/Utensil to Dress Bathe Eat: Sometimes | 7 | 7 | 2
  Week 64: Device/Utensil to Dress Bathe Eat: Often | 3 | 5 | 2
  Week 64: Device/Utensil to Dress Bathe Eat: Always | 1 | 1 | 2
  Week 64: Other Aids Or Devices: number analyzed (Participants) | 773 | 782 | 799
  Week 64: Other Aids Or Devices: Never | 733 | 720 | 771
  Week 64: Other Aids Or Devices: Rarely | 6 | 9 | 11
  Week 64: Other Aids Or Devices: Sometimes | 19 | 26 | 8
  Week 64: Other Aids Or Devices: Often | 12 | 20 | 6
  Week 64: Other Aids Or Devices: Always | 3 | 7 | 3
  Week 80: Walking Aid Use: number analyzed (Participants) | 432 | 396 | 424
  Week 80: Walking Aid Use: Never | 373 | 322 | 386
  Week 80: Walking Aid Use: Rarely | 12 | 10 | 6
  Week 80: Walking Aid Use: Sometimes | 25 | 25 | 17
  Week 80: Walking Aid Use: Often | 14 | 17 | 7
  Week 80: Walking Aid Use: Always | 8 | 22 | 8
  Week 80: Wheelchair Use: number analyzed (Participants) | 432 | 396 | 424
  Week 80: Wheelchair Use: Never | 430 | 389 | 421
  Week 80: Wheelchair Use: Rarely | 0 | 2 | 2
  Week 80: Wheelchair Use: Sometimes | 1 | 4 | 1
  Week 80: Wheelchair Use: Often | 0 | 0 | 0
  Week 80: Wheelchair Use: Always | 1 | 1 | 0
  Week 80: Device/Utensil to Dress Bathe Eat: number analyzed (Participants) | 432 | 396 | 424
  Week 80: Device/Utensil to Dress Bathe Eat: Never | 425 | 383 | 422
  Week 80: Device/Utensil to Dress Bathe Eat: Rarely | 0 | 0 | 1
  Week 80: Device/Utensil to Dress Bathe Eat: Sometimes | 2 | 6 | 1
  Week 80: Device/Utensil to Dress Bathe Eat: Often | 3 | 5 | 0
  Week 80: Device/Utensil to Dress Bathe Eat: Always | 2 | 2 | 0
  Week 80: Other Aids Or Devices: number analyzed (Participants) | 432 | 396 | 424
  Week 80: Other Aids Or Devices: Never | 416 | 375 | 410
  Week 80: Other Aids Or Devices: Rarely | 4 | 3 | 4
  Week 80: Other Aids Or Devices: Sometimes | 5 | 11 | 4
  Week 80: Other Aids Or Devices: Often | 5 | 4 | 2
  Week 80: Other Aids Or Devices: Always | 2 | 3 | 4

63. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Participants Who Quit Job Due to Osteoarthritis
Description: OA HCRU assessed healthcare usage during the last 3 months (for Baseline and Week 80) and past 8 weeks (for Week 64). Domain evaluated was number of participants who quit job due to OA.
Time Frame: Baseline, Weeks 64 and 80
Population: as for outcome 46
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 995
Participants
  Baseline: number analyzed (Participants) | 1001 | 997 | 995
  Baseline | 47 | 55 | 65
  Week 64: number analyzed (Participants) | 773 | 782 | 799
  Week 64 | 28 | 35 | 26
  Week 80: number analyzed (Participants) | 432 | 396 | 424
  Week 80 | 12 | 18 | 6

64. Secondary Outcome: Health Care Resource Utilization (HCRU): Duration Since Quitting Job Due to Osteoarthritis
Description: OA HCRU assessed healthcare usage during the last 3 months (for Baseline and Week 80) and past 8 weeks (for Week 64). Domain evaluated was duration since quitting job due to OA.
Time Frame: Baseline, Weeks 64 and 80
Population: ITT population was analyzed. One additional participant apart from the ones who had responded for quitting job responded to duration since quitting job. Here 'Overall number of participants analyzed'=participants evaluable for this outcome measure. Here, "Number analyzed" =participants evaluable at specified time point for each arm, respectively.
Measure: Median (Full Range); unit: years
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 47 | 55 | 66
years
  Baseline | 2.0 [0.1 to 15.4] | 1.8 [0.3 to 20.0] | 2.4 [0.1 to 80.0]
  Week 64: number analyzed (Participants) | 33 | 38 | 32
  Week 64 | 2.4 [0.2 to 18.6] | 1.8 [0.1 to 31.0] | 4.0 [0.1 to 90.0]
  Week 80: number analyzed (Participants) | 12 | 18 | 6
  Week 80 | 2.0 [0.3 to 30.4] | 2.0 [0.1 to 50.0] | 1.8 [0.2 to 20.4]

65. Secondary Outcome: Number of Participants With Categorical Change From Baseline in Lower Extremity Activity Scale (LEAS) at Weeks 4, 8, 16, 24, 56 and 80
Description: The LEAS is a self-administered scale to assess activity level in participants having total knee arthroplasty. The LEAS scale reflected four levels of lower-extremity activity (1)housebound(unable to walk or a minimal ability to walk) (2)more ordinary walking about the house (3)walking about the community (4)walking about the community as well as substantial work or exercise. It consisted of 12 questions resulting in 18-level scale that allowed participants to select a single description that most represented his or her self-perceived activity level. The final score was simply the number of the descriptor selected by the participant as being most representative of his or her activity level. The minimum possible score was 1(entirely bedbound) and the maximum possible score was 18(currently competitive athlete). Higher score indicated increased activity. Categorical changes from baseline were reported in terms of improvement (Change >0), No change and worsening (Change less than [<] 0).
Time Frame: Baseline, Weeks 4, 8, 16, 24, 56 and 80
Population: as for outcome 46
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1000 | 995 | 994
Participants
  Change at Week 4: Improvement | 423 | 421 | 411
  Change at Week 4: No Change | 370 | 394 | 369
  Change at Week 4: Worsening | 207 | 180 | 214
  Change at Week 8: Improvement | 454 | 443 | 445
  Change at Week 8: No Change | 325 | 362 | 348
  Change at Week 8: Worsening | 221 | 190 | 201
  Change at Week 16: Improvement | 488 | 470 | 477
  Change at Week 16: No Change | 288 | 312 | 312
  Change at Week 16: Worsening | 224 | 213 | 205
  Change at Week 24: Improvement | 478 | 458 | 467
  Change at Week 24: No Change | 277 | 302 | 291
  Change at Week 24: Worsening | 245 | 235 | 236
  Change at Week 56: Improvement | 486 | 429 | 461
  Change at Week 56: No Change | 270 | 314 | 300
  Change at Week 56: Worsening | 244 | 252 | 233
  Change at Week 80: number analyzed (Participants) | 438 | 408 | 432
  Change at Week 80: Improvement | 220 | 196 | 227
  Change at Week 80: No Change | 105 | 97 | 125
  Change at Week 80: Worsening | 113 | 115 | 80
Statistical Analysis 1: Comparison: Tanezumab 2.5 mg vs NSAID; Week 4: Cochran-Mantel-Haenszel test for row mean scores differ, stratified by the combinations of the three stratification factors (index joint, highest Kellgren-Lawrence grade and NSAID); Test type: Superiority; p = 0.6037, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 65, analysis 1]; Test type: Superiority; p = 0.1928, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Tanezumab 2.5 mg vs NSAID; Week 8: Cochran-Mantel-Haenszel test for row mean scores differ, stratified by the combinations of the three stratification factors (index joint, highest Kellgren-Lawrence grade and NSAID); Test type: Superiority; p = 0.7204, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 65, analysis 3]; Test type: Superiority; p = 0.7969, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Tanezumab 2.5 mg vs NSAID; [analysis description as in outcome 48, analysis 1]; Test type: Superiority; p = 0.7857, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 48, analysis 1]; Test type: Superiority; p = 0.6627, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Tanezumab 2.5 mg vs NSAID; Week 24: Cochran-Mantel-Haenszel test for row mean scores differ, stratified by the combinations of the three stratification factors (index joint, highest Kellgren-Lawrence grade and NSAID); Test type: Superiority; p = 0.9867, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 65, analysis 7]; Test type: Superiority; p = 0.8190, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: Tanezumab 2.5 mg vs NSAID; [analysis description as in outcome 48, analysis 3]; Test type: Superiority; p = 0.7284, Cochran-Mantel-Haenszel
Statistical Analysis 10: Comparison: Tanezumab 5 mg vs NSAID; [analysis description as in outcome 48, analysis 3]; Test type: Superiority; p = 0.1545, Cochran-Mantel-Haenszel

66. Secondary Outcome: Change From Baseline in Average Daily Minutes of Physical Activity at Weeks 16 and 56
Description: Participant activity level was assessed using actigraphy. Participants continuously wore the accelerometer (apart for water activities) in the morning until going to bed at night for 7 or 14 consecutive days while going about their usual daily activities. Participants maintained a log (electronic or written) to record when the accelerometer was put on in the morning and removed at night (or if removed for any other purpose).
Time Frame: Baseline, Weeks 16 and 56
Population: Accelerometry analysis set = All participants treated with tanezumab or matching placebo SC who had any baseline or post-baseline accelerometry data. 'Overall number of participants analyzed'=participants evaluable for this outcome measure. Here, "Number analyzed" =participants who were evaluable at specified time point for each arm, respectively.
Measure: Median (Full Range); unit: minutes
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 36 | 46 | 44
minutes
  Baseline | 97.0 [22.6 to 164.9] | 107.1 [50.5 to 195.5] | 99.2 [13.9 to 176.9]
  Change at Week 16: number analyzed (Participants) | 20 | 29 | 24
  Change at Week 16 | 3.9 [-39.5 to 60.1] | 2.9 [-49.4 to 45.1] | -4.2 [-45.5 to 67.8]
  Change at Week 56: number analyzed (Participants) | 7 | 8 | 10
  Change at Week 56 | -8.9 [-63.5 to 16.9] | -10.1 [-25.4 to 30.2] | 3.9 [-17.7 to 15.3]

67. Secondary Outcome: Change From Baseline in Average Daily Physical Activity Counts at Weeks 16 and 56
Description: An average daily physical activity count was measured using actigraphy. Participants continuously wore the accelerometer (apart for water activities) in the morning until going to bed at night for 7 or 14 consecutive days while going about their usual daily activities. Participants maintained a log (electronic or written) to record when the accelerometer was put on in the morning and removed at night (or if removed for any other purpose).
Time Frame: Baseline, Weeks 16 and 56
Population: as for outcome 66
Measure: Median (Full Range); unit: physical activity counts
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 36 | 46 | 44
physical activity counts
  Baseline | 75244 [12385 to 129724] | 95911 [25816 to 428586] | 74414 [8136.6 to 253672]
  Change at Week 16: number analyzed (Participants) | 20 | 29 | 24
  Change at Week 16 | -470.0 [-32693 to 225384] | -2261 [-114000 to 125895] | 1202.9 [-70004 to 300461]
  Change at Week 56: number analyzed (Participants) | 7 | 8 | 10
  Change at Week 56 | -14552 [-42956 to 24607] | -8313 [-60556 to 53888] | 4414.3 [-15896 to 56451]

68. Secondary Outcome: Change From Baseline in Average Daily Minutes of Moderate to Vigorous Physical Activity at Weeks 16 and 56
Description: An average daily physical activity count was measured using actigraphy which was then sorted into three intensity thresholds: light (100 - less than {<1500} counts moderate (1,500 - <6500 counts), and vigorous (>=6500 counts). Participants continuously wore the accelerometer (apart for water activities) in the morning until going to bed at night for 7 or 14 consecutive days while going about their usual daily activities. Participants maintained a log (electronic or written) to record when the accelerometer was put on in the morning and removed at night (or if removed for any other purpose).
Time Frame: Baseline, Weeks 16 and 56
Population: as for outcome 66
Measure: Median (Full Range); unit: minutes
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 36 | 46 | 44
minutes
  Baseline | 41.2 [2.2 to 80.4] | 53.1 [7.3 to 156.0] | 41.9 [0.7 to 117.0]
  Change at Week 16: number analyzed (Participants) | 20 | 29 | 24
  Change at Week 16 | 0.7 [-25.3 to 62.7] | -1.6 [-72.2 to 78.8] | -0.1 [-39.2 to 68.7]
  Change at Week 56: number analyzed (Participants) | 7 | 8 | 10
  Change at Week 56 | -3.8 [-27.5 to 23.5] | 2.7 [-27.5 to 38.5] | 7.4 [-13.4 to 40.7]

69. Secondary Outcome: Change From Baseline in Average Daily Minutes of Bouted (Sustained) Moderate to Vigorous Physical Activity at Weeks 16 and 56
Description: An average daily physical activity count was measured using actigraphy which was then sorted into three intensity thresholds: light (100 - <1,500 counts) moderate (1,500 - <6,500 counts), and vigorous (>=6,500 counts). Participants continuously wore the accelerometer (apart for water activities) in the morning until going to bed at night for 7 or 14 consecutive days while going about their usual daily activities. Participants maintained a log (electronic or written) to record when the accelerometer was put on in the morning and removed at night (or if removed for any other purpose).A "bout" of moderate to vigorous activity was defined as 10 or more consecutive minutes above the moderate physical activity level threshold, with allowance for interruptions of 1 or 2 minutes below the threshold.
Time Frame: Baseline, Weeks 16 and 56
Population: as for outcome 66
Measure: Median (Full Range); unit: minutes
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 36 | 46 | 44
minutes
  Baseline | 0.0 [0.0 to 16.5] | 0.0 [0.0 to 111.5] | 0.0 [0.0 to 42.4]
  Change at Week 16: number analyzed (Participants) | 20 | 29 | 24
  Change at Week 16 | 0.0 [-13.1 to 25.9] | 0.0 [-73.3 to 13.0] | 0.0 [-12.6 to 64.8]
  Change at Week 56: number analyzed (Participants) | 7 | 8 | 10
  Change at Week 56 | 0.0 [-5.8 to 0.0] | -1.4 [-11.5 to 8.2] | 0.0 [-2.0 to 6.5]

70. Secondary Outcome: Change From Baseline in Average Daily Step Count at Weeks 16 and 56
Description: Average daily step count was measured using actigraphy. Participants continuously wore the accelerometer (apart for water activities) in the morning until going to bed at night for 7 or 14 consecutive days while going about their usual daily activities. Participants maintained a log (electronic or written) to record when the accelerometer was put on in the morning and removed at night (or if removed for any other purpose).
Time Frame: Baseline, Weeks 16 and 56
Population: as for outcome 66
Measure: Median (Full Range); unit: step count
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 36 | 46 | 44
step count
  Baseline | 4851.0 [827.6 to 9206.5] | 5834.8 [2041.0 to 17895] | 4779.0 [1015.6 to 11759]
  Change at Week 16: number analyzed (Participants) | 20 | 29 | 24
  Change at Week 16 | 350.9 [-4970 to 5017.9] | 87.8 [-9415 to 5849.9] | -705.7 [-3286 to 6270.4]
  Change at Week 56: number analyzed (Participants) | 7 | 8 | 10
  Change at Week 56 | -1938 [-4055 to 138.3] | -543.2 [-1856 to 3609.9] | 242.6 [-4411 to 3312.2]

71. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to Week 80 that were absent before treatment or that worsened relative to pre-treatment state. AEs included both serious and non-serious AEs. Clinically significant physical examination abnormalities were reported as AEs.
Time Frame: Baseline up to Week 80
Population: Safety population included all participants treated with tanezumab or placebo SC.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
Participants
  AEs | 681 | 744 | 666
  SAEs | 78 | 110 | 66

72. Secondary Outcome: Number of Participants With Treatment-Related Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to Week 80 that were absent before treatment or that worsened relative to pre-treatment state. Relatedness to study drug was assessed by the investigator.
Time Frame: Baseline up to Week 80
Population: Safety population included all participants treated with tanezumab or placebo SC.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
Participants
  Treatment Related AEs | 190 | 250 | 179
  Treatment Related SAEs | 7 | 20 | 7

73. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities With Regard to Normal Baseline
Description: Primary Abnormality criteria: HGB, hematocrit, RBC count <0.8* lower limit of normal(LLN); Ery. mean corpuscular volume/hemoglobin/ HGB concentration, RBCs distribution width <0.9*LLN, >1.1*upper limit of normal(ULN); platelets <0.5*LLN,>1.75*ULN; Leukocytes <0.6*LLN, >1.5*ULN; Lymphocytes, Neutrophils <0.8*LLN, >1.2*ULN; Basophils,Eosinophils,Monocytes>1.2*ULN; Prothrombin time/Intl. normalized ratio>1.1*ULN; total bilirubin>1.5*ULN; aspartate aminotransferase,alanine aminotransferase,gamma GT,LDH,alkaline phosphatase >3.0*ULN; total protein; albumin<0.8*LLN, >1.2*ULN; blood urea nitrogen,creatinine,Cholesterol,triglycerides >1.3*ULN; Urate>1.2*ULN; sodium<0.95*LLN,>1.05*ULN; potassium,chloride,calcium,magnesium,bicarbonate <0.9*LLN, >1.1*ULN; phosphate<0.8*LLN, >1.2*ULN; glucose<0.6*LLN, >1.5*ULN; HGB A1C >1.3*ULN; creatine kinase>2.0*ULN, specific gravity<1.003, >1.030; pH<4.5, >8;Urine erythrocytes,Leukocytes>=20.
Time Frame: Baseline up to Week 80
Population: Safety population included all participants treated with tanezumab or placebo SC. Here 'Overall number of participants analyzed' = participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 877 | 897 | 884
Participants | 109 | 102 | 121

74. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities With Regard to Abnormal Baseline
Description: Primary Abnormality criteria: hemoglobin; hematocrit; RBC count < 0.8*LLN; Ery. mean corpuscular volume/ hemoglobin/ HGB concentration, erythrocytes distribution width <0.9*LLN, >1.1*ULN; platelets <0.5*LLN,>1.75*upper limit of normal (ULN); white blood cell count<0.6*LLN, >1.5*ULN; Lymphocytes, Lymphocytes/Leukocytes, Neutrophils, Neutrophils/Leukocytes <0.8*LLN, >1.2*ULN; Basophils, Eosinophils, Monocytes >1.2*ULN; total bilirubin>1.5*ULN; aspartate aminotransferase, alanine aminotransferase, gamma GT,LDH, alkaline phosphatase >3.0*ULN; total protein; albumin<0.8*LLN, >1.2*ULN; blood urea nitrogen, creatinine, Cholesterol, triglycerides >1.3*ULN; Urate >1.2*ULN; sodium <0.95*LLN,>1.05*ULN; potassium, chloride, calcium, magnesium, bicarbonate <0.9*LLN, >1.1*ULN; phosphate <0.8*LLN, >1.2*ULN; glucose <0.6*LLN, >1.5*ULN; Hemoglobin A1C >1.3*ULN; creatine kinase >2.0*ULN; specific gravity<1.003, >1.030; Urine erythrocytes,Leukocytes>=20; Hyaline Casts>=1.
Time Frame: Baseline up to Week 80
Population: as for outcome 73
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 706 | 731 | 691
Participants | 78 | 61 | 84

75. Secondary Outcome: Change From Baseline in Blood Pressure (BP) at Weeks 2, 4, 8, 16, 24, 32, 40, 48, 56, 64 and 80
Description: Measurement of BP included sitting systolic blood pressure (SBP) and diastolic blood pressure (DBP).
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 32, 40, 48, 56, 64 and 80
Population: Safety population included all participants treated with tanezumab or placebo SC. Here, "Number analyzed" signifies those participants who were evaluable for this outcome measure for specified categories.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
millimeters of mercury (mmHg)
  SBP: Baseline | 128.9 (12.91) | 129.3 (13.43) | 128.8 (13.26)
  SBP: Change at Week 2: number analyzed (Participants) | 973 | 971 | 966
  SBP: Change at Week 2 | -2.7 (11.69) | -4.2 (11.92) | -1.2 (11.24)
  SBP: Change at Week 4: number analyzed (Participants) | 967 | 955 | 949
  SBP: Change at Week 4 | -4.0 (11.44) | -4.9 (12.68) | -1.8 (11.29)
  SBP: Change at Week 8: number analyzed (Participants) | 930 | 926 | 918
  SBP: Change at Week 8 | -2.9 (12.16) | -3.8 (12.60) | -1.8 (11.68)
  SBP: Change at Week 16: number analyzed (Participants) | 635 | 637 | 601
  SBP: Change at Week 16 | -3.0 (11.66) | -3.7 (12.95) | -1.3 (12.37)
  SBP: Change at Week 24: number analyzed (Participants) | 545 | 542 | 528
  SBP: Change at Week 24 | -3.0 (12.35) | -3.1 (13.49) | -1.7 (11.83)
  SBP: Change at Week 32: number analyzed (Participants) | 518 | 512 | 505
  SBP: Change at Week 32 | -2.8 (11.95) | -3.3 (13.70) | -1.7 (13.49)
  SBP: Change at Week 40: number analyzed (Participants) | 492 | 474 | 482
  SBP: Change at Week 40 | -2.5 (11.35) | -3.8 (14.41) | -2.3 (13.42)
  SBP: Change at Week 48: number analyzed (Participants) | 471 | 449 | 459
  SBP: Change at Week 48 | -2.7 (12.21) | -3.0 (13.29) | -2.2 (12.97)
  SBP: Change at Week 56: number analyzed (Participants) | 446 | 421 | 445
  SBP: Change at Week 56 | -3.1 (11.76) | -3.4 (13.78) | -2.2 (12.64)
  SBP: Change at Week 64: number analyzed (Participants) | 430 | 407 | 435
  SBP: Change at Week 64 | -2.1 (13.40) | -2.1 (13.56) | -2.8 (13.33)
  SBP: Change at Week 80: number analyzed (Participants) | 423 | 390 | 415
  SBP: Change at Week 80 | -1.0 (13.24) | -1.3 (13.71) | -2.3 (13.31)
  DBP: Baseline | 79.3 (8.56) | 79.1 (8.68) | 79.3 (8.57)
  DBP: Change at Week 2: number analyzed (Participants) | 973 | 971 | 966
  DBP: Change at Week 2 | -1.3 (8.29) | -2.1 (7.96) | -1.1 (7.84)
  DBP: Change at Week 4: number analyzed (Participants) | 967 | 955 | 949
  DBP: Change at Week 4 | -2.2 (8.06) | -2.5 (8.10) | -1.4 (8.19)
  DBP: Change at Week 8: number analyzed (Participants) | 930 | 926 | 918
  DBP: Change at Week 8 | -1.1 (7.84) | -1.7 (8.24) | -1.1 (8.23)
  DBP: Change at Week 16: number analyzed (Participants) | 635 | 637 | 601
  DBP: Change at Week 16 | -1.3 (8.14) | -1.8 (8.53) | -1.1 (8.30)
  DBP: Change at Week 24: number analyzed (Participants) | 545 | 542 | 528
  DBP: Change at Week 24 | -1.3 (8.39) | -1.7 (8.91) | -1.4 (8.26)
  DBP: Change at Week 32: number analyzed (Participants) | 518 | 512 | 505
  DBP: Change at Week 32 | -1.3 (8.28) | -1.4 (9.14) | -1.2 (8.91)
  DBP: Change at Week 40: number analyzed (Participants) | 492 | 474 | 482
  DBP: Change at Week 40 | -1.2 (8.07) | -2.0 (8.90) | -1.1 (8.69)
  DBP: Change at Week 48: number analyzed (Participants) | 471 | 449 | 459
  DBP: Change at Week 48 | -0.9 (8.82) | -1.8 (8.89) | -1.5 (8.65)
  DBP: Change at Week 56: number analyzed (Participants) | 446 | 421 | 445
  DBP: Change at Week 56 | -1.8 (8.61) | -1.9 (9.11) | -1.2 (8.69)
  DBP: Change at Week 64: number analyzed (Participants) | 430 | 407 | 435
  DBP: Change at Week 64 | -0.8 (8.63) | -0.8 (9.23) | -1.7 (9.03)
  DBP: Change at Week 80: number analyzed (Participants) | 423 | 390 | 415
  DBP: Change at Week 80 | -0.6 (8.73) | -0.6 (9.66) | -1.2 (9.35)

76. Secondary Outcome: Change From Baseline in Heart Rate at Weeks 2, 4, 8, 16, 24, 32, 40, 48, 56, 64 and 80
Description: Heart rate (pulse rate) was measured at sitting position.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 32, 40, 48, 56, 64 and 80
Population: Safety population included all participants treated with tanezumab or placebo SC. Here, "Number analyzed" =participants who were evaluable at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 998 | 996
beats per minute
  Baseline | 70.8 (9.09) | 70.5 (9.66) | 70.6 (9.36)
  Change at Week 2: number analyzed (Participants) | 973 | 971 | 966
  Change at Week 2 | 1.8 (8.65) | 2.0 (8.50) | 1.1 (8.31)
  Change at Week 4: number analyzed (Participants) | 967 | 955 | 949
  Change at Week 4 | 1.6 (9.00) | 2.0 (9.03) | 1.2 (8.75)
  Change at Week 8: number analyzed (Participants) | 930 | 926 | 917
  Change at Week 8 | 0.7 (9.06) | 0.8 (8.54) | 0.1 (8.78)
  Change at Week 16: number analyzed (Participants) | 635 | 637 | 601
  Change at Week 16 | 0.5 (9.37) | 0.5 (9.14) | 0.8 (8.86)
  Change at Week 24: number analyzed (Participants) | 545 | 542 | 528
  Change at Week 24 | 0.4 (9.46) | 0.7 (9.36) | 0.8 (9.24)
  Change at Week 32: number analyzed (Participants) | 518 | 512 | 505
  Change at Week 32 | 1.2 (9.67) | 1.6 (9.34) | 1.7 (9.70)
  Change at Week 40: number analyzed (Participants) | 492 | 474 | 482
  Change at Week 40 | 1.2 (9.89) | 1.6 (9.40) | 1.4 (8.71)
  Change at Week 48: number analyzed (Participants) | 471 | 448 | 458
  Change at Week 48 | 0.6 (9.86) | 1.0 (9.34) | 1.3 (9.44)
  Change at Week 56: number analyzed (Participants) | 446 | 421 | 445
  Change at Week 56 | 0.2 (9.51) | 0.1 (10.15) | -0.0 (9.28)
  Change at Week 64: number analyzed (Participants) | 430 | 407 | 435
  Change at Week 64 | 1.5 (9.81) | 1.5 (9.55) | 0.5 (9.84)
  Change at Week 80: number analyzed (Participants) | 423 | 390 | 415
  Change at Week 80 | 0.9 (10.24) | 0.6 (9.97) | 0.9 (9.61)

77. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters at Weeks 56 and 80
Description: A 12-lead ECG was recorded after participants had rested for at least 5 minutes in the supine position in a quiet environment. All standard intervals (PR, QRS, QT, QTcF, QTcB, RR intervals) were collected. ECG abnormalities included: 1) QT interval, QT interval corrected using Bazett's formula (QTcB) and QT interval corrected using Fridericia's formula (QTcF): increase from baseline greater than (>) 30 millisecond (ms) or 60 ms; absolute value > 450 ms, >480 ms and > 500 ms; 2) heart rate (HR) : absolute value <=50 bpm and decrease from baseline >=20 bpm; absolute value >=120 beats per minute (bpm) and increase from baseline >=20 bpm; 3) PR interval: absolute value >=220 ms and increase from baseline >=20 ms; 4) QRS interval: absolute value >= 120 ms.
Time Frame: Baseline, Weeks 56 and 80
Population: Safety population included all participants treated with tanezumab or placebo SC. 'Overall number of participants analyzed'=participants evaluable for this outcome measure. Here, "Number analyzed" =participants who were evaluable at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 995 | 995
milliseconds
  RR Interval: Baseline | 940.5 (136.21) | 940.1 (144.48) | 936.1 (142.31)
  RR Interval:Change at Week 56: number analyzed (Participants) | 440 | 413 | 441
  RR Interval:Change at Week 56 | -26.3 (123.23) | -22.6 (128.58) | -14.9 (128.73)
  RR Interval:Change at Week 80: number analyzed (Participants) | 419 | 381 | 410
  RR Interval:Change at Week 80 | -33.6 (119.23) | -32.4 (126.08) | -34.3 (133.83)
  PR Interval: Baseline: number analyzed (Participants) | 996 | 990 | 991
  PR Interval: Baseline | 165.0 (27.43) | 165.9 (25.45) | 163.9 (23.98)
  PR Interval:Change at Week 56: number analyzed (Participants) | 435 | 410 | 434
  PR Interval:Change at Week 56 | 1.7 (12.98) | 0.6 (13.33) | 1.7 (14.40)
  PR Interval:Change at Week 80: number analyzed (Participants) | 412 | 378 | 401
  PR Interval:Change at Week 80 | 0.3 (13.39) | -0.8 (14.70) | 0.6 (13.80)
  QRS Interval: Baseline | 94.9 (13.12) | 94.6 (13.65) | 94.3 (13.16)
  QRS Interval:Change at Week 56: number analyzed (Participants) | 440 | 413 | 441
  QRS Interval:Change at Week 56 | 0.2 (8.22) | 0.4 (8.30) | -0.4 (7.39)
  QRS Interval:Change at Week 80: number analyzed (Participants) | 419 | 381 | 410
  QRS Interval:Change at Week 80 | -0.2 (8.12) | 1.0 (8.64) | -0.1 (7.81)
  QT Interval: Baseline: number analyzed (Participants) | 999 | 994 | 994
  QT Interval: Baseline | 405.0 (28.86) | 403.8 (30.08) | 404.3 (29.33)
  QT Interval:Change at Week 56: number analyzed (Participants) | 437 | 413 | 440
  QT Interval:Change at Week 56 | -3.5 (24.07) | -4.5 (25.06) | -2.9 (26.58)
  QT Interval:Change at Week 80: number analyzed (Participants) | 417 | 381 | 408
  QT Interval:Change at Week 80 | -6.2 (22.56) | -6.8 (24.46) | -6.0 (25.34)
  QTCB Interval: Baseline: number analyzed (Participants) | 999 | 994 | 994
  QTCB Interval: Baseline | 419.3 (21.85) | 418.5 (21.96) | 419.7 (21.60)
  QTCB Interval:Change at Week 56: number analyzed (Participants) | 437 | 413 | 440
  QTCB Interval:Change at Week 56 | 2.3 (18.82) | 0.5 (17.83) | 0.2 (19.66)
  QTCB Interval:Change at Week 80: number analyzed (Participants) | 417 | 381 | 408
  QTCB Interval:Change at Week 80 | 1.5 (19.37) | 0.2 (17.98) | 1.7 (19.06)
  QTCF Interval: Baseline: number analyzed (Participants) | 999 | 994 | 994
  QTCF Interval: Baseline | 414.2 (19.96) | 413.3 (20.09) | 414.3 (19.49)
  QTCF Interval:Change at Week 56: number analyzed (Participants) | 437 | 413 | 440
  QTCF Interval:Change at Week 56 | 0.3 (16.24) | -1.2 (15.55) | -0.8 (17.50)
  QTCF Interval:Change at Week 80: number analyzed (Participants) | 417 | 381 | 408
  QTCF Interval:Change at Week 80 | -1.2 (16.16) | -2.1 (15.55) | -1.0 (16.21)

78. Secondary Outcome: Change From Baseline in Heart Rate (as Assessed by ECG) at Weeks 56 and 80
Description: Heart rate was measured at sitting position.
Time Frame: Baseline, Weeks 56 and 80
Population: as for outcome 77
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1002 | 995 | 995
beats per minute
  Baseline | 65.2 (9.70) | 65.4 (10.30) | 65.6 (10.36)
  Change at Week 56: number analyzed (Participants) | 440 | 413 | 441
  Change at Week 56 | 2.0 (9.10) | 1.7 (9.72) | 1.0 (9.95)
  Change at Week 80: number analyzed (Participants) | 419 | 381 | 410
  Change at Week 80 | 2.7 (9.00) | 2.3 (9.34) | 2.5 (10.02)

79. Secondary Outcome: Number of Participants With Confirmed Orthostatic Hypotension
Description: Orthostatic hypotension was defined as postural change (supine to standing) that met the following criteria: For systolic BP <=150 mmHg (mean supine): Reduction in systolic BP>=20 mmHg or reduction in diastolic BP>=10 mmHg at the 1 and/or 3 minute standing BP measurements. For systolic BP >150 mmHg (mean supine): Reduction in systolic BP>=30 mmHg or reduction in diastolic BP>=15 mmHg at the 1 and/or 3 minute standing BP measurements. If the 1 minute or 3 minute standing BP in a sequence met the orthostatic hypotension criteria, then that sequence was considered positive. If 2 of 2 or 2 of 3 sequences were positive, then orthostatic hypotension was considered confirmed.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 32, 40, 48, 56, 64 and 80
Population: as for outcome 77
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1001 | 996 | 996
Participants
  Baseline | 0 | 3 | 1
  Week 2: number analyzed (Participants) | 956 | 957 | 954
  Week 2 | 2 | 4 | 2
  Week 4: number analyzed (Participants) | 949 | 938 | 937
  Week 4 | 1 | 1 | 2
  Week 8: number analyzed (Participants) | 917 | 918 | 914
  Week 8 | 0 | 2 | 1
  Week 16: number analyzed (Participants) | 677 | 697 | 654
  Week 16 | 1 | 1 | 0
  Week 24: number analyzed (Participants) | 544 | 538 | 525
  Week 24 | 0 | 1 | 1
  Week 32: number analyzed (Participants) | 511 | 503 | 497
  Week 32 | 2 | 2 | 0
  Week 40: number analyzed (Participants) | 488 | 472 | 480
  Week 40 | 1 | 1 | 1
  Week 48: number analyzed (Participants) | 467 | 447 | 459
  Week 48 | 2 | 2 | 0
  Week 56: number analyzed (Participants) | 441 | 419 | 442
  Week 56 | 1 | 1 | 1
  Week 64: number analyzed (Participants) | 429 | 402 | 425
  Week 64 | 0 | 1 | 3
  Week 80: number analyzed (Participants) | 420 | 386 | 414
  Week 80 | 0 | 1 | 0

80. Secondary Outcome: Change From Baseline in Survey of Autonomic Symptom (SAS) Scores at Weeks 24, 56 and 80
Description: The SAS is a 12 item (11 for females) questionnaire, from which the total number of symptoms (0-12 for males and 0-11 for females) is calculated. Each positive symptom is rated from 1 (not at all) to 5 (a lot). The total impact score was the sum of all symptom rating scores, with 0 assigned where the participant did not have the particular symptom. The range for the total impact score is 0-60 for males and 0-55 for females, higher scores indicating higher impact.
Time Frame: Baseline, Weeks 24, 56 and 80
Population: as for outcome 77
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1000 | 997 | 996
units on a scale
  Number of symptoms reported: Baseline | 0.47 (0.76) | 0.53 (0.78) | 0.49 (0.76)
  Number of symptoms reported: Change at Week 24: number analyzed (Participants) | 546 | 543 | 532
  Number of symptoms reported: Change at Week 24 | 0.21 (1.13) | 0.18 (1.22) | 0.11 (1.20)
  Number of symptoms reported: Change at Week 56: number analyzed (Participants) | 448 | 421 | 443
  Number of symptoms reported: Change at Week 56 | 0.28 (1.19) | 0.33 (1.34) | 0.22 (1.21)
  Number of symptoms reported: Change at Week 80: number analyzed (Participants) | 423 | 391 | 414
  Number of symptoms reported: Change at Week 80 | 0.89 (1.39) | 0.94 (1.43) | 0.74 (1.22)
  Total symptom impact score: Baseline | 1.10 (1.84) | 1.23 (1.89) | 1.13 (1.82)
  Total symptom impact score: Change at Week 24: number analyzed (Participants) | 546 | 543 | 532
  Total symptom impact score: Change at Week 24 | 0.66 (2.90) | 0.52 (3.19) | 0.33 (2.99)
  Total symptom impact score: Change at Week 56: number analyzed (Participants) | 448 | 421 | 443
  Total symptom impact score: Change at Week 56 | 0.97 (3.29) | 1.21 (4.01) | 0.82 (3.40)
  Total symptom impact score: Change at Week 80: number analyzed (Participants) | 423 | 391 | 414
  Total symptom impact score: Change at Week 80 | 1.33 (3.85) | 1.31 (4.36) | 0.89 (3.65)

81. Secondary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Weeks 2, 4, 8, 16, 24, 32, 40, 48, 56, 64 and 80
Description: NIS is a standardized instrument used to evaluate participant for signs of peripheral neuropathy. NIS is the sum of scores of 37 items, from both the left and right side, where 24 items scored from 0 (normal) to 4 (paralysis), higher score indicated higher abnormality/impairment and 13 items scored from 0 (normal), 1 (decreased) and 2 (absent), higher score indicated higher impairment. NIS possible overall score ranged from 0 (no impairment) to 244 (maximum impairment), higher scores indicated increased impairment.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 32, 40, 48, 56, 64 and 80
Population: as for outcome 77
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
Number analyzed (Participants) | 1000 | 995 | 994
units on a scale
  Baseline | 1.85 (4.30) | 1.70 (4.45) | 1.87 (4.47)
  Change at Week 2: number analyzed (Participants) | 971 | 965 | 951
  Change at Week 2 | -0.22 (2.15) | -0.13 (1.40) | -0.15 (1.67)
  Change at Week 4: number analyzed (Participants) | 986 | 981 | 977
  Change at Week 4 | -0.16 (2.06) | -0.17 (1.92) | -0.19 (2.32)
  Change at Week 8: number analyzed (Participants) | 988 | 988 | 982
  Change at Week 8 | -0.27 (2.28) | -0.22 (2.08) | -0.36 (2.55)
  Change at Week 16: number analyzed (Participants) | 989 | 988 | 982
  Change at Week 16 | -0.27 (2.32) | -0.31 (2.48) | -0.47 (3.06)
  Change at Week 24: number analyzed (Participants) | 989 | 988 | 982
  Change at Week 24 | -0.32 (2.39) | -0.35 (2.76) | -0.49 (3.08)
  Change at Week 32: number analyzed (Participants) | 989 | 988 | 982
  Change at Week 32 | -0.37 (2.46) | -0.40 (2.75) | -0.53 (3.17)
  Change at Week 40: number analyzed (Participants) | 989 | 988 | 982
  Change at Week 40 | -0.35 (2.42) | -0.43 (2.80) | -0.53 (3.32)
  Change at Week 48: number analyzed (Participants) | 989 | 988 | 982
  Change at Week 48 | -0.37 (2.46) | -0.49 (3.13) | -0.55 (3.21)
  Change at Week 56: number analyzed (Participants) | 989 | 988 | 982
  Change at Week 56 | -0.35 (2.48) | -0.52 (3.26) | -0.58 (3.22)
  Change at Week 64: number analyzed (Participants) | 989 | 988 | 982
  Change at Week 64 | -0.32 (2.60) | -0.47 (3.24) | -0.57 (3.20)
  Change at Week 80: number analyzed (Participants) | 989 | 988 | 982
  Change at Week 80 | -0.35 (2.53) | -0.47 (3.35) | -0.62 (3.28)

82. Secondary Outcome: Number of Participants With Anti-Tanezumab Antibodies
Description: Human serum anti-drug antibody (ADA) samples were analyzed for the presence or absence of anti-tanezumab antibodies by using a semi quantitative enzyme linked immunosorbent assay (ELISA).
Time Frame: Baseline, Weeks 8, 16, 32, 48, 56, 64 and 80
Population: as for outcome 76
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 1002 | 998
Participants
  Baseline: number analyzed (Participants) | 993 | 985
  Baseline | 116 | 83
  Week 8: number analyzed (Participants) | 923 | 920
  Week 8 | 120 | 93
  Week 16: number analyzed (Participants) | 618 | 616
  Week 16 | 98 | 83
  Week 32: number analyzed (Participants) | 512 | 503
  Week 32 | 108 | 81
  Week 48: number analyzed (Participants) | 466 | 444
  Week 48 | 96 | 78
  Week 56: number analyzed (Participants) | 436 | 412
  Week 56 | 82 | 66
  Week 64: number analyzed (Participants) | 420 | 390
  Week 64 | 69 | 60
  Week 80: number analyzed (Participants) | 414 | 384
  Week 80 | 50 | 42

ADVERSE EVENTS:
Time Frame: Baseline up to Week 56
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Analysis performed on safety set.
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | NSAID
All-Cause Mortality (participants affected / at risk) | 4/1002 | 5/998 | 1/996
Serious Adverse Events (participants affected / at risk) | 51/1002 | 80/998 | 46/996
Other Adverse Events (participants affected / at risk) | 301/1002 | 318/998 | 264/996
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab 2.5 mg (N=1002) | Tanezumab 5 mg (N=998) | NSAID (N=996)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 3
Aortic valve incompetence (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 1
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0
Myocardial rupture (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Prinzmetal angina (Cardiac disorders) | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Entropion (Eye disorders) | 1 | 0 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Sensation of foreign body (General disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 2 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0 | 0
Escherichia pyelonephritis (Infections and infestations) | 0 | 1 | 0
Extradural abscess (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
Intervertebral discitis (Infections and infestations) | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Pelvic abscess (Infections and infestations) | 0 | 1 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 1
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Testicular abscess (Infections and infestations) | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 1 | 0
Adjacent segment degeneration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 3 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 9 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 | 17 | 4
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rapidly progressive osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 11 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Subchondral insufficiency fracture (Musculoskeletal and connective tissue disorders) | 1 | 4 | 2
Thoracic spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Cervix neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Brain stem infarction (Nervous system disorders) | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Cervical cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab 2.5 mg (N=1002) | Tanezumab 5 mg (N=998) | NSAID (N=996)
Nasopharyngitis (Infections and infestations) | 57 | 67 | 40
Upper respiratory tract infection (Infections and infestations) | 57 | 45 | 59
Fall (Injury, poisoning and procedural complications) | 65 | 52 | 46
Arthralgia (Musculoskeletal and connective tissue disorders) | 131 | 160 | 117
Back pain (Musculoskeletal and connective tissue disorders) | 34 | 55 | 34
Headache (Nervous system disorders) | 56 | 45 | 25

LIMITATIONS AND CAVEATS:
2 deaths occurred after end of study and are captured in All- cause mortality section.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT02528188/SAP_000.pdf
  • Study Protocol (2006-05-15): https://cdn.clinicaltrials.gov/large-docs/88/NCT02528188/Prot_001.pdf